CLINICAL TRIAL: NCT06964165
Title: Cohort C: Open-label Phase 2, Randomized, Controlled Multicenter Study Comparing Niraparib Versus Platinum-Taxane Doublet Chemotherapy as Neoadjuvant Treatment in Participants With Homologous Recombination-Deficient Stage III/IV Ovarian Cancer
Brief Title: A Study Comparing Niraparib Versus Platinum-Taxane Doublet Chemotherapy as Neoadjuvant Treatment in Participants With Homologous Recombination-Deficient Stage III/IV Ovarian Cancer (COHORT-C)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study stopped after meeting pre-specified futility criteria
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 213357-COHORT-C; 2023-505097-16 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Neoplasms
Keywords: Ovarian Cancer; Homologous Recombination Deficiency (HRD); Interval debulking surgery (IDS); Niraparib; Paclitaxel; Carboplatin
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort C (Niraparib) (Experimental)
  Interventions: Drug: Niraparib
- Cohort C (Carboplatin + Paclitaxel) (Experimental)
  Interventions: Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Niraparib — Niraparib will be administered
  Arms: Cohort C (Niraparib)
Drug: Carboplatin — Carboplatin will be administered
  Arms: Cohort C (Carboplatin + Paclitaxel)
Drug: Paclitaxel — Paclitaxel will be administered
  Arms: Cohort C (Carboplatin + Paclitaxel)

SUMMARY:
The goal of the study is to learn whether Niraparib or Platinum-Taxane Doublet chemotherapy is better in treating participants with Homologous Recombination Deficient (HRd) Stage III/IV Ovarian Cancer (OC). This study is a sub-study of the Master protocol -OPAL (NCT03574779)

ELIGIBILITY:
Inclusion Criteria:

* Participant has newly diagnosed Stage III or IV ovarian, fallopian tube, or primary peritoneal cancer according to the International Federation of Gynecology and Obstetrics staging criteria.
* Participants must provide sufficient tumor tissue at Prescreening and agree to undergo a central HRD tumor testing using a fully validated assay. The participants must be HRd as per central HRD tumor testing result for eligibility.

  1. Participants with a documented germline breast cancer susceptibility gene (BRCA) 1/2 deleterious or suspected deleterious mutations by Sponsor's permitted test (e.g., BRACAnalysis CDx) may be allowed to enroll prior to receiving the central test results, provided all inclusion criteria are met. However, tumor sample submitted by these participants will still be required for central HRD confirmation. The list of Sponsor's permitted tests will be provided by the Sponsor.
  2. All participants must agree to provide tumor tissue collected from IDS.
  3. Participant must provide 2 formalin-fixed paraffin-embedded tissue blocks (or slides if blocks are not available) with sufficient tumor content (as confirmed by the Sponsor's designated central and/or testing laboratory) for central HRD testing at Prescreening and for exploratory biomarker testing at Prescreening or Screening. If sufficient tumor tissue is provided at Prescreening, participants do not need to provide additional tissue at Screening.
* Participant must have completed 1 run-in cycle of carboplatin-paclitaxel and not experienced disease progression after this treatment. Completion is defined as receiving ≥50% of the prescribed dose of therapy within 5 weeks.
* Participant must not have known contraindication or uncontrolled hypersensitivity to carboplatin and paclitaxel and their excipients and no known pre-existing conditions that would preclude treatment with these agents.
* Participant must not have known contraindication or uncontrolled hypersensitivity to niraparib and its excipients.
* Participant must not have symptomatic ascites or pleural effusions as defined by the following criterion: presence of fluid in the abdominal or pleural cavities requiring removal within 1 week prior to signing the informed consent.
* Participant must agree to complete Patient-reported outcome (PRO) and work productivity questionnaires throughout the study.

Exclusion Criteria:

* Participant has low-grade or Grade 1 epithelial Ovarian Cancer (OC) or mucinous, germ cell, transitional cell, carcinosarcoma, or undifferentiated tumor.
* Participant has contraindications to surgery.
* Participant has a bowel obstruction by clinical symptoms or Computed tomography (CT) scan, subocclusive mesenteric disease, abdominal or gastrointestinal fistula, gastrointestinal perforation, or intra-abdominal abscess.
* Participant has any known history or current diagnosis of Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukemia (AML).
* Participant is at increased bleeding risk due to concurrent conditions (e.g., major injuries or major surgery within the past 28 days prior to the start of study treatment and/or history of hemorrhagic stroke, transient ischemic attack, subarachnoid hemorrhage, or clinically significant hemorrhage within the past 3 months).
* Participant is immunocompromised. Participants with splenectomy are allowed. Participants with known Human immunodeficiency virus (HIV) are allowed if they meet all of the following criteria:

  1. Cluster of differentiation 4-positive T cell count ≥350/μL and viral load <400 copies/mL
  2. No history of Acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within 12 months prior to enrollment
  3. No history of HIV-associated malignancy for the past 5 years
  4. Concurrent antiretroviral therapy as per the most current National Institutes of Health Guidelines for the Use of Antiretroviral Agents in Adults and Adolescents Living with HIV started >4 weeks prior to study enrollment
* Participant received prior treatment for high-grade non-mucinous epithelial ovarian, fallopian tube, or peritoneal cancer (e.g., prior surgery, immunotherapy, anticancer therapy [with the exception of 1 run-in cycle of carboplatin-paclitaxel], or radiation therapy).
* Participant has an active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy is not considered a form of systemic therapy (e.g., thyroid hormone or insulin).
* Participant is unable to swallow orally administered medication or has a gastrointestinal disorder likely to interfere with absorption of the study medication.
* Participant received whole blood transfusions in the 2 weeks prior to entry to the study (packed red blood cells and platelet transfusions are acceptable outside of 2 weeks prior to treatment).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (10):
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Scarborough, Maine
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Seattle, Washington
- Canada (2):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Spain (4):
  - GSK Investigational Site, A Coruña, ES
  - GSK Investigational Site, Madrid, ES
  - GSK Investigational Site, Málaga, ES
  - GSK Investigational Site, Pamplona, ES

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is a sub study of the master protocol (NCT03574779).
Groups:
- Platinum-taxane: Participants with ovarian cancer received platinum-taxane doublet chemotherapy as solution for intravenous infusion for three 21-day cycles (Cycles 1, 2 and 3). After 3 cycles of treatment, the participants underwent interval debulking surgery (IDS) with recovery period of up to 6 weeks. After IDS, all participants received another three 21-day cycles of platinum-taxane doublet chemotherapy (Cycles 4, 5, and 6), with the last cycle (Cycle 6) being optional followed by niraparib maintenance treatment for up to 36 months or until an adverse event (AE), progression of disease (PD) per RECIST v1.1.
- Niraparib: Participants with ovarian cancer received 100 milligram (mg) Niraparib capsules orally for three 21-day cycles (Cycles 1, 2 and 3). After 3 cycles of treatment, the participants underwent IDS with recovery period of up to 6 weeks. After IDS, all participants received three 21-day cycles of platinum-taxane doublet chemotherapy (Cycles 4, 5, and 6), with the last cycle (Cycle 6) being optional, followed by niraparib maintenance treatment for up to 36 months or until an AE, PD per RECIST v1.1. Participants with screening actual body weight greater than or equal (≥) to 77 kg and screening platelets count ≥ 150000 cells per microliter were administered 300 mg of Niraparib. Participants with screening actual body weight less than 77 kg or screening platelets count less than 150000 cells per microliter were administered 200 mg of niraparib.
Period: Overall Study
Arm/Group | Platinum-taxane | Niraparib
Started | 17 | 19
Completed | 0 | 0
Not Completed | 17 | 19
Not completed — Death | 4 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Study terminated by sponsor | 12 | 10
Not completed — Participant discontinued due to relocation to a long-term care facility | 0 | 1
Not completed — Participant removed due to non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Platinum-taxane | Niraparib | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 61.0 (13.67) | 58.4 (12.26) | 59.6 (12.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Pre-Interval Debulking Surgery (IDS) Unconfirmed Overall Response Rate (ORR)
Description: Pre-IDS unconfirmed ORR is defined as the percentage of participants with unconfirmed complete or partial response on study treatment pre-IDS as assessed per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by the Investigator. Complete Response (CR) is defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. Partial Response (PR) is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters
Time Frame: Up to approximately 102 weeks
Population: Intent-to-Treat population included all randomized participants whether or not randomized treatment was administered.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Platinum-taxane | Niraparib
Number analyzed (Participants) | 17 | 19
Percentage of Participants | 70.6 [44.04 to 89.69] | 31.6 [16.34 to 67.71]
Statistical Analysis 1: Comparison: Platinum-taxane vs Niraparib; Test type: Other; Difference in pre-IDS ORR = -39, 80% CI 2-sided [-56.8 to -17.7]

2. Secondary Outcome: Number of Participants With Cancer Antigen (CA)-125 Progression by Gynecological Cancer InterGroup (GCIG) CA-125 Response Criteria
Description: Serum samples were collected to assess CA-125 progression based on the GCIG CA-125 response criteria, which is defined as follows: Criteria 1 - For participants with elevated CA-125 levels pre-treatment that reduced to the normal range during the study, progression is defined as CA-125 ≥2× Upper limit of normal (ULN) on 2 occasions at least 1 week apart.; Criteria 2 - For participants with elevated CA-125 levels pre-treatment that did not reduce to the normal range during the study, progression is defined as CA-125 ≥2× the nadir value on 2 occasions at least 1 week apart.; Criteria 3 - For participants with CA-125 levels in the normal range pre-treatment, progression is defined as CA-125 ≥2× ULN on 2 occasions at least 1 week apart.
Time Frame: At week 24
Population: Intent-to-Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-taxane | Niraparib
Number analyzed (Participants) | 17 | 19
Participants
  Criteria 1 | 0 | 0
  Criteria 2 | 0 | 0
  Criteria 3 | 0 | 0

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of treatment randomization to the date of first documentation of disease progression (PD) per RECIST v1.1 or death by any cause, whichever occurs first, as determined by the Investigator. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g. percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5mm.
Time Frame: Up to approximately 154 weeks
Population: As pre-specified in Section 2 of the Statistical Analysis Plan, analyses was not performed due to low maturity (<30%) for PFS data, resulting from insufficient number of participants with events within the length of follow-up in assessing the number of events.
Arm/Group | Platinum-taxane | Niraparib
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of treatment randomization to the date of death by any cause.
Time Frame: Up to approximately 154 weeks
Population: As pre-specified in Section 2 of the Statistical Analysis Plan, analyses was not performed due to low maturity (<30%) for OS data, resulting from insufficient number of participants with events within the length of follow-up in assessing the number of events.
Arm/Group | Platinum-taxane | Niraparib
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to First Subsequent Treatment (TFST)
Description: TFST is defined as the time from the date of treatment randomization to the date of first subsequent anticancer therapy or death.
Time Frame: Up to approximately 154 weeks
Population: As pre-specified in Section 2 of the Statistical Analysis Plan, analyses was not performed due to low maturity (<30%) for TFST data, resulting from insufficient number of participants with events within the length of follow-up in assessing the number of events.
Arm/Group | Platinum-taxane | Niraparib
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Frequency and Severity of Items as Measured by Patient Reported Outcomes of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Description: The PRO-CTCAE is a patient-reported outcome measure developed to evaluate symptomatic toxicity in participants of cancer clinical studies. It characterizes the frequency and severity of adverse events using a standardized scoring system. Responses include 0 ("never" OR "none" OR "Not at all"); 1 ("Rarely" OR "Mild" OR "A little bit"); 2 ("Occasionally" OR "Moderate" OR "Somewhat"); 3 ("Frequently" OR "Severe" OR "Quite a bit") and 4 ("almost constantly" OR "very severe" OR "Very much"), with a higher score indicating a higher frequency and severity of adverse events.
Time Frame: Baseline (Predose), Day 8 and 15 of Cycle 1; Day 1, 8 and 15 of Cycle 2 and Cycle 3; Pre-IDS Evaluation, and End of Treatment (Up to approximately 154 weeks).
Population: Intent to Treat Population is included as the Overall Number of Participants Analyzed. 'Number Analyzed' refers to participants evaluable at the specified time points. The "0" participants analyzed represents that data was not collected or available for analysis at that particular time point for the respective Arms/Groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-taxane | Niraparib
Number analyzed (Participants) | 17 | 19
Participants
  Probs Tasting Food/Drink, Baseline, Severity, 0=None: number analyzed (Participants) | 14 | 17
  Probs Tasting Food/Drink, Baseline, Severity, 0=None | 10 | 9
  Probs Tasting Food/Drink, Baseline, Severity, 1=Mild: number analyzed (Participants) | 14 | 17
  Probs Tasting Food/Drink, Baseline, Severity, 1=Mild | 3 | 4
  Probs Tasting Food/Drink, Baseline, Severity, 2=Moderate: number analyzed (Participants) | 14 | 17
  Probs Tasting Food/Drink, Baseline, Severity, 2=Moderate | 1 | 3
  Probs Tasting Food/Drink, Baseline, Severity, 3=Severe: number analyzed (Participants) | 14 | 17
  Probs Tasting Food/Drink, Baseline, Severity, 3=Severe | 0 | 1
  Probs Tasting Food/Drink, Baseline, Severity, 4=Very severe: number analyzed (Participants) | 14 | 17
  Probs Tasting Food/Drink, Baseline, Severity, 4=Very severe | 0 | 0
  Probs Tasting Food/Drink, Cycle 1 Day 8, Severity, 0=None: number analyzed (Participants) | 11 | 15
  Probs Tasting Food/Drink, Cycle 1 Day 8, Severity, 0=None | 6 | 7
  Probs Tasting Food/Drink, Cycle 1 Day 8, Severity, 1=Mild: number analyzed (Participants) | 11 | 15
  Probs Tasting Food/Drink, Cycle 1 Day 8, Severity, 1=Mild | 3 | 5
  Probs Tasting Food/Drink, Cycle 1 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 11 | 15
  Probs Tasting Food/Drink, Cycle 1 Day 8, Severity, 2=Moderate | 2 | 2
  Probs Tasting Food/Drink, Cycle 1 Day 8, Severity, 3=Severe: number analyzed (Participants) | 11 | 15
  Probs Tasting Food/Drink, Cycle 1 Day 8, Severity, 3=Severe | 0 | 1
  Probs Tasting Food/Drink, Cycle 1 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 11 | 15
  Probs Tasting Food/Drink, Cycle 1 Day 8, Severity, 4=Very severe | 0 | 0
  Probs Tasting Food/Drink, Cycle 1 Day 15, Severity, 0=None: number analyzed (Participants) | 14 | 13
  Probs Tasting Food/Drink, Cycle 1 Day 15, Severity, 0=None | 12 | 6
  Probs Tasting Food/Drink, Cycle 1 Day 15, Severity, 1=Mild: number analyzed (Participants) | 14 | 13
  Probs Tasting Food/Drink, Cycle 1 Day 15, Severity, 1=Mild | 1 | 5
  Probs Tasting Food/Drink, Cycle 1 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 14 | 13
  Probs Tasting Food/Drink, Cycle 1 Day 15, Severity, 2=Moderate | 1 | 2
  Probs Tasting Food/Drink, Cycle 1 Day 15, Severity, 3=Severe: number analyzed (Participants) | 14 | 13
  Probs Tasting Food/Drink, Cycle 1 Day 15, Severity, 3=Severe | 0 | 0
  Probs Tasting Food/Drink, Cycle 1 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 14 | 13
  Probs Tasting Food/Drink, Cycle 1 Day 15, Severity, 4=Very severe | 0 | 0
  Probs Tasting Food/Drink, Cycle 2 Day 1, Severity, 0=None: number analyzed (Participants) | 11 | 14
  Probs Tasting Food/Drink, Cycle 2 Day 1, Severity, 0=None | 9 | 8
  Probs Tasting Food/Drink, Cycle 2 Day 1, Severity, 1=Mild: number analyzed (Participants) | 11 | 14
  Probs Tasting Food/Drink, Cycle 2 Day 1, Severity, 1=Mild | 2 | 4
  Probs Tasting Food/Drink, Cycle 2 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 11 | 14
  Probs Tasting Food/Drink, Cycle 2 Day 1, Severity, 2=Moderate | 0 | 1
  Probs Tasting Food/Drink, Cycle 2 Day 1, Severity, 3=Severe: number analyzed (Participants) | 11 | 14
  Probs Tasting Food/Drink, Cycle 2 Day 1, Severity, 3=Severe | 0 | 1
  Probs Tasting Food/Drink, Cycle 2 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 11 | 14
  Probs Tasting Food/Drink, Cycle 2 Day 1, Severity, 4=Very severe | 0 | 0
  Probs Tasting Food/Drink, Cycle 2 Day 8, Severity, 0=None: number analyzed (Participants) | 11 | 11
  Probs Tasting Food/Drink, Cycle 2 Day 8, Severity, 0=None | 6 | 6
  Probs Tasting Food/Drink, Cycle 2 Day 8, Severity, 1=Mild: number analyzed (Participants) | 11 | 11
  Probs Tasting Food/Drink, Cycle 2 Day 8, Severity, 1=Mild | 3 | 4
  Probs Tasting Food/Drink, Cycle 2 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 11 | 11
  Probs Tasting Food/Drink, Cycle 2 Day 8, Severity, 2=Moderate | 1 | 0
  Probs Tasting Food/Drink, Cycle 2 Day 8, Severity, 3=Severe: number analyzed (Participants) | 11 | 11
  Probs Tasting Food/Drink, Cycle 2 Day 8, Severity, 3=Severe | 1 | 1
  Probs Tasting Food/Drink, Cycle 2 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 11 | 11
  Probs Tasting Food/Drink, Cycle 2 Day 8, Severity, 4=Very severe | 0 | 0
  Probs Tasting Food/Drink, Cycle 2 Day 15, Severity, 0=None: number analyzed (Participants) | 13 | 14
  Probs Tasting Food/Drink, Cycle 2 Day 15, Severity, 0=None | 8 | 10
  Probs Tasting Food/Drink, Cycle 2 Day 15, Severity, 1=Mild: number analyzed (Participants) | 13 | 14
  Probs Tasting Food/Drink, Cycle 2 Day 15, Severity, 1=Mild | 5 | 3
  Probs Tasting Food/Drink, Cycle 2 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 13 | 14
  Probs Tasting Food/Drink, Cycle 2 Day 15, Severity, 2=Moderate | 0 | 0
  Probs Tasting Food/Drink, Cycle 2 Day 15, Severity, 3=Severe: number analyzed (Participants) | 13 | 14
  Probs Tasting Food/Drink, Cycle 2 Day 15, Severity, 3=Severe | 0 | 1
  Probs Tasting Food/Drink, Cycle 2 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 13 | 14
  Probs Tasting Food/Drink, Cycle 2 Day 15, Severity, 4=Very severe | 0 | 0
  Probs Tasting Food/Drink, Cycle 3 Day 1, Severity, 0=None: number analyzed (Participants) | 14 | 14
  Probs Tasting Food/Drink, Cycle 3 Day 1, Severity, 0=None | 12 | 8
  Probs Tasting Food/Drink, Cycle 3 Day 1, Severity, 1=Mild: number analyzed (Participants) | 14 | 14
  Probs Tasting Food/Drink, Cycle 3 Day 1, Severity, 1=Mild | 2 | 4
  Probs Tasting Food/Drink, Cycle 3 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 14 | 14
  Probs Tasting Food/Drink, Cycle 3 Day 1, Severity, 2=Moderate | 0 | 1
  Probs Tasting Food/Drink, Cycle 3 Day 1, Severity, 3=Severe: number analyzed (Participants) | 14 | 14
  Probs Tasting Food/Drink, Cycle 3 Day 1, Severity, 3=Severe | 0 | 1
  Probs Tasting Food/Drink, Cycle 3 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 14 | 14
  Probs Tasting Food/Drink, Cycle 3 Day 1, Severity, 4=Very severe | 0 | 0
  Probs Tasting Food/Drink, Cycle 3 Day 8, Severity, 0=None: number analyzed (Participants) | 10 | 10
  Probs Tasting Food/Drink, Cycle 3 Day 8, Severity, 0=None | 1 | 6
  Probs Tasting Food/Drink, Cycle 3 Day 8, Severity, 1=Mild: number analyzed (Participants) | 10 | 10
  Probs Tasting Food/Drink, Cycle 3 Day 8, Severity, 1=Mild | 3 | 3
  Probs Tasting Food/Drink, Cycle 3 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 10 | 10
  Probs Tasting Food/Drink, Cycle 3 Day 8, Severity, 2=Moderate | 4 | 0
  Probs Tasting Food/Drink, Cycle 3 Day 8, Severity, 3=Severe: number analyzed (Participants) | 10 | 10
  Probs Tasting Food/Drink, Cycle 3 Day 8, Severity, 3=Severe | 2 | 1
  Probs Tasting Food/Drink, Cycle 3 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 10 | 10
  Probs Tasting Food/Drink, Cycle 3 Day 8, Severity, 4=Very severe | 0 | 0
  Probs Tasting Food/Drink, Cycle 3 Day 15, Severity, 0=None: number analyzed (Participants) | 5 | 7
  Probs Tasting Food/Drink, Cycle 3 Day 15, Severity, 0=None | 3 | 4
  Probs Tasting Food/Drink, Cycle 3 Day 15, Severity, 1=Mild: number analyzed (Participants) | 5 | 7
  Probs Tasting Food/Drink, Cycle 3 Day 15, Severity, 1=Mild | 2 | 3
  Probs Tasting Food/Drink, Cycle 3 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 5 | 7
  Probs Tasting Food/Drink, Cycle 3 Day 15, Severity, 2=Moderate | 0 | 0
  Probs Tasting Food/Drink, Cycle 3 Day 15, Severity, 3=Severe: number analyzed (Participants) | 5 | 7
  Probs Tasting Food/Drink, Cycle 3 Day 15, Severity, 3=Severe | 0 | 0
  Probs Tasting Food/Drink, Cycle 3 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 5 | 7
  Probs Tasting Food/Drink, Cycle 3 Day 15, Severity, 4=Very severe | 0 | 0
  Probs Tasting Food/Drink, Pre-IDS Evaluation, Severity, 0=None: number analyzed (Participants) | 2 | 1
  Probs Tasting Food/Drink, Pre-IDS Evaluation, Severity, 0=None | 1 | 0
  Probs Tasting Food/Drink, Pre-IDS Evaluation, Severity, 1=Mild: number analyzed (Participants) | 2 | 1
  Probs Tasting Food/Drink, Pre-IDS Evaluation, Severity, 1=Mild | 1 | 1
  Probs Tasting Food/Drink, Pre-IDS Evaluation, Severity, 2=Moderate: number analyzed (Participants) | 2 | 1
  Probs Tasting Food/Drink, Pre-IDS Evaluation, Severity, 2=Moderate | 0 | 0
  Probs Tasting Food/Drink, Pre-IDS Evaluation, Severity, 3=Severe: number analyzed (Participants) | 2 | 1
  Probs Tasting Food/Drink, Pre-IDS Evaluation, Severity, 3=Severe | 0 | 0
  Probs Tasting Food/Drink, Pre-IDS Evaluation, Severity, 4=Very severe: number analyzed (Participants) | 2 | 1
  Probs Tasting Food/Drink, Pre-IDS Evaluation, Severity, 4=Very severe | 0 | 0
  Probs Tasting Food/Drink, End Of Treatment, Severity, 0=None: number analyzed (Participants) | 0 | 5
  Probs Tasting Food/Drink, End Of Treatment, Severity, 0=None |  | 2
  Probs Tasting Food/Drink, End Of Treatment, Severity, 1=Mild: number analyzed (Participants) | 0 | 5
  Probs Tasting Food/Drink, End Of Treatment, Severity, 1=Mild |  | 3
  Probs Tasting Food/Drink, End Of Treatment, Severity, 2=Moderate: number analyzed (Participants) | 0 | 5
  Probs Tasting Food/Drink, End Of Treatment, Severity, 2=Moderate |  | 0
  Probs Tasting Food/Drink, End Of Treatment, Severity, 3=Severe: number analyzed (Participants) | 0 | 5
  Probs Tasting Food/Drink, End Of Treatment, Severity, 3=Severe |  | 0
  Probs Tasting Food/Drink, End Of Treatment, Severity, 4=Very severe: number analyzed (Participants) | 0 | 5
  Probs Tasting Food/Drink, End Of Treatment, Severity, 4=Very severe |  | 0
  Nausea, Baseline, Severity, 0=None: number analyzed (Participants) | 7 | 9
  Nausea, Baseline, Severity, 0=None | 1 | 2
  Nausea, Baseline, Severity, 1=Mild: number analyzed (Participants) | 7 | 9
  Nausea, Baseline, Severity, 1=Mild | 5 | 5
  Nausea, Baseline, Severity, 2=Moderate: number analyzed (Participants) | 7 | 9
  Nausea, Baseline, Severity, 2=Moderate | 1 | 1
  Nausea, Baseline, Severity, 3=Severe: number analyzed (Participants) | 7 | 9
  Nausea, Baseline, Severity, 3=Severe | 0 | 0
  Nausea, Baseline, Severity, 4=Very severe: number analyzed (Participants) | 7 | 9
  Nausea, Baseline, Severity, 4=Very severe | 0 | 1
  Nausea, Baseline, Frequency, 0=Never: number analyzed (Participants) | 14 | 17
  Nausea, Baseline, Frequency, 0=Never | 7 | 8
  Nausea, Baseline, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 17
  Nausea, Baseline, Frequency, 1=Rarely | 6 | 5
  Nausea, Baseline, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 17
  Nausea, Baseline, Frequency, 2=Occasionally | 1 | 4
  Nausea, Baseline, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 17
  Nausea, Baseline, Frequency, 3=Frequently | 0 | 0
  Nausea, Baseline, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 17
  Nausea, Baseline, Frequency, 4=Almost constantly | 0 | 0
  Nausea, Cycle 1 Day 8, Severity, 0=None: number analyzed (Participants) | 9 | 7
  Nausea, Cycle 1 Day 8, Severity, 0=None | 1 | 0
  Nausea, Cycle 1 Day 8, Severity, 1=Mild: number analyzed (Participants) | 9 | 7
  Nausea, Cycle 1 Day 8, Severity, 1=Mild | 3 | 2
  Nausea, Cycle 1 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 9 | 7
  Nausea, Cycle 1 Day 8, Severity, 2=Moderate | 5 | 3
  Nausea, Cycle 1 Day 8, Severity, 3=Severe: number analyzed (Participants) | 9 | 7
  Nausea, Cycle 1 Day 8, Severity, 3=Severe | 0 | 2
  Nausea, Cycle 1 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 9 | 7
  Nausea, Cycle 1 Day 8, Severity, 4=Very severe | 0 | 0
  Nausea, Cycle 1 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 15
  Nausea, Cycle 1 Day 8, Frequency, 0=Never | 2 | 8
  Nausea, Cycle 1 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 15
  Nausea, Cycle 1 Day 8, Frequency, 1=Rarely | 4 | 2
  Nausea, Cycle 1 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 15
  Nausea, Cycle 1 Day 8, Frequency, 2=Occasionally | 4 | 3
  Nausea, Cycle 1 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 15
  Nausea, Cycle 1 Day 8, Frequency, 3=Frequently | 1 | 1
  Nausea, Cycle 1 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 15
  Nausea, Cycle 1 Day 8, Frequency, 4=Almost constantly | 0 | 1
  Nausea, Cycle 1 Day 15, Severity, 0=None: number analyzed (Participants) | 6 | 6
  Nausea, Cycle 1 Day 15, Severity, 0=None | 1 | 0
  Nausea, Cycle 1 Day 15, Severity, 1=Mild: number analyzed (Participants) | 6 | 6
  Nausea, Cycle 1 Day 15, Severity, 1=Mild | 3 | 2
  Nausea, Cycle 1 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 6 | 6
  Nausea, Cycle 1 Day 15, Severity, 2=Moderate | 2 | 3
  Nausea, Cycle 1 Day 15, Severity, 3=Severe: number analyzed (Participants) | 6 | 6
  Nausea, Cycle 1 Day 15, Severity, 3=Severe | 0 | 1
  Nausea, Cycle 1 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 6 | 6
  Nausea, Cycle 1 Day 15, Severity, 4=Very severe | 0 | 0
  Nausea, Cycle 1 Day 15, Frequency, 0=Never: number analyzed (Participants) | 14 | 13
  Nausea, Cycle 1 Day 15, Frequency, 0=Never | 8 | 7
  Nausea, Cycle 1 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 13
  Nausea, Cycle 1 Day 15, Frequency, 1=Rarely | 3 | 2
  Nausea, Cycle 1 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 13
  Nausea, Cycle 1 Day 15, Frequency, 2=Occasionally | 3 | 3
  Nausea, Cycle 1 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 13
  Nausea, Cycle 1 Day 15, Frequency, 3=Frequently | 0 | 1
  Nausea, Cycle 1 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 13
  Nausea, Cycle 1 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Nausea, Cycle 2 Day 1, Severity, 0=None: number analyzed (Participants) | 2 | 7
  Nausea, Cycle 2 Day 1, Severity, 0=None | 1 | 1
  Nausea, Cycle 2 Day 1, Severity, 1=Mild: number analyzed (Participants) | 2 | 7
  Nausea, Cycle 2 Day 1, Severity, 1=Mild | 0 | 3
  Nausea, Cycle 2 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 2 | 7
  Nausea, Cycle 2 Day 1, Severity, 2=Moderate | 1 | 1
  Nausea, Cycle 2 Day 1, Severity, 3=Severe: number analyzed (Participants) | 2 | 7
  Nausea, Cycle 2 Day 1, Severity, 3=Severe | 0 | 2
  Nausea, Cycle 2 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 2 | 7
  Nausea, Cycle 2 Day 1, Severity, 4=Very severe | 0 | 0
  Nausea, Cycle 2 Day 1, Frequency, 0=Never: number analyzed (Participants) | 11 | 14
  Nausea, Cycle 2 Day 1, Frequency, 0=Never | 9 | 7
  Nausea, Cycle 2 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 14
  Nausea, Cycle 2 Day 1, Frequency, 1=Rarely | 2 | 3
  Nausea, Cycle 2 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 14
  Nausea, Cycle 2 Day 1, Frequency, 2=Occasionally | 0 | 3
  Nausea, Cycle 2 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 14
  Nausea, Cycle 2 Day 1, Frequency, 3=Frequently | 0 | 0
  Nausea, Cycle 2 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 14
  Nausea, Cycle 2 Day 1, Frequency, 4=Almost constantly | 0 | 1
  Nausea, Cycle 2 Day 8, Severity, 0=None: number analyzed (Participants) | 5 | 5
  Nausea, Cycle 2 Day 8, Severity, 0=None | 1 | 2
  Nausea, Cycle 2 Day 8, Severity, 1=Mild: number analyzed (Participants) | 5 | 5
  Nausea, Cycle 2 Day 8, Severity, 1=Mild | 4 | 1
  Nausea, Cycle 2 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 5 | 5
  Nausea, Cycle 2 Day 8, Severity, 2=Moderate | 0 | 1
  Nausea, Cycle 2 Day 8, Severity, 3=Severe: number analyzed (Participants) | 5 | 5
  Nausea, Cycle 2 Day 8, Severity, 3=Severe | 0 | 1
  Nausea, Cycle 2 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 5 | 5
  Nausea, Cycle 2 Day 8, Severity, 4=Very severe | 0 | 0
  Nausea, Cycle 2 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 11
  Nausea, Cycle 2 Day 8, Frequency, 0=Never | 6 | 6
  Nausea, Cycle 2 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 11
  Nausea, Cycle 2 Day 8, Frequency, 1=Rarely | 3 | 3
  Nausea, Cycle 2 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 11
  Nausea, Cycle 2 Day 8, Frequency, 2=Occasionally | 2 | 1
  Nausea, Cycle 2 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 11
  Nausea, Cycle 2 Day 8, Frequency, 3=Frequently | 0 | 1
  Nausea, Cycle 2 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 11
  Nausea, Cycle 2 Day 8, Frequency, 4=Almost constantly | 0 | 0
  Nausea, Cycle 2 Day 15, Severity, 0=None: number analyzed (Participants) | 2 | 6
  Nausea, Cycle 2 Day 15, Severity, 0=None | 0 | 2
  Nausea, Cycle 2 Day 15, Severity, 1=Mild: number analyzed (Participants) | 2 | 6
  Nausea, Cycle 2 Day 15, Severity, 1=Mild | 2 | 1
  Nausea, Cycle 2 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 2 | 6
  Nausea, Cycle 2 Day 15, Severity, 2=Moderate | 0 | 2
  Nausea, Cycle 2 Day 15, Severity, 3=Severe: number analyzed (Participants) | 2 | 6
  Nausea, Cycle 2 Day 15, Severity, 3=Severe | 0 | 1
  Nausea, Cycle 2 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 2 | 6
  Nausea, Cycle 2 Day 15, Severity, 4=Very severe | 0 | 0
  Nausea, Cycle 2 Day 15, Frequency, 0=Never: number analyzed (Participants) | 13 | 14
  Nausea, Cycle 2 Day 15, Frequency, 0=Never | 11 | 8
  Nausea, Cycle 2 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 13 | 14
  Nausea, Cycle 2 Day 15, Frequency, 1=Rarely | 1 | 3
  Nausea, Cycle 2 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 13 | 14
  Nausea, Cycle 2 Day 15, Frequency, 2=Occasionally | 1 | 1
  Nausea, Cycle 2 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 13 | 14
  Nausea, Cycle 2 Day 15, Frequency, 3=Frequently | 0 | 2
  Nausea, Cycle 2 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 13 | 14
  Nausea, Cycle 2 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Nausea, Cycle 3 Day 1, Severity, 0=None: number analyzed (Participants) | 2 | 6
  Nausea, Cycle 3 Day 1, Severity, 0=None | 0 | 0
  Nausea, Cycle 3 Day 1, Severity, 1=Mild: number analyzed (Participants) | 2 | 6
  Nausea, Cycle 3 Day 1, Severity, 1=Mild | 2 | 3
  Nausea, Cycle 3 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 2 | 6
  Nausea, Cycle 3 Day 1, Severity, 2=Moderate | 0 | 1
  Nausea, Cycle 3 Day 1, Severity, 3=Severe: number analyzed (Participants) | 2 | 6
  Nausea, Cycle 3 Day 1, Severity, 3=Severe | 0 | 1
  Nausea, Cycle 3 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 2 | 6
  Nausea, Cycle 3 Day 1, Severity, 4=Very severe | 0 | 1
  Nausea, Cycle 3 Day 1, Frequency, 0=Never: number analyzed (Participants) | 14 | 14
  Nausea, Cycle 3 Day 1, Frequency, 0=Never | 12 | 8
  Nausea, Cycle 3 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 14
  Nausea, Cycle 3 Day 1, Frequency, 1=Rarely | 2 | 3
  Nausea, Cycle 3 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 14
  Nausea, Cycle 3 Day 1, Frequency, 2=Occasionally | 0 | 0
  Nausea, Cycle 3 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 14
  Nausea, Cycle 3 Day 1, Frequency, 3=Frequently | 0 | 2
  Nausea, Cycle 3 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 14
  Nausea, Cycle 3 Day 1, Frequency, 4=Almost constantly | 0 | 1
  Nausea, Cycle 3 Day 8, Severity, 0=None: number analyzed (Participants) | 5 | 5
  Nausea, Cycle 3 Day 8, Severity, 0=None | 1 | 1
  Nausea, Cycle 3 Day 8, Severity, 1=Mild: number analyzed (Participants) | 5 | 5
  Nausea, Cycle 3 Day 8, Severity, 1=Mild | 1 | 2
  Nausea, Cycle 3 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 5 | 5
  Nausea, Cycle 3 Day 8, Severity, 2=Moderate | 2 | 1
  Nausea, Cycle 3 Day 8, Severity, 3=Severe: number analyzed (Participants) | 5 | 5
  Nausea, Cycle 3 Day 8, Severity, 3=Severe | 1 | 1
  Nausea, Cycle 3 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 5 | 5
  Nausea, Cycle 3 Day 8, Severity, 4=Very severe | 0 | 0
  Nausea, Cycle 3 Day 8, Frequency, 0=Never: number analyzed (Participants) | 10 | 10
  Nausea, Cycle 3 Day 8, Frequency, 0=Never | 5 | 5
  Nausea, Cycle 3 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 10 | 10
  Nausea, Cycle 3 Day 8, Frequency, 1=Rarely | 2 | 2
  Nausea, Cycle 3 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 10 | 10
  Nausea, Cycle 3 Day 8, Frequency, 2=Occasionally | 0 | 2
  Nausea, Cycle 3 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 10 | 10
  Nausea, Cycle 3 Day 8, Frequency, 3=Frequently | 3 | 1
  Nausea, Cycle 3 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 10 | 10
  Nausea, Cycle 3 Day 8, Frequency, 4=Almost constantly | 0 | 0
  Nausea, Cycle 3 Day 15, Severity, 0=None: number analyzed (Participants) | 4 | 3
  Nausea, Cycle 3 Day 15, Severity, 0=None | 0 | 2
  Nausea, Cycle 3 Day 15, Severity, 1=Mild: number analyzed (Participants) | 4 | 3
  Nausea, Cycle 3 Day 15, Severity, 1=Mild | 3 | 0
  Nausea, Cycle 3 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 4 | 3
  Nausea, Cycle 3 Day 15, Severity, 2=Moderate | 1 | 1
  Nausea, Cycle 3 Day 15, Severity, 3=Severe: number analyzed (Participants) | 4 | 3
  Nausea, Cycle 3 Day 15, Severity, 3=Severe | 0 | 0
  Nausea, Cycle 3 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 4 | 3
  Nausea, Cycle 3 Day 15, Severity, 4=Very severe | 0 | 0
  Nausea, Cycle 3 Day 15, Frequency, 0=Never: number analyzed (Participants) | 5 | 7
  Nausea, Cycle 3 Day 15, Frequency, 0=Never | 1 | 4
  Nausea, Cycle 3 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 5 | 7
  Nausea, Cycle 3 Day 15, Frequency, 1=Rarely | 3 | 2
  Nausea, Cycle 3 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 5 | 7
  Nausea, Cycle 3 Day 15, Frequency, 2=Occasionally | 1 | 1
  Nausea, Cycle 3 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 5 | 7
  Nausea, Cycle 3 Day 15, Frequency, 3=Frequently | 0 | 0
  Nausea, Cycle 3 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 5 | 7
  Nausea, Cycle 3 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Nausea, Pre-IDS Evaluation, Frequency, 0=Never: number analyzed (Participants) | 2 | 1
  Nausea, Pre-IDS Evaluation, Frequency, 0=Never | 2 | 1
  Nausea, Pre-IDS Evaluation, Frequency, 1=Rarely: number analyzed (Participants) | 2 | 1
  Nausea, Pre-IDS Evaluation, Frequency, 1=Rarely | 0 | 0
  Nausea, Pre-IDS Evaluation, Frequency, 2=Occasionally: number analyzed (Participants) | 2 | 1
  Nausea, Pre-IDS Evaluation, Frequency, 2=Occasionally | 0 | 0
  Nausea, Pre-IDS Evaluation, Frequency, 3=Frequently: number analyzed (Participants) | 2 | 1
  Nausea, Pre-IDS Evaluation, Frequency, 3=Frequently | 0 | 0
  Nausea, Pre-IDS Evaluation, Frequency, 4=Almost constantly: number analyzed (Participants) | 2 | 1
  Nausea, Pre-IDS Evaluation, Frequency, 4=Almost constantly | 0 | 0
  Nausea, End Of Treatment, Severity, 0=None: number analyzed (Participants) | 0 | 4
  Nausea, End Of Treatment, Severity, 0=None |  | 1
  Nausea, End Of Treatment, Severity, 1=Mild: number analyzed (Participants) | 0 | 4
  Nausea, End Of Treatment, Severity, 1=Mild |  | 3
  Nausea, End Of Treatment, Severity, 2=Moderate: number analyzed (Participants) | 0 | 4
  Nausea, End Of Treatment, Severity, 2=Moderate |  | 0
  Nausea, End Of Treatment, Severity, 3=Severe: number analyzed (Participants) | 0 | 4
  Nausea, End Of Treatment, Severity, 3=Severe |  | 0
  Nausea, End Of Treatment, Severity, 4=Very severe: number analyzed (Participants) | 0 | 4
  Nausea, End Of Treatment, Severity, 4=Very severe |  | 0
  Nausea, End Of Treatment, Frequency, 0=Never: number analyzed (Participants) | 0 | 5
  Nausea, End Of Treatment, Frequency, 0=Never |  | 1
  Nausea, End Of Treatment, Frequency, 1=Rarely: number analyzed (Participants) | 0 | 5
  Nausea, End Of Treatment, Frequency, 1=Rarely |  | 3
  Nausea, End Of Treatment, Frequency, 2=Occasionally: number analyzed (Participants) | 0 | 5
  Nausea, End Of Treatment, Frequency, 2=Occasionally |  | 1
  Nausea, End Of Treatment, Frequency, 3=Frequently: number analyzed (Participants) | 0 | 5
  Nausea, End Of Treatment, Frequency, 3=Frequently |  | 0
  Nausea, End Of Treatment, Frequency, 4=Almost constantly: number analyzed (Participants) | 0 | 5
  Nausea, End Of Treatment, Frequency, 4=Almost constantly |  | 0
  Vomiting, Baseline, Severity, 0=None: number analyzed (Participants) | 1 | 1
  Vomiting, Baseline, Severity, 0=None | 0 | 0
  Vomiting, Baseline, Severity, 1=Mild: number analyzed (Participants) | 1 | 1
  Vomiting, Baseline, Severity, 1=Mild | 1 | 0
  Vomiting, Baseline, Severity, 2=Moderate: number analyzed (Participants) | 1 | 1
  Vomiting, Baseline, Severity, 2=Moderate | 0 | 1
  Vomiting, Baseline, Severity, 3=Severe: number analyzed (Participants) | 1 | 1
  Vomiting, Baseline, Severity, 3=Severe | 0 | 0
  Vomiting, Baseline, Severity, 4=Very severe: number analyzed (Participants) | 1 | 1
  Vomiting, Baseline, Severity, 4=Very severe | 0 | 0
  Vomiting, Baseline, Frequency, 0=Never: number analyzed (Participants) | 14 | 17
  Vomiting, Baseline, Frequency, 0=Never | 13 | 16
  Vomiting, Baseline, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 17
  Vomiting, Baseline, Frequency, 1=Rarely | 1 | 0
  Vomiting, Baseline, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 17
  Vomiting, Baseline, Frequency, 2=Occasionally | 0 | 1
  Vomiting, Baseline, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 17
  Vomiting, Baseline, Frequency, 3=Frequently | 0 | 0
  Vomiting, Baseline, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 17
  Vomiting, Baseline, Frequency, 4=Almost constantly | 0 | 0
  Vomiting, Cycle 1 Day 8, Severity, 0=None: number analyzed (Participants) | 1 | 3
  Vomiting, Cycle 1 Day 8, Severity, 0=None | 0 | 0
  Vomiting, Cycle 1 Day 8, Severity, 1=Mild: number analyzed (Participants) | 1 | 3
  Vomiting, Cycle 1 Day 8, Severity, 1=Mild | 1 | 2
  Vomiting, Cycle 1 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 1 | 3
  Vomiting, Cycle 1 Day 8, Severity, 2=Moderate | 0 | 1
  Vomiting, Cycle 1 Day 8, Severity, 3=Severe: number analyzed (Participants) | 1 | 3
  Vomiting, Cycle 1 Day 8, Severity, 3=Severe | 0 | 0
  Vomiting, Cycle 1 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 1 | 3
  Vomiting, Cycle 1 Day 8, Severity, 4=Very severe | 0 | 0
  Vomiting, Cycle 1 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 15
  Vomiting, Cycle 1 Day 8, Frequency, 0=Never | 10 | 12
  Vomiting, Cycle 1 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 15
  Vomiting, Cycle 1 Day 8, Frequency, 1=Rarely | 1 | 2
  Vomiting, Cycle 1 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 15
  Vomiting, Cycle 1 Day 8, Frequency, 2=Occasionally | 0 | 1
  Vomiting, Cycle 1 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 15
  Vomiting, Cycle 1 Day 8, Frequency, 3=Frequently | 0 | 0
  Vomiting, Cycle 1 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 15
  Vomiting, Cycle 1 Day 8, Frequency, 4=Almost constantly | 0 | 0
  Vomiting, Cycle 1 Day 15, Severity, 0=None: number analyzed (Participants) | 0 | 1
  Vomiting, Cycle 1 Day 15, Severity, 0=None |  | 0
  Vomiting, Cycle 1 Day 15, Severity, 1=Mild: number analyzed (Participants) | 0 | 1
  Vomiting, Cycle 1 Day 15, Severity, 1=Mild |  | 1
  Vomiting, Cycle 1 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 0 | 1
  Vomiting, Cycle 1 Day 15, Severity, 2=Moderate |  | 0
  Vomiting, Cycle 1 Day 15, Severity, 3=Severe: number analyzed (Participants) | 0 | 1
  Vomiting, Cycle 1 Day 15, Severity, 3=Severe |  | 0
  Vomiting, Cycle 1 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 0 | 1
  Vomiting, Cycle 1 Day 15, Severity, 4=Very severe |  | 0
  Vomiting, Cycle 1 Day 15, Frequency, 0=Never: number analyzed (Participants) | 14 | 13
  Vomiting, Cycle 1 Day 15, Frequency, 0=Never | 14 | 12
  Vomiting, Cycle 1 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 13
  Vomiting, Cycle 1 Day 15, Frequency, 1=Rarely | 0 | 1
  Vomiting, Cycle 1 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 13
  Vomiting, Cycle 1 Day 15, Frequency, 2=Occasionally | 0 | 0
  Vomiting, Cycle 1 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 13
  Vomiting, Cycle 1 Day 15, Frequency, 3=Frequently | 0 | 0
  Vomiting, Cycle 1 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 13
  Vomiting, Cycle 1 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Vomiting, Cycle 2 Day 1, Severity, 0=None: number analyzed (Participants) | 0 | 2
  Vomiting, Cycle 2 Day 1, Severity, 0=None |  | 0
  Vomiting, Cycle 2 Day 1, Severity, 1=Mild: number analyzed (Participants) | 0 | 2
  Vomiting, Cycle 2 Day 1, Severity, 1=Mild |  | 1
  Vomiting, Cycle 2 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 0 | 2
  Vomiting, Cycle 2 Day 1, Severity, 2=Moderate |  | 1
  Vomiting, Cycle 2 Day 1, Severity, 3=Severe: number analyzed (Participants) | 0 | 2
  Vomiting, Cycle 2 Day 1, Severity, 3=Severe |  | 0
  Vomiting, Cycle 2 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 0 | 2
  Vomiting, Cycle 2 Day 1, Severity, 4=Very severe |  | 0
  Vomiting, Cycle 2 Day 1, Frequency, 0=Never: number analyzed (Participants) | 11 | 14
  Vomiting, Cycle 2 Day 1, Frequency, 0=Never | 11 | 12
  Vomiting, Cycle 2 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 14
  Vomiting, Cycle 2 Day 1, Frequency, 1=Rarely | 0 | 2
  Vomiting, Cycle 2 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 14
  Vomiting, Cycle 2 Day 1, Frequency, 2=Occasionally | 0 | 0
  Vomiting, Cycle 2 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 14
  Vomiting, Cycle 2 Day 1, Frequency, 3=Frequently | 0 | 0
  Vomiting, Cycle 2 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 14
  Vomiting, Cycle 2 Day 1, Frequency, 4=Almost constantly | 0 | 0
  Vomiting, Cycle 2 Day 8, Severity, 0=None: number analyzed (Participants) | 1 | 2
  Vomiting, Cycle 2 Day 8, Severity, 0=None | 0 | 0
  Vomiting, Cycle 2 Day 8, Severity, 1=Mild: number analyzed (Participants) | 1 | 2
  Vomiting, Cycle 2 Day 8, Severity, 1=Mild | 1 | 1
  Vomiting, Cycle 2 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 1 | 2
  Vomiting, Cycle 2 Day 8, Severity, 2=Moderate | 0 | 1
  Vomiting, Cycle 2 Day 8, Severity, 3=Severe: number analyzed (Participants) | 1 | 2
  Vomiting, Cycle 2 Day 8, Severity, 3=Severe | 0 | 0
  Vomiting, Cycle 2 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 1 | 2
  Vomiting, Cycle 2 Day 8, Severity, 4=Very severe | 0 | 0
  Vomiting, Cycle 2 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 11
  Vomiting, Cycle 2 Day 8, Frequency, 0=Never | 10 | 9
  Vomiting, Cycle 2 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 11
  Vomiting, Cycle 2 Day 8, Frequency, 1=Rarely | 1 | 2
  Vomiting, Cycle 2 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 11
  Vomiting, Cycle 2 Day 8, Frequency, 2=Occasionally | 0 | 0
  Vomiting, Cycle 2 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 11
  Vomiting, Cycle 2 Day 8, Frequency, 3=Frequently | 0 | 0
  Vomiting, Cycle 2 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 11
  Vomiting, Cycle 2 Day 8, Frequency, 4=Almost constantly | 0 | 0
  Vomiting, Cycle 2 Day 15, Severity, 0=None: number analyzed (Participants) | 1 | 1
  Vomiting, Cycle 2 Day 15, Severity, 0=None | 0 | 1
  Vomiting, Cycle 2 Day 15, Severity, 1=Mild: number analyzed (Participants) | 1 | 1
  Vomiting, Cycle 2 Day 15, Severity, 1=Mild | 1 | 0
  Vomiting, Cycle 2 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 1 | 1
  Vomiting, Cycle 2 Day 15, Severity, 2=Moderate | 0 | 0
  Vomiting, Cycle 2 Day 15, Severity, 3=Severe: number analyzed (Participants) | 1 | 1
  Vomiting, Cycle 2 Day 15, Severity, 3=Severe | 0 | 0
  Vomiting, Cycle 2 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 1 | 1
  Vomiting, Cycle 2 Day 15, Severity, 4=Very severe | 0 | 0
  Vomiting, Cycle 2 Day 15, Frequency, 0=Never: number analyzed (Participants) | 13 | 14
  Vomiting, Cycle 2 Day 15, Frequency, 0=Never | 12 | 13
  Vomiting, Cycle 2 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 13 | 14
  Vomiting, Cycle 2 Day 15, Frequency, 1=Rarely | 1 | 1
  Vomiting, Cycle 2 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 13 | 14
  Vomiting, Cycle 2 Day 15, Frequency, 2=Occasionally | 0 | 0
  Vomiting, Cycle 2 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 13 | 14
  Vomiting, Cycle 2 Day 15, Frequency, 3=Frequently | 0 | 0
  Vomiting, Cycle 2 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 13 | 14
  Vomiting, Cycle 2 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Vomiting, Cycle 3 Day 1, Severity, 0=None: number analyzed (Participants) | 0 | 3
  Vomiting, Cycle 3 Day 1, Severity, 0=None |  | 0
  Vomiting, Cycle 3 Day 1, Severity, 1=Mild: number analyzed (Participants) | 0 | 3
  Vomiting, Cycle 3 Day 1, Severity, 1=Mild |  | 1
  Vomiting, Cycle 3 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 0 | 3
  Vomiting, Cycle 3 Day 1, Severity, 2=Moderate |  | 0
  Vomiting, Cycle 3 Day 1, Severity, 3=Severe: number analyzed (Participants) | 0 | 3
  Vomiting, Cycle 3 Day 1, Severity, 3=Severe |  | 2
  Vomiting, Cycle 3 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 0 | 3
  Vomiting, Cycle 3 Day 1, Severity, 4=Very severe |  | 0
  Vomiting, Cycle 3 Day 1, Frequency, 0=Never: number analyzed (Participants) | 14 | 14
  Vomiting, Cycle 3 Day 1, Frequency, 0=Never | 14 | 11
  Vomiting, Cycle 3 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 14
  Vomiting, Cycle 3 Day 1, Frequency, 1=Rarely | 0 | 2
  Vomiting, Cycle 3 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 14
  Vomiting, Cycle 3 Day 1, Frequency, 2=Occasionally | 0 | 0
  Vomiting, Cycle 3 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 14
  Vomiting, Cycle 3 Day 1, Frequency, 3=Frequently | 0 | 1
  Vomiting, Cycle 3 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 14
  Vomiting, Cycle 3 Day 1, Frequency, 4=Almost constantly | 0 | 0
  Vomiting, Cycle 3 Day 8, Severity, 0=None: number analyzed (Participants) | 1 | 1
  Vomiting, Cycle 3 Day 8, Severity, 0=None | 0 | 0
  Vomiting, Cycle 3 Day 8, Severity, 1=Mild: number analyzed (Participants) | 1 | 1
  Vomiting, Cycle 3 Day 8, Severity, 1=Mild | 0 | 0
  Vomiting, Cycle 3 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 1 | 1
  Vomiting, Cycle 3 Day 8, Severity, 2=Moderate | 1 | 1
  Vomiting, Cycle 3 Day 8, Severity, 3=Severe: number analyzed (Participants) | 1 | 1
  Vomiting, Cycle 3 Day 8, Severity, 3=Severe | 0 | 0
  Vomiting, Cycle 3 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 1 | 1
  Vomiting, Cycle 3 Day 8, Severity, 4=Very severe | 0 | 0
  Vomiting, Cycle 3 Day 8, Frequency, 0=Never: number analyzed (Participants) | 10 | 10
  Vomiting, Cycle 3 Day 8, Frequency, 0=Never | 9 | 9
  Vomiting, Cycle 3 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 10 | 10
  Vomiting, Cycle 3 Day 8, Frequency, 1=Rarely | 0 | 0
  Vomiting, Cycle 3 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 10 | 10
  Vomiting, Cycle 3 Day 8, Frequency, 2=Occasionally | 1 | 1
  Vomiting, Cycle 3 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 10 | 10
  Vomiting, Cycle 3 Day 8, Frequency, 3=Frequently | 0 | 0
  Vomiting, Cycle 3 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 10 | 10
  Vomiting, Cycle 3 Day 8, Frequency, 4=Almost constantly | 0 | 0
  Vomiting, Cycle 3 Day 15, Severity, 0=None: number analyzed (Participants) | 0 | 2
  Vomiting, Cycle 3 Day 15, Severity, 0=None |  | 1
  Vomiting, Cycle 3 Day 15, Severity, 1=Mild: number analyzed (Participants) | 0 | 2
  Vomiting, Cycle 3 Day 15, Severity, 1=Mild |  | 0
  Vomiting, Cycle 3 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 0 | 2
  Vomiting, Cycle 3 Day 15, Severity, 2=Moderate |  | 1
  Vomiting, Cycle 3 Day 15, Severity, 3=Severe: number analyzed (Participants) | 0 | 2
  Vomiting, Cycle 3 Day 15, Severity, 3=Severe |  | 0
  Vomiting, Cycle 3 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 0 | 2
  Vomiting, Cycle 3 Day 15, Severity, 4=Very severe |  | 0
  Vomiting, Cycle 3 Day 15, Frequency, 0=Never: number analyzed (Participants) | 5 | 7
  Vomiting, Cycle 3 Day 15, Frequency, 0=Never | 5 | 5
  Vomiting, Cycle 3 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 5 | 7
  Vomiting, Cycle 3 Day 15, Frequency, 1=Rarely | 0 | 1
  Vomiting, Cycle 3 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 5 | 7
  Vomiting, Cycle 3 Day 15, Frequency, 2=Occasionally | 0 | 1
  Vomiting, Cycle 3 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 5 | 7
  Vomiting, Cycle 3 Day 15, Frequency, 3=Frequently | 0 | 0
  Vomiting, Cycle 3 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 5 | 7
  Vomiting, Cycle 3 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Vomiting, Pre-IDS Evaluation, Frequency, 0=Never: number analyzed (Participants) | 2 | 1
  Vomiting, Pre-IDS Evaluation, Frequency, 0=Never | 2 | 1
  Vomiting, Pre-IDS Evaluation, Frequency, 1=Rarely: number analyzed (Participants) | 2 | 1
  Vomiting, Pre-IDS Evaluation, Frequency, 1=Rarely | 0 | 0
  Vomiting, Pre-IDS Evaluation, Frequency, 2=Occasionally: number analyzed (Participants) | 2 | 1
  Vomiting, Pre-IDS Evaluation, Frequency, 2=Occasionally | 0 | 0
  Vomiting, Pre-IDS Evaluation, Frequency, 3=Frequently: number analyzed (Participants) | 2 | 1
  Vomiting, Pre-IDS Evaluation, Frequency, 3=Frequently | 0 | 0
  Vomiting, Pre-IDS Evaluation, Frequency, 4=Almost constantly: number analyzed (Participants) | 2 | 1
  Vomiting, Pre-IDS Evaluation, Frequency, 4=Almost constantly | 0 | 0
  Vomiting, End Of Treatment, Severity, 0=None: number analyzed (Participants) | 0 | 1
  Vomiting, End Of Treatment, Severity, 0=None |  | 0
  Vomiting, End Of Treatment, Severity, 1=Mild: number analyzed (Participants) | 0 | 1
  Vomiting, End Of Treatment, Severity, 1=Mild |  | 1
  Vomiting, End Of Treatment, Severity, 2=Moderate: number analyzed (Participants) | 0 | 1
  Vomiting, End Of Treatment, Severity, 2=Moderate |  | 0
  Vomiting, End Of Treatment, Severity, 3=Severe: number analyzed (Participants) | 0 | 1
  Vomiting, End Of Treatment, Severity, 3=Severe |  | 0
  Vomiting, End Of Treatment, Severity, 4=Very severe: number analyzed (Participants) | 0 | 1
  Vomiting, End Of Treatment, Severity, 4=Very severe |  | 0
  Vomiting, End Of Treatment, Frequency, 0=Never: number analyzed (Participants) | 0 | 5
  Vomiting, End Of Treatment, Frequency, 0=Never |  | 4
  Vomiting, End Of Treatment, Frequency, 1=Rarely: number analyzed (Participants) | 0 | 5
  Vomiting, End Of Treatment, Frequency, 1=Rarely |  | 0
  Vomiting, End Of Treatment, Frequency, 2=Occasionally: number analyzed (Participants) | 0 | 5
  Vomiting, End Of Treatment, Frequency, 2=Occasionally |  | 1
  Vomiting, End Of Treatment, Frequency, 3=Frequently: number analyzed (Participants) | 0 | 5
  Vomiting, End Of Treatment, Frequency, 3=Frequently |  | 0
  Vomiting, End Of Treatment, Frequency, 4=Almost constantly: number analyzed (Participants) | 0 | 5
  Vomiting, End Of Treatment, Frequency, 4=Almost constantly |  | 0
  Bloating of Abdomen, Baseline, Severity, 0=None: number analyzed (Participants) | 11 | 8
  Bloating of Abdomen, Baseline, Severity, 0=None | 0 | 0
  Bloating of Abdomen, Baseline, Severity, 1=Mild: number analyzed (Participants) | 11 | 8
  Bloating of Abdomen, Baseline, Severity, 1=Mild | 7 | 5
  Bloating of Abdomen, Baseline, Severity, 2=Moderate: number analyzed (Participants) | 11 | 8
  Bloating of Abdomen, Baseline, Severity, 2=Moderate | 3 | 3
  Bloating of Abdomen, Baseline, Severity, 3=Severe: number analyzed (Participants) | 11 | 8
  Bloating of Abdomen, Baseline, Severity, 3=Severe | 1 | 0
  Bloating of Abdomen, Baseline, Severity, 4=Very severe: number analyzed (Participants) | 11 | 8
  Bloating of Abdomen, Baseline, Severity, 4=Very severe | 0 | 0
  Bloating of Abdomen, Baseline, Frequency, 0=Never: number analyzed (Participants) | 14 | 17
  Bloating of Abdomen, Baseline, Frequency, 0=Never | 3 | 9
  Bloating of Abdomen, Baseline, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 17
  Bloating of Abdomen, Baseline, Frequency, 1=Rarely | 5 | 3
  Bloating of Abdomen, Baseline, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 17
  Bloating of Abdomen, Baseline, Frequency, 2=Occasionally | 3 | 4
  Bloating of Abdomen, Baseline, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 17
  Bloating of Abdomen, Baseline, Frequency, 3=Frequently | 1 | 1
  Bloating of Abdomen, Baseline, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 17
  Bloating of Abdomen, Baseline, Frequency, 4=Almost constantly | 2 | 0
  Bloating of Abdomen, Cycle 1 Day 8, Severity, 0=None: number analyzed (Participants) | 8 | 9
  Bloating of Abdomen, Cycle 1 Day 8, Severity, 0=None | 0 | 0
  Bloating of Abdomen, Cycle 1 Day 8, Severity, 1=Mild: number analyzed (Participants) | 8 | 9
  Bloating of Abdomen, Cycle 1 Day 8, Severity, 1=Mild | 3 | 5
  Bloating of Abdomen, Cycle 1 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 8 | 9
  Bloating of Abdomen, Cycle 1 Day 8, Severity, 2=Moderate | 4 | 3
  Bloating of Abdomen, Cycle 1 Day 8, Severity, 3=Severe: number analyzed (Participants) | 8 | 9
  Bloating of Abdomen, Cycle 1 Day 8, Severity, 3=Severe | 1 | 1
  Bloating of Abdomen, Cycle 1 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 8 | 9
  Bloating of Abdomen, Cycle 1 Day 8, Severity, 4=Very severe | 0 | 0
  Bloating of Abdomen, Cycle 1 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 15
  Bloating of Abdomen, Cycle 1 Day 8, Frequency, 0=Never | 3 | 6
  Bloating of Abdomen, Cycle 1 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 15
  Bloating of Abdomen, Cycle 1 Day 8, Frequency, 1=Rarely | 1 | 3
  Bloating of Abdomen, Cycle 1 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 15
  Bloating of Abdomen, Cycle 1 Day 8, Frequency, 2=Occasionally | 5 | 4
  Bloating of Abdomen, Cycle 1 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 15
  Bloating of Abdomen, Cycle 1 Day 8, Frequency, 3=Frequently | 1 | 0
  Bloating of Abdomen, Cycle 1 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 15
  Bloating of Abdomen, Cycle 1 Day 8, Frequency, 4=Almost constantly | 1 | 2
  Bloating of Abdomen, Cycle 1 Day 15, Severity, 0=None: number analyzed (Participants) | 8 | 9
  Bloating of Abdomen, Cycle 1 Day 15, Severity, 0=None | 0 | 0
  Bloating of Abdomen, Cycle 1 Day 15, Severity, 1=Mild: number analyzed (Participants) | 8 | 9
  Bloating of Abdomen, Cycle 1 Day 15, Severity, 1=Mild | 5 | 2
  Bloating of Abdomen, Cycle 1 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 8 | 9
  Bloating of Abdomen, Cycle 1 Day 15, Severity, 2=Moderate | 3 | 5
  Bloating of Abdomen, Cycle 1 Day 15, Severity, 3=Severe: number analyzed (Participants) | 8 | 9
  Bloating of Abdomen, Cycle 1 Day 15, Severity, 3=Severe | 0 | 1
  Bloating of Abdomen, Cycle 1 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 8 | 9
  Bloating of Abdomen, Cycle 1 Day 15, Severity, 4=Very severe | 0 | 1
  Bloating of Abdomen, Cycle 1 Day 15, Frequency, 0=Never: number analyzed (Participants) | 14 | 13
  Bloating of Abdomen, Cycle 1 Day 15, Frequency, 0=Never | 6 | 4
  Bloating of Abdomen, Cycle 1 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 13
  Bloating of Abdomen, Cycle 1 Day 15, Frequency, 1=Rarely | 5 | 3
  Bloating of Abdomen, Cycle 1 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 13
  Bloating of Abdomen, Cycle 1 Day 15, Frequency, 2=Occasionally | 0 | 4
  Bloating of Abdomen, Cycle 1 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 13
  Bloating of Abdomen, Cycle 1 Day 15, Frequency, 3=Frequently | 2 | 0
  Bloating of Abdomen, Cycle 1 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 13
  Bloating of Abdomen, Cycle 1 Day 15, Frequency, 4=Almost constantly | 1 | 2
  Bloating of Abdomen, Cycle 2 Day 1, Severity, 0=None: number analyzed (Participants) | 7 | 6
  Bloating of Abdomen, Cycle 2 Day 1, Severity, 0=None | 0 | 0
  Bloating of Abdomen, Cycle 2 Day 1, Severity, 1=Mild: number analyzed (Participants) | 7 | 6
  Bloating of Abdomen, Cycle 2 Day 1, Severity, 1=Mild | 7 | 3
  Bloating of Abdomen, Cycle 2 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 7 | 6
  Bloating of Abdomen, Cycle 2 Day 1, Severity, 2=Moderate | 0 | 3
  Bloating of Abdomen, Cycle 2 Day 1, Severity, 3=Severe: number analyzed (Participants) | 7 | 6
  Bloating of Abdomen, Cycle 2 Day 1, Severity, 3=Severe | 0 | 0
  Bloating of Abdomen, Cycle 2 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 7 | 6
  Bloating of Abdomen, Cycle 2 Day 1, Severity, 4=Very severe | 0 | 0
  Bloating of Abdomen, Cycle 2 Day 1, Frequency, 0=Never: number analyzed (Participants) | 11 | 14
  Bloating of Abdomen, Cycle 2 Day 1, Frequency, 0=Never | 4 | 8
  Bloating of Abdomen, Cycle 2 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 14
  Bloating of Abdomen, Cycle 2 Day 1, Frequency, 1=Rarely | 6 | 3
  Bloating of Abdomen, Cycle 2 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 14
  Bloating of Abdomen, Cycle 2 Day 1, Frequency, 2=Occasionally | 1 | 3
  Bloating of Abdomen, Cycle 2 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 14
  Bloating of Abdomen, Cycle 2 Day 1, Frequency, 3=Frequently | 0 | 0
  Bloating of Abdomen, Cycle 2 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 14
  Bloating of Abdomen, Cycle 2 Day 1, Frequency, 4=Almost constantly | 0 | 0
  Bloating of Abdomen, Cycle 2 Day 8, Severity, 0=None: number analyzed (Participants) | 8 | 7
  Bloating of Abdomen, Cycle 2 Day 8, Severity, 0=None | 0 | 0
  Bloating of Abdomen, Cycle 2 Day 8, Severity, 1=Mild: number analyzed (Participants) | 8 | 7
  Bloating of Abdomen, Cycle 2 Day 8, Severity, 1=Mild | 4 | 4
  Bloating of Abdomen, Cycle 2 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 8 | 7
  Bloating of Abdomen, Cycle 2 Day 8, Severity, 2=Moderate | 2 | 3
  Bloating of Abdomen, Cycle 2 Day 8, Severity, 3=Severe: number analyzed (Participants) | 8 | 7
  Bloating of Abdomen, Cycle 2 Day 8, Severity, 3=Severe | 2 | 0
  Bloating of Abdomen, Cycle 2 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 8 | 7
  Bloating of Abdomen, Cycle 2 Day 8, Severity, 4=Very severe | 0 | 0
  Bloating of Abdomen, Cycle 2 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 11
  Bloating of Abdomen, Cycle 2 Day 8, Frequency, 0=Never | 3 | 4
  Bloating of Abdomen, Cycle 2 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 11
  Bloating of Abdomen, Cycle 2 Day 8, Frequency, 1=Rarely | 3 | 4
  Bloating of Abdomen, Cycle 2 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 11
  Bloating of Abdomen, Cycle 2 Day 8, Frequency, 2=Occasionally | 3 | 2
  Bloating of Abdomen, Cycle 2 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 11
  Bloating of Abdomen, Cycle 2 Day 8, Frequency, 3=Frequently | 2 | 1
  Bloating of Abdomen, Cycle 2 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 11
  Bloating of Abdomen, Cycle 2 Day 8, Frequency, 4=Almost constantly | 0 | 0
  Bloating of Abdomen, Cycle 2 Day 15, Severity, 0=None: number analyzed (Participants) | 7 | 9
  Bloating of Abdomen, Cycle 2 Day 15, Severity, 0=None | 0 | 1
  Bloating of Abdomen, Cycle 2 Day 15, Severity, 1=Mild: number analyzed (Participants) | 7 | 9
  Bloating of Abdomen, Cycle 2 Day 15, Severity, 1=Mild | 5 | 3
  Bloating of Abdomen, Cycle 2 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 7 | 9
  Bloating of Abdomen, Cycle 2 Day 15, Severity, 2=Moderate | 2 | 2
  Bloating of Abdomen, Cycle 2 Day 15, Severity, 3=Severe: number analyzed (Participants) | 7 | 9
  Bloating of Abdomen, Cycle 2 Day 15, Severity, 3=Severe | 0 | 3
  Bloating of Abdomen, Cycle 2 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 7 | 9
  Bloating of Abdomen, Cycle 2 Day 15, Severity, 4=Very severe | 0 | 0
  Bloating of Abdomen, Cycle 2 Day 15, Frequency, 0=Never: number analyzed (Participants) | 13 | 14
  Bloating of Abdomen, Cycle 2 Day 15, Frequency, 0=Never | 6 | 5
  Bloating of Abdomen, Cycle 2 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 13 | 14
  Bloating of Abdomen, Cycle 2 Day 15, Frequency, 1=Rarely | 2 | 4
  Bloating of Abdomen, Cycle 2 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 13 | 14
  Bloating of Abdomen, Cycle 2 Day 15, Frequency, 2=Occasionally | 4 | 1
  Bloating of Abdomen, Cycle 2 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 13 | 14
  Bloating of Abdomen, Cycle 2 Day 15, Frequency, 3=Frequently | 1 | 4
  Bloating of Abdomen, Cycle 2 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 13 | 14
  Bloating of Abdomen, Cycle 2 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Bloating of Abdomen, Cycle 3 Day 1, Severity, 0=None: number analyzed (Participants) | 7 | 10
  Bloating of Abdomen, Cycle 3 Day 1, Severity, 0=None | 1 | 0
  Bloating of Abdomen, Cycle 3 Day 1, Severity, 1=Mild: number analyzed (Participants) | 7 | 10
  Bloating of Abdomen, Cycle 3 Day 1, Severity, 1=Mild | 4 | 6
  Bloating of Abdomen, Cycle 3 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 7 | 10
  Bloating of Abdomen, Cycle 3 Day 1, Severity, 2=Moderate | 2 | 3
  Bloating of Abdomen, Cycle 3 Day 1, Severity, 3=Severe: number analyzed (Participants) | 7 | 10
  Bloating of Abdomen, Cycle 3 Day 1, Severity, 3=Severe | 0 | 1
  Bloating of Abdomen, Cycle 3 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 7 | 10
  Bloating of Abdomen, Cycle 3 Day 1, Severity, 4=Very severe | 0 | 0
  Bloating of Abdomen, Cycle 3 Day 1, Frequency, 0=Never: number analyzed (Participants) | 14 | 14
  Bloating of Abdomen, Cycle 3 Day 1, Frequency, 0=Never | 7 | 4
  Bloating of Abdomen, Cycle 3 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 14
  Bloating of Abdomen, Cycle 3 Day 1, Frequency, 1=Rarely | 2 | 5
  Bloating of Abdomen, Cycle 3 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 14
  Bloating of Abdomen, Cycle 3 Day 1, Frequency, 2=Occasionally | 2 | 4
  Bloating of Abdomen, Cycle 3 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 14
  Bloating of Abdomen, Cycle 3 Day 1, Frequency, 3=Frequently | 3 | 1
  Bloating of Abdomen, Cycle 3 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 14
  Bloating of Abdomen, Cycle 3 Day 1, Frequency, 4=Almost constantly | 0 | 0
  Bloating of Abdomen, Cycle 3 Day 8, Severity, 0=None: number analyzed (Participants) | 6 | 9
  Bloating of Abdomen, Cycle 3 Day 8, Severity, 0=None | 1 | 0
  Bloating of Abdomen, Cycle 3 Day 8, Severity, 1=Mild: number analyzed (Participants) | 6 | 9
  Bloating of Abdomen, Cycle 3 Day 8, Severity, 1=Mild | 2 | 5
  Bloating of Abdomen, Cycle 3 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 6 | 9
  Bloating of Abdomen, Cycle 3 Day 8, Severity, 2=Moderate | 2 | 3
  Bloating of Abdomen, Cycle 3 Day 8, Severity, 3=Severe: number analyzed (Participants) | 6 | 9
  Bloating of Abdomen, Cycle 3 Day 8, Severity, 3=Severe | 1 | 1
  Bloating of Abdomen, Cycle 3 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 6 | 9
  Bloating of Abdomen, Cycle 3 Day 8, Severity, 4=Very severe | 0 | 0
  Bloating of Abdomen, Cycle 3 Day 8, Frequency, 0=Never: number analyzed (Participants) | 10 | 10
  Bloating of Abdomen, Cycle 3 Day 8, Frequency, 0=Never | 4 | 1
  Bloating of Abdomen, Cycle 3 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 10 | 10
  Bloating of Abdomen, Cycle 3 Day 8, Frequency, 1=Rarely | 2 | 4
  Bloating of Abdomen, Cycle 3 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 10 | 10
  Bloating of Abdomen, Cycle 3 Day 8, Frequency, 2=Occasionally | 3 | 3
  Bloating of Abdomen, Cycle 3 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 10 | 10
  Bloating of Abdomen, Cycle 3 Day 8, Frequency, 3=Frequently | 0 | 2
  Bloating of Abdomen, Cycle 3 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 10 | 10
  Bloating of Abdomen, Cycle 3 Day 8, Frequency, 4=Almost constantly | 1 | 0
  Bloating of Abdomen, Cycle 3 Day 15, Severity, 0=None: number analyzed (Participants) | 2 | 5
  Bloating of Abdomen, Cycle 3 Day 15, Severity, 0=None | 1 | 0
  Bloating of Abdomen, Cycle 3 Day 15, Severity, 1=Mild: number analyzed (Participants) | 2 | 5
  Bloating of Abdomen, Cycle 3 Day 15, Severity, 1=Mild | 1 | 3
  Bloating of Abdomen, Cycle 3 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 2 | 5
  Bloating of Abdomen, Cycle 3 Day 15, Severity, 2=Moderate | 0 | 2
  Bloating of Abdomen, Cycle 3 Day 15, Severity, 3=Severe: number analyzed (Participants) | 2 | 5
  Bloating of Abdomen, Cycle 3 Day 15, Severity, 3=Severe | 0 | 0
  Bloating of Abdomen, Cycle 3 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 2 | 5
  Bloating of Abdomen, Cycle 3 Day 15, Severity, 4=Very severe | 0 | 0
  Bloating of Abdomen, Cycle 3 Day 15, Frequency, 0=Never: number analyzed (Participants) | 5 | 7
  Bloating of Abdomen, Cycle 3 Day 15, Frequency, 0=Never | 3 | 2
  Bloating of Abdomen, Cycle 3 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 5 | 7
  Bloating of Abdomen, Cycle 3 Day 15, Frequency, 1=Rarely | 1 | 3
  Bloating of Abdomen, Cycle 3 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 5 | 7
  Bloating of Abdomen, Cycle 3 Day 15, Frequency, 2=Occasionally | 1 | 0
  Bloating of Abdomen, Cycle 3 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 5 | 7
  Bloating of Abdomen, Cycle 3 Day 15, Frequency, 3=Frequently | 0 | 2
  Bloating of Abdomen, Cycle 3 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 5 | 7
  Bloating of Abdomen, Cycle 3 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Bloating of Abdomen, Pre-IDS Evaluation, Frequency, 0=Never: number analyzed (Participants) | 2 | 1
  Bloating of Abdomen, Pre-IDS Evaluation, Frequency, 0=Never | 2 | 1
  Bloating of Abdomen, Pre-IDS Evaluation, Frequency, 1=Rarely: number analyzed (Participants) | 2 | 1
  Bloating of Abdomen, Pre-IDS Evaluation, Frequency, 1=Rarely | 0 | 0
  Bloating of Abdomen, Pre-IDS Evaluation, Frequency, 2=Occasionally: number analyzed (Participants) | 2 | 1
  Bloating of Abdomen, Pre-IDS Evaluation, Frequency, 2=Occasionally | 0 | 0
  Bloating of Abdomen, Pre-IDS Evaluation, Frequency, 3=Frequently: number analyzed (Participants) | 2 | 1
  Bloating of Abdomen, Pre-IDS Evaluation, Frequency, 3=Frequently | 0 | 0
  Bloating of Abdomen, Pre-IDS Evaluation, Frequency, 4=Almost constantly: number analyzed (Participants) | 2 | 1
  Bloating of Abdomen, Pre-IDS Evaluation, Frequency, 4=Almost constantly | 0 | 0
  Bloating of Abdomen, End Of Treatment, Severity, 0=None: number analyzed (Participants) | 0 | 4
  Bloating of Abdomen, End Of Treatment, Severity, 0=None |  | 0
  Bloating of Abdomen, End Of Treatment, Severity, 1=Mild: number analyzed (Participants) | 0 | 4
  Bloating of Abdomen, End Of Treatment, Severity, 1=Mild |  | 2
  Bloating of Abdomen, End Of Treatment, Severity, 2=Moderate: number analyzed (Participants) | 0 | 4
  Bloating of Abdomen, End Of Treatment, Severity, 2=Moderate |  | 1
  Bloating of Abdomen, End Of Treatment, Severity, 3=Severe: number analyzed (Participants) | 0 | 4
  Bloating of Abdomen, End Of Treatment, Severity, 3=Severe |  | 1
  Bloating of Abdomen, End Of Treatment, Severity, 4=Very severe: number analyzed (Participants) | 0 | 4
  Bloating of Abdomen, End Of Treatment, Severity, 4=Very severe |  | 0
  Bloating of Abdomen, End Of Treatment, Frequency, 0=Never: number analyzed (Participants) | 0 | 5
  Bloating of Abdomen, End Of Treatment, Frequency, 0=Never |  | 1
  Bloating of Abdomen, End Of Treatment, Frequency, 1=Rarely: number analyzed (Participants) | 0 | 5
  Bloating of Abdomen, End Of Treatment, Frequency, 1=Rarely |  | 1
  Bloating of Abdomen, End Of Treatment, Frequency, 2=Occasionally: number analyzed (Participants) | 0 | 5
  Bloating of Abdomen, End Of Treatment, Frequency, 2=Occasionally |  | 1
  Bloating of Abdomen, End Of Treatment, Frequency, 3=Frequently: number analyzed (Participants) | 0 | 5
  Bloating of Abdomen, End Of Treatment, Frequency, 3=Frequently |  | 1
  Bloating of Abdomen, End Of Treatment, Frequency, 4=Almost constantly: number analyzed (Participants) | 0 | 5
  Bloating of Abdomen, End Of Treatment, Frequency, 4=Almost constantly |  | 1
  Constipation, Baseline, Severity, 0=None: number analyzed (Participants) | 14 | 17
  Constipation, Baseline, Severity, 0=None | 8 | 9
  Constipation, Baseline, Severity, 1=Mild: number analyzed (Participants) | 14 | 17
  Constipation, Baseline, Severity, 1=Mild | 3 | 6
  Constipation, Baseline, Severity, 2=Moderate: number analyzed (Participants) | 14 | 17
  Constipation, Baseline, Severity, 2=Moderate | 1 | 2
  Constipation, Baseline, Severity, 3=Severe: number analyzed (Participants) | 14 | 17
  Constipation, Baseline, Severity, 3=Severe | 1 | 0
  Constipation, Baseline, Severity, 4=Very severe: number analyzed (Participants) | 14 | 17
  Constipation, Baseline, Severity, 4=Very severe | 1 | 0
  Constipation, Cycle 1 Day 8, Severity, 0=None: number analyzed (Participants) | 11 | 15
  Constipation, Cycle 1 Day 8, Severity, 0=None | 5 | 8
  Constipation, Cycle 1 Day 8, Severity, 1=Mild: number analyzed (Participants) | 11 | 15
  Constipation, Cycle 1 Day 8, Severity, 1=Mild | 0 | 2
  Constipation, Cycle 1 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 11 | 15
  Constipation, Cycle 1 Day 8, Severity, 2=Moderate | 3 | 2
  Constipation, Cycle 1 Day 8, Severity, 3=Severe: number analyzed (Participants) | 11 | 15
  Constipation, Cycle 1 Day 8, Severity, 3=Severe | 3 | 3
  Constipation, Cycle 1 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 11 | 15
  Constipation, Cycle 1 Day 8, Severity, 4=Very severe | 0 | 0
  Constipation, Cycle 1 Day 15, Severity, 0=None: number analyzed (Participants) | 14 | 13
  Constipation, Cycle 1 Day 15, Severity, 0=None | 10 | 6
  Constipation, Cycle 1 Day 15, Severity, 1=Mild: number analyzed (Participants) | 14 | 13
  Constipation, Cycle 1 Day 15, Severity, 1=Mild | 4 | 4
  Constipation, Cycle 1 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 14 | 13
  Constipation, Cycle 1 Day 15, Severity, 2=Moderate | 0 | 1
  Constipation, Cycle 1 Day 15, Severity, 3=Severe: number analyzed (Participants) | 14 | 13
  Constipation, Cycle 1 Day 15, Severity, 3=Severe | 0 | 1
  Constipation, Cycle 1 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 14 | 13
  Constipation, Cycle 1 Day 15, Severity, 4=Very severe | 0 | 1
  Constipation, Cycle 2 Day 1, Severity, 0=None: number analyzed (Participants) | 11 | 14
  Constipation, Cycle 2 Day 1, Severity, 0=None | 8 | 6
  Constipation, Cycle 2 Day 1, Severity, 1=Mild: number analyzed (Participants) | 11 | 14
  Constipation, Cycle 2 Day 1, Severity, 1=Mild | 2 | 5
  Constipation, Cycle 2 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 11 | 14
  Constipation, Cycle 2 Day 1, Severity, 2=Moderate | 1 | 2
  Constipation, Cycle 2 Day 1, Severity, 3=Severe: number analyzed (Participants) | 11 | 14
  Constipation, Cycle 2 Day 1, Severity, 3=Severe | 0 | 0
  Constipation, Cycle 2 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 11 | 14
  Constipation, Cycle 2 Day 1, Severity, 4=Very severe | 0 | 1
  Constipation, Cycle 2 Day 8, Severity, 0=None: number analyzed (Participants) | 11 | 11
  Constipation, Cycle 2 Day 8, Severity, 0=None | 6 | 5
  Constipation, Cycle 2 Day 8, Severity, 1=Mild: number analyzed (Participants) | 11 | 11
  Constipation, Cycle 2 Day 8, Severity, 1=Mild | 2 | 4
  Constipation, Cycle 2 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 11 | 11
  Constipation, Cycle 2 Day 8, Severity, 2=Moderate | 2 | 2
  Constipation, Cycle 2 Day 8, Severity, 3=Severe: number analyzed (Participants) | 11 | 11
  Constipation, Cycle 2 Day 8, Severity, 3=Severe | 1 | 0
  Constipation, Cycle 2 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 11 | 11
  Constipation, Cycle 2 Day 8, Severity, 4=Very severe | 0 | 0
  Constipation, Cycle 2 Day 15, Severity, 0=None: number analyzed (Participants) | 13 | 14
  Constipation, Cycle 2 Day 15, Severity, 0=None | 10 | 8
  Constipation, Cycle 2 Day 15, Severity, 1=Mild: number analyzed (Participants) | 13 | 14
  Constipation, Cycle 2 Day 15, Severity, 1=Mild | 3 | 2
  Constipation, Cycle 2 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 13 | 14
  Constipation, Cycle 2 Day 15, Severity, 2=Moderate | 0 | 3
  Constipation, Cycle 2 Day 15, Severity, 3=Severe: number analyzed (Participants) | 13 | 14
  Constipation, Cycle 2 Day 15, Severity, 3=Severe | 0 | 1
  Constipation, Cycle 2 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 13 | 14
  Constipation, Cycle 2 Day 15, Severity, 4=Very severe | 0 | 0
  Constipation, Cycle 3 Day 1, Severity, 0=None: number analyzed (Participants) | 14 | 14
  Constipation, Cycle 3 Day 1, Severity, 0=None | 11 | 6
  Constipation, Cycle 3 Day 1, Severity, 1=Mild: number analyzed (Participants) | 14 | 14
  Constipation, Cycle 3 Day 1, Severity, 1=Mild | 2 | 1
  Constipation, Cycle 3 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 14 | 14
  Constipation, Cycle 3 Day 1, Severity, 2=Moderate | 1 | 5
  Constipation, Cycle 3 Day 1, Severity, 3=Severe: number analyzed (Participants) | 14 | 14
  Constipation, Cycle 3 Day 1, Severity, 3=Severe | 0 | 1
  Constipation, Cycle 3 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 14 | 14
  Constipation, Cycle 3 Day 1, Severity, 4=Very severe | 0 | 1
  Constipation, Cycle 3 Day 8, Severity, 0=None: number analyzed (Participants) | 10 | 10
  Constipation, Cycle 3 Day 8, Severity, 0=None | 4 | 4
  Constipation, Cycle 3 Day 8, Severity, 1=Mild: number analyzed (Participants) | 10 | 10
  Constipation, Cycle 3 Day 8, Severity, 1=Mild | 5 | 2
  Constipation, Cycle 3 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 10 | 10
  Constipation, Cycle 3 Day 8, Severity, 2=Moderate | 1 | 2
  Constipation, Cycle 3 Day 8, Severity, 3=Severe: number analyzed (Participants) | 10 | 10
  Constipation, Cycle 3 Day 8, Severity, 3=Severe | 0 | 2
  Constipation, Cycle 3 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 10 | 10
  Constipation, Cycle 3 Day 8, Severity, 4=Very severe | 0 | 0
  Constipation, Cycle 3 Day 15, Severity, 0=None: number analyzed (Participants) | 5 | 7
  Constipation, Cycle 3 Day 15, Severity, 0=None | 4 | 3
  Constipation, Cycle 3 Day 15, Severity, 1=Mild: number analyzed (Participants) | 5 | 7
  Constipation, Cycle 3 Day 15, Severity, 1=Mild | 1 | 3
  Constipation, Cycle 3 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 5 | 7
  Constipation, Cycle 3 Day 15, Severity, 2=Moderate | 0 | 1
  Constipation, Cycle 3 Day 15, Severity, 3=Severe: number analyzed (Participants) | 5 | 7
  Constipation, Cycle 3 Day 15, Severity, 3=Severe | 0 | 0
  Constipation, Cycle 3 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 5 | 7
  Constipation, Cycle 3 Day 15, Severity, 4=Very severe | 0 | 0
  Constipation, Pre-IDS Evaluation, Severity, 0=None: number analyzed (Participants) | 2 | 1
  Constipation, Pre-IDS Evaluation, Severity, 0=None | 2 | 0
  Constipation, Pre-IDS Evaluation, Severity, 1=Mild: number analyzed (Participants) | 2 | 1
  Constipation, Pre-IDS Evaluation, Severity, 1=Mild | 0 | 0
  Constipation, Pre-IDS Evaluation, Severity, 2=Moderate: number analyzed (Participants) | 2 | 1
  Constipation, Pre-IDS Evaluation, Severity, 2=Moderate | 0 | 0
  Constipation, Pre-IDS Evaluation, Severity, 3=Severe: number analyzed (Participants) | 2 | 1
  Constipation, Pre-IDS Evaluation, Severity, 3=Severe | 0 | 0
  Constipation, Pre-IDS Evaluation, Severity, 4=Very severe: number analyzed (Participants) | 2 | 1
  Constipation, Pre-IDS Evaluation, Severity, 4=Very severe | 0 | 1
  Constipation, End Of Treatment, Severity, 0=None: number analyzed (Participants) | 0 | 5
  Constipation, End Of Treatment, Severity, 0=None |  | 2
  Constipation, End Of Treatment, Severity, 1=Mild: number analyzed (Participants) | 0 | 5
  Constipation, End Of Treatment, Severity, 1=Mild |  | 3
  Constipation, End Of Treatment, Severity, 2=Moderate: number analyzed (Participants) | 0 | 5
  Constipation, End Of Treatment, Severity, 2=Moderate |  | 0
  Constipation, End Of Treatment, Severity, 3=Severe: number analyzed (Participants) | 0 | 5
  Constipation, End Of Treatment, Severity, 3=Severe |  | 0
  Constipation, End Of Treatment, Severity, 4=Very severe: number analyzed (Participants) | 0 | 5
  Constipation, End Of Treatment, Severity, 4=Very severe |  | 0
  Loose/Watery Stools, Baseline, Frequency, 0=Never: number analyzed (Participants) | 14 | 17
  Loose/Watery Stools, Baseline, Frequency, 0=Never | 8 | 10
  Loose/Watery Stools, Baseline, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 17
  Loose/Watery Stools, Baseline, Frequency, 1=Rarely | 2 | 5
  Loose/Watery Stools, Baseline, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 17
  Loose/Watery Stools, Baseline, Frequency, 2=Occasionally | 4 | 1
  Loose/Watery Stools, Baseline, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 17
  Loose/Watery Stools, Baseline, Frequency, 3=Frequently | 0 | 1
  Loose/Watery Stools, Baseline, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 17
  Loose/Watery Stools, Baseline, Frequency, 4=Almost constantly | 0 | 0
  Loose/Watery Stools, Cycle 1 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 15
  Loose/Watery Stools, Cycle 1 Day 8, Frequency, 0=Never | 8 | 11
  Loose/Watery Stools, Cycle 1 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 15
  Loose/Watery Stools, Cycle 1 Day 8, Frequency, 1=Rarely | 1 | 3
  Loose/Watery Stools, Cycle 1 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 15
  Loose/Watery Stools, Cycle 1 Day 8, Frequency, 2=Occasionally | 2 | 1
  Loose/Watery Stools, Cycle 1 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 15
  Loose/Watery Stools, Cycle 1 Day 8, Frequency, 3=Frequently | 0 | 0
  Loose/Watery Stools, Cycle 1 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 15
  Loose/Watery Stools, Cycle 1 Day 8, Frequency, 4=Almost constantly | 0 | 0
  Loose/Watery Stools, Cycle 1 Day 15, Frequency, 0=Never: number analyzed (Participants) | 14 | 13
  Loose/Watery Stools, Cycle 1 Day 15, Frequency, 0=Never | 11 | 10
  Loose/Watery Stools, Cycle 1 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 13
  Loose/Watery Stools, Cycle 1 Day 15, Frequency, 1=Rarely | 2 | 2
  Loose/Watery Stools, Cycle 1 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 13
  Loose/Watery Stools, Cycle 1 Day 15, Frequency, 2=Occasionally | 1 | 1
  Loose/Watery Stools, Cycle 1 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 13
  Loose/Watery Stools, Cycle 1 Day 15, Frequency, 3=Frequently | 0 | 0
  Loose/Watery Stools, Cycle 1 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 13
  Loose/Watery Stools, Cycle 1 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Loose/Watery Stools, Cycle 2 Day 1, Frequency, 0=Never: number analyzed (Participants) | 11 | 14
  Loose/Watery Stools, Cycle 2 Day 1, Frequency, 0=Never | 9 | 12
  Loose/Watery Stools, Cycle 2 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 14
  Loose/Watery Stools, Cycle 2 Day 1, Frequency, 1=Rarely | 0 | 1
  Loose/Watery Stools, Cycle 2 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 14
  Loose/Watery Stools, Cycle 2 Day 1, Frequency, 2=Occasionally | 1 | 0
  Loose/Watery Stools, Cycle 2 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 14
  Loose/Watery Stools, Cycle 2 Day 1, Frequency, 3=Frequently | 1 | 1
  Loose/Watery Stools, Cycle 2 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 14
  Loose/Watery Stools, Cycle 2 Day 1, Frequency, 4=Almost constantly | 0 | 0
  Loose/Watery Stools, Cycle 2 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 11
  Loose/Watery Stools, Cycle 2 Day 8, Frequency, 0=Never | 7 | 9
  Loose/Watery Stools, Cycle 2 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 11
  Loose/Watery Stools, Cycle 2 Day 8, Frequency, 1=Rarely | 2 | 2
  Loose/Watery Stools, Cycle 2 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 11
  Loose/Watery Stools, Cycle 2 Day 8, Frequency, 2=Occasionally | 2 | 0
  Loose/Watery Stools, Cycle 2 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 11
  Loose/Watery Stools, Cycle 2 Day 8, Frequency, 3=Frequently | 0 | 0
  Loose/Watery Stools, Cycle 2 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 11
  Loose/Watery Stools, Cycle 2 Day 8, Frequency, 4=Almost constantly | 0 | 0
  Loose/Watery Stools, Cycle 2 Day 15, Frequency, 0=Never: number analyzed (Participants) | 13 | 14
  Loose/Watery Stools, Cycle 2 Day 15, Frequency, 0=Never | 8 | 12
  Loose/Watery Stools, Cycle 2 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 13 | 14
  Loose/Watery Stools, Cycle 2 Day 15, Frequency, 1=Rarely | 1 | 1
  Loose/Watery Stools, Cycle 2 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 13 | 14
  Loose/Watery Stools, Cycle 2 Day 15, Frequency, 2=Occasionally | 3 | 1
  Loose/Watery Stools, Cycle 2 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 13 | 14
  Loose/Watery Stools, Cycle 2 Day 15, Frequency, 3=Frequently | 1 | 0
  Loose/Watery Stools, Cycle 2 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 13 | 14
  Loose/Watery Stools, Cycle 2 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Loose/Watery Stools, Cycle 3 Day 1, Frequency, 0=Never: number analyzed (Participants) | 14 | 14
  Loose/Watery Stools, Cycle 3 Day 1, Frequency, 0=Never | 8 | 12
  Loose/Watery Stools, Cycle 3 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 14
  Loose/Watery Stools, Cycle 3 Day 1, Frequency, 1=Rarely | 4 | 1
  Loose/Watery Stools, Cycle 3 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 14
  Loose/Watery Stools, Cycle 3 Day 1, Frequency, 2=Occasionally | 0 | 1
  Loose/Watery Stools, Cycle 3 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 14
  Loose/Watery Stools, Cycle 3 Day 1, Frequency, 3=Frequently | 1 | 0
  Loose/Watery Stools, Cycle 3 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 14
  Loose/Watery Stools, Cycle 3 Day 1, Frequency, 4=Almost constantly | 1 | 0
  Loose/Watery Stools, Cycle 3 Day 8, Frequency, 0=Never: number analyzed (Participants) | 10 | 10
  Loose/Watery Stools, Cycle 3 Day 8, Frequency, 0=Never | 7 | 8
  Loose/Watery Stools, Cycle 3 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 10 | 10
  Loose/Watery Stools, Cycle 3 Day 8, Frequency, 1=Rarely | 0 | 1
  Loose/Watery Stools, Cycle 3 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 10 | 10
  Loose/Watery Stools, Cycle 3 Day 8, Frequency, 2=Occasionally | 0 | 0
  Loose/Watery Stools, Cycle 3 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 10 | 10
  Loose/Watery Stools, Cycle 3 Day 8, Frequency, 3=Frequently | 2 | 1
  Loose/Watery Stools, Cycle 3 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 10 | 10
  Loose/Watery Stools, Cycle 3 Day 8, Frequency, 4=Almost constantly | 1 | 0
  Loose/Watery Stools, Cycle 3 Day 15, Frequency, 0=Never: number analyzed (Participants) | 5 | 7
  Loose/Watery Stools, Cycle 3 Day 15, Frequency, 0=Never | 1 | 5
  Loose/Watery Stools, Cycle 3 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 5 | 7
  Loose/Watery Stools, Cycle 3 Day 15, Frequency, 1=Rarely | 2 | 2
  Loose/Watery Stools, Cycle 3 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 5 | 7
  Loose/Watery Stools, Cycle 3 Day 15, Frequency, 2=Occasionally | 2 | 0
  Loose/Watery Stools, Cycle 3 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 5 | 7
  Loose/Watery Stools, Cycle 3 Day 15, Frequency, 3=Frequently | 0 | 0
  Loose/Watery Stools, Cycle 3 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 5 | 7
  Loose/Watery Stools, Cycle 3 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Loose/Watery Stools, Pre-IDS Evaluation, Frequency, 0=Never: number analyzed (Participants) | 2 | 1
  Loose/Watery Stools, Pre-IDS Evaluation, Frequency, 0=Never | 2 | 1
  Loose/Watery Stools, Pre-IDS Evaluation, Frequency, 1=Rarely: number analyzed (Participants) | 2 | 1
  Loose/Watery Stools, Pre-IDS Evaluation, Frequency, 1=Rarely | 0 | 0
  Loose/Watery Stools, Pre-IDS Evaluation, Frequency, 2=Occasionally: number analyzed (Participants) | 2 | 1
  Loose/Watery Stools, Pre-IDS Evaluation, Frequency, 2=Occasionally | 0 | 0
  Loose/Watery Stools, Pre-IDS Evaluation, Frequency, 3=Frequently: number analyzed (Participants) | 2 | 1
  Loose/Watery Stools, Pre-IDS Evaluation, Frequency, 3=Frequently | 0 | 0
  Loose/Watery Stools, Pre-IDS Evaluation, Frequency, 4=Almost constantly: number analyzed (Participants) | 2 | 1
  Loose/Watery Stools, Pre-IDS Evaluation, Frequency, 4=Almost constantly | 0 | 0
  Loose/Watery Stools, End Of Treatment, Frequency, 0=Never: number analyzed (Participants) | 0 | 5
  Loose/Watery Stools, End Of Treatment, Frequency, 0=Never |  | 3
  Loose/Watery Stools, End Of Treatment, Frequency, 1=Rarely: number analyzed (Participants) | 0 | 5
  Loose/Watery Stools, End Of Treatment, Frequency, 1=Rarely |  | 1
  Loose/Watery Stools, End Of Treatment, Frequency, 2=Occasionally: number analyzed (Participants) | 0 | 5
  Loose/Watery Stools, End Of Treatment, Frequency, 2=Occasionally |  | 1
  Loose/Watery Stools, End Of Treatment, Frequency, 3=Frequently: number analyzed (Participants) | 0 | 5
  Loose/Watery Stools, End Of Treatment, Frequency, 3=Frequently |  | 0
  Loose/Watery Stools, End Of Treatment, Frequency, 4=Almost constantly: number analyzed (Participants) | 0 | 5
  Loose/Watery Stools, End Of Treatment, Frequency, 4=Almost constantly |  | 0
  Pain in the Abdomen, Baseline, Severity, 0=None: number analyzed (Participants) | 12 | 11
  Pain in the Abdomen, Baseline, Severity, 0=None | 0 | 1
  Pain in the Abdomen, Baseline, Severity, 1=Mild: number analyzed (Participants) | 12 | 11
  Pain in the Abdomen, Baseline, Severity, 1=Mild | 6 | 5
  Pain in the Abdomen, Baseline, Severity, 2=Moderate: number analyzed (Participants) | 12 | 11
  Pain in the Abdomen, Baseline, Severity, 2=Moderate | 6 | 4
  Pain in the Abdomen, Baseline, Severity, 3=Severe: number analyzed (Participants) | 12 | 11
  Pain in the Abdomen, Baseline, Severity, 3=Severe | 0 | 1
  Pain in the Abdomen, Baseline, Severity, 4=Very severe: number analyzed (Participants) | 12 | 11
  Pain in the Abdomen, Baseline, Severity, 4=Very severe | 0 | 0
  Pain in the Abdomen, Baseline, Frequency, 0=Never: number analyzed (Participants) | 14 | 17
  Pain in the Abdomen, Baseline, Frequency, 0=Never | 2 | 6
  Pain in the Abdomen, Baseline, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 17
  Pain in the Abdomen, Baseline, Frequency, 1=Rarely | 6 | 5
  Pain in the Abdomen, Baseline, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 17
  Pain in the Abdomen, Baseline, Frequency, 2=Occasionally | 3 | 4
  Pain in the Abdomen, Baseline, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 17
  Pain in the Abdomen, Baseline, Frequency, 3=Frequently | 2 | 2
  Pain in the Abdomen, Baseline, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 17
  Pain in the Abdomen, Baseline, Frequency, 4=Almost constantly | 1 | 0
  Pain in the Abdomen, Cycle 1 Day 8, Severity, 0=None: number analyzed (Participants) | 10 | 9
  Pain in the Abdomen, Cycle 1 Day 8, Severity, 0=None | 0 | 0
  Pain in the Abdomen, Cycle 1 Day 8, Severity, 1=Mild: number analyzed (Participants) | 10 | 9
  Pain in the Abdomen, Cycle 1 Day 8, Severity, 1=Mild | 4 | 2
  Pain in the Abdomen, Cycle 1 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 10 | 9
  Pain in the Abdomen, Cycle 1 Day 8, Severity, 2=Moderate | 4 | 5
  Pain in the Abdomen, Cycle 1 Day 8, Severity, 3=Severe: number analyzed (Participants) | 10 | 9
  Pain in the Abdomen, Cycle 1 Day 8, Severity, 3=Severe | 1 | 2
  Pain in the Abdomen, Cycle 1 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 10 | 9
  Pain in the Abdomen, Cycle 1 Day 8, Severity, 4=Very severe | 1 | 0
  Pain in the Abdomen, Cycle 1 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 15
  Pain in the Abdomen, Cycle 1 Day 8, Frequency, 0=Never | 1 | 6
  Pain in the Abdomen, Cycle 1 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 15
  Pain in the Abdomen, Cycle 1 Day 8, Frequency, 1=Rarely | 3 | 1
  Pain in the Abdomen, Cycle 1 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 15
  Pain in the Abdomen, Cycle 1 Day 8, Frequency, 2=Occasionally | 3 | 5
  Pain in the Abdomen, Cycle 1 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 15
  Pain in the Abdomen, Cycle 1 Day 8, Frequency, 3=Frequently | 3 | 2
  Pain in the Abdomen, Cycle 1 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 15
  Pain in the Abdomen, Cycle 1 Day 8, Frequency, 4=Almost constantly | 1 | 1
  Pain in the Abdomen, Cycle 1 Day 15, Severity, 0=None: number analyzed (Participants) | 11 | 9
  Pain in the Abdomen, Cycle 1 Day 15, Severity, 0=None | 0 | 0
  Pain in the Abdomen, Cycle 1 Day 15, Severity, 1=Mild: number analyzed (Participants) | 11 | 9
  Pain in the Abdomen, Cycle 1 Day 15, Severity, 1=Mild | 8 | 4
  Pain in the Abdomen, Cycle 1 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 11 | 9
  Pain in the Abdomen, Cycle 1 Day 15, Severity, 2=Moderate | 2 | 4
  Pain in the Abdomen, Cycle 1 Day 15, Severity, 3=Severe: number analyzed (Participants) | 11 | 9
  Pain in the Abdomen, Cycle 1 Day 15, Severity, 3=Severe | 1 | 1
  Pain in the Abdomen, Cycle 1 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 11 | 9
  Pain in the Abdomen, Cycle 1 Day 15, Severity, 4=Very severe | 0 | 0
  Pain in the Abdomen, Cycle 1 Day 15, Frequency, 0=Never: number analyzed (Participants) | 14 | 13
  Pain in the Abdomen, Cycle 1 Day 15, Frequency, 0=Never | 3 | 4
  Pain in the Abdomen, Cycle 1 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 13
  Pain in the Abdomen, Cycle 1 Day 15, Frequency, 1=Rarely | 6 | 2
  Pain in the Abdomen, Cycle 1 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 13
  Pain in the Abdomen, Cycle 1 Day 15, Frequency, 2=Occasionally | 4 | 5
  Pain in the Abdomen, Cycle 1 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 13
  Pain in the Abdomen, Cycle 1 Day 15, Frequency, 3=Frequently | 1 | 1
  Pain in the Abdomen, Cycle 1 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 13
  Pain in the Abdomen, Cycle 1 Day 15, Frequency, 4=Almost constantly | 0 | 1
  Pain in the Abdomen, Cycle 2 Day 1, Severity, 0=None: number analyzed (Participants) | 7 | 5
  Pain in the Abdomen, Cycle 2 Day 1, Severity, 0=None | 0 | 0
  Pain in the Abdomen, Cycle 2 Day 1, Severity, 1=Mild: number analyzed (Participants) | 7 | 5
  Pain in the Abdomen, Cycle 2 Day 1, Severity, 1=Mild | 4 | 1
  Pain in the Abdomen, Cycle 2 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 7 | 5
  Pain in the Abdomen, Cycle 2 Day 1, Severity, 2=Moderate | 3 | 3
  Pain in the Abdomen, Cycle 2 Day 1, Severity, 3=Severe: number analyzed (Participants) | 7 | 5
  Pain in the Abdomen, Cycle 2 Day 1, Severity, 3=Severe | 0 | 1
  Pain in the Abdomen, Cycle 2 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 7 | 5
  Pain in the Abdomen, Cycle 2 Day 1, Severity, 4=Very severe | 0 | 0
  Pain in the Abdomen, Cycle 2 Day 1, Frequency, 0=Never: number analyzed (Participants) | 11 | 14
  Pain in the Abdomen, Cycle 2 Day 1, Frequency, 0=Never | 4 | 9
  Pain in the Abdomen, Cycle 2 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 14
  Pain in the Abdomen, Cycle 2 Day 1, Frequency, 1=Rarely | 4 | 1
  Pain in the Abdomen, Cycle 2 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 14
  Pain in the Abdomen, Cycle 2 Day 1, Frequency, 2=Occasionally | 3 | 4
  Pain in the Abdomen, Cycle 2 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 14
  Pain in the Abdomen, Cycle 2 Day 1, Frequency, 3=Frequently | 0 | 0
  Pain in the Abdomen, Cycle 2 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 14
  Pain in the Abdomen, Cycle 2 Day 1, Frequency, 4=Almost constantly | 0 | 0
  Pain in the Abdomen, Cycle 2 Day 8, Severity, 0=None: number analyzed (Participants) | 7 | 5
  Pain in the Abdomen, Cycle 2 Day 8, Severity, 0=None | 1 | 0
  Pain in the Abdomen, Cycle 2 Day 8, Severity, 1=Mild: number analyzed (Participants) | 7 | 5
  Pain in the Abdomen, Cycle 2 Day 8, Severity, 1=Mild | 2 | 2
  Pain in the Abdomen, Cycle 2 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 7 | 5
  Pain in the Abdomen, Cycle 2 Day 8, Severity, 2=Moderate | 3 | 3
  Pain in the Abdomen, Cycle 2 Day 8, Severity, 3=Severe: number analyzed (Participants) | 7 | 5
  Pain in the Abdomen, Cycle 2 Day 8, Severity, 3=Severe | 1 | 0
  Pain in the Abdomen, Cycle 2 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 7 | 5
  Pain in the Abdomen, Cycle 2 Day 8, Severity, 4=Very severe | 0 | 0
  Pain in the Abdomen, Cycle 2 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 11
  Pain in the Abdomen, Cycle 2 Day 8, Frequency, 0=Never | 4 | 6
  Pain in the Abdomen, Cycle 2 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 11
  Pain in the Abdomen, Cycle 2 Day 8, Frequency, 1=Rarely | 1 | 2
  Pain in the Abdomen, Cycle 2 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 11
  Pain in the Abdomen, Cycle 2 Day 8, Frequency, 2=Occasionally | 4 | 3
  Pain in the Abdomen, Cycle 2 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 11
  Pain in the Abdomen, Cycle 2 Day 8, Frequency, 3=Frequently | 1 | 0
  Pain in the Abdomen, Cycle 2 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 11
  Pain in the Abdomen, Cycle 2 Day 8, Frequency, 4=Almost constantly | 1 | 0
  Pain in the Abdomen, Cycle 2 Day 15, Severity, 0=None: number analyzed (Participants) | 7 | 9
  Pain in the Abdomen, Cycle 2 Day 15, Severity, 0=None | 0 | 0
  Pain in the Abdomen, Cycle 2 Day 15, Severity, 1=Mild: number analyzed (Participants) | 7 | 9
  Pain in the Abdomen, Cycle 2 Day 15, Severity, 1=Mild | 7 | 5
  Pain in the Abdomen, Cycle 2 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 7 | 9
  Pain in the Abdomen, Cycle 2 Day 15, Severity, 2=Moderate | 0 | 3
  Pain in the Abdomen, Cycle 2 Day 15, Severity, 3=Severe: number analyzed (Participants) | 7 | 9
  Pain in the Abdomen, Cycle 2 Day 15, Severity, 3=Severe | 0 | 1
  Pain in the Abdomen, Cycle 2 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 7 | 9
  Pain in the Abdomen, Cycle 2 Day 15, Severity, 4=Very severe | 0 | 0
  Pain in the Abdomen, Cycle 2 Day 15, Frequency, 0=Never: number analyzed (Participants) | 13 | 14
  Pain in the Abdomen, Cycle 2 Day 15, Frequency, 0=Never | 6 | 5
  Pain in the Abdomen, Cycle 2 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 13 | 14
  Pain in the Abdomen, Cycle 2 Day 15, Frequency, 1=Rarely | 1 | 5
  Pain in the Abdomen, Cycle 2 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 13 | 14
  Pain in the Abdomen, Cycle 2 Day 15, Frequency, 2=Occasionally | 6 | 3
  Pain in the Abdomen, Cycle 2 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 13 | 14
  Pain in the Abdomen, Cycle 2 Day 15, Frequency, 3=Frequently | 0 | 1
  Pain in the Abdomen, Cycle 2 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 13 | 14
  Pain in the Abdomen, Cycle 2 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Pain in the Abdomen, Cycle 3 Day 1, Severity, 0=None: number analyzed (Participants) | 8 | 8
  Pain in the Abdomen, Cycle 3 Day 1, Severity, 0=None | 1 | 0
  Pain in the Abdomen, Cycle 3 Day 1, Severity, 1=Mild: number analyzed (Participants) | 8 | 8
  Pain in the Abdomen, Cycle 3 Day 1, Severity, 1=Mild | 4 | 6
  Pain in the Abdomen, Cycle 3 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 8 | 8
  Pain in the Abdomen, Cycle 3 Day 1, Severity, 2=Moderate | 2 | 1
  Pain in the Abdomen, Cycle 3 Day 1, Severity, 3=Severe: number analyzed (Participants) | 8 | 8
  Pain in the Abdomen, Cycle 3 Day 1, Severity, 3=Severe | 1 | 1
  Pain in the Abdomen, Cycle 3 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 8 | 8
  Pain in the Abdomen, Cycle 3 Day 1, Severity, 4=Very severe | 0 | 0
  Pain in the Abdomen, Cycle 3 Day 1, Frequency, 0=Never: number analyzed (Participants) | 14 | 14
  Pain in the Abdomen, Cycle 3 Day 1, Frequency, 0=Never | 6 | 6
  Pain in the Abdomen, Cycle 3 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 14
  Pain in the Abdomen, Cycle 3 Day 1, Frequency, 1=Rarely | 3 | 3
  Pain in the Abdomen, Cycle 3 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 14
  Pain in the Abdomen, Cycle 3 Day 1, Frequency, 2=Occasionally | 3 | 4
  Pain in the Abdomen, Cycle 3 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 14
  Pain in the Abdomen, Cycle 3 Day 1, Frequency, 3=Frequently | 1 | 1
  Pain in the Abdomen, Cycle 3 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 14
  Pain in the Abdomen, Cycle 3 Day 1, Frequency, 4=Almost constantly | 1 | 0
  Pain in the Abdomen, Cycle 3 Day 8, Severity, 0=None: number analyzed (Participants) | 8 | 7
  Pain in the Abdomen, Cycle 3 Day 8, Severity, 0=None | 0 | 0
  Pain in the Abdomen, Cycle 3 Day 8, Severity, 1=Mild: number analyzed (Participants) | 8 | 7
  Pain in the Abdomen, Cycle 3 Day 8, Severity, 1=Mild | 4 | 3
  Pain in the Abdomen, Cycle 3 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 8 | 7
  Pain in the Abdomen, Cycle 3 Day 8, Severity, 2=Moderate | 2 | 3
  Pain in the Abdomen, Cycle 3 Day 8, Severity, 3=Severe: number analyzed (Participants) | 8 | 7
  Pain in the Abdomen, Cycle 3 Day 8, Severity, 3=Severe | 2 | 1
  Pain in the Abdomen, Cycle 3 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 8 | 7
  Pain in the Abdomen, Cycle 3 Day 8, Severity, 4=Very severe | 0 | 0
  Pain in the Abdomen, Cycle 3 Day 8, Frequency, 0=Never: number analyzed (Participants) | 10 | 10
  Pain in the Abdomen, Cycle 3 Day 8, Frequency, 0=Never | 2 | 3
  Pain in the Abdomen, Cycle 3 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 10 | 10
  Pain in the Abdomen, Cycle 3 Day 8, Frequency, 1=Rarely | 3 | 3
  Pain in the Abdomen, Cycle 3 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 10 | 10
  Pain in the Abdomen, Cycle 3 Day 8, Frequency, 2=Occasionally | 2 | 2
  Pain in the Abdomen, Cycle 3 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 10 | 10
  Pain in the Abdomen, Cycle 3 Day 8, Frequency, 3=Frequently | 3 | 2
  Pain in the Abdomen, Cycle 3 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 10 | 10
  Pain in the Abdomen, Cycle 3 Day 8, Frequency, 4=Almost constantly | 0 | 0
  Pain in the Abdomen, Cycle 3 Day 15, Severity, 0=None: number analyzed (Participants) | 5 | 4
  Pain in the Abdomen, Cycle 3 Day 15, Severity, 0=None | 2 | 0
  Pain in the Abdomen, Cycle 3 Day 15, Severity, 1=Mild: number analyzed (Participants) | 5 | 4
  Pain in the Abdomen, Cycle 3 Day 15, Severity, 1=Mild | 2 | 3
  Pain in the Abdomen, Cycle 3 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 5 | 4
  Pain in the Abdomen, Cycle 3 Day 15, Severity, 2=Moderate | 1 | 1
  Pain in the Abdomen, Cycle 3 Day 15, Severity, 3=Severe: number analyzed (Participants) | 5 | 4
  Pain in the Abdomen, Cycle 3 Day 15, Severity, 3=Severe | 0 | 0
  Pain in the Abdomen, Cycle 3 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 5 | 4
  Pain in the Abdomen, Cycle 3 Day 15, Severity, 4=Very severe | 0 | 0
  Pain in the Abdomen, Cycle 3 Day 15, Frequency, 0=Never: number analyzed (Participants) | 5 | 7
  Pain in the Abdomen, Cycle 3 Day 15, Frequency, 0=Never | 0 | 3
  Pain in the Abdomen, Cycle 3 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 5 | 7
  Pain in the Abdomen, Cycle 3 Day 15, Frequency, 1=Rarely | 2 | 1
  Pain in the Abdomen, Cycle 3 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 5 | 7
  Pain in the Abdomen, Cycle 3 Day 15, Frequency, 2=Occasionally | 3 | 2
  Pain in the Abdomen, Cycle 3 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 5 | 7
  Pain in the Abdomen, Cycle 3 Day 15, Frequency, 3=Frequently | 0 | 1
  Pain in the Abdomen, Cycle 3 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 5 | 7
  Pain in the Abdomen, Cycle 3 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Pain in the Abdomen, Pre-IDS Evaluation, Frequency, 0=Never: number analyzed (Participants) | 2 | 1
  Pain in the Abdomen, Pre-IDS Evaluation, Frequency, 0=Never | 2 | 1
  Pain in the Abdomen, Pre-IDS Evaluation, Frequency, 1=Rarely: number analyzed (Participants) | 2 | 1
  Pain in the Abdomen, Pre-IDS Evaluation, Frequency, 1=Rarely | 0 | 0
  Pain in the Abdomen, Pre-IDS Evaluation, Frequency, 2=Occasionally: number analyzed (Participants) | 2 | 1
  Pain in the Abdomen, Pre-IDS Evaluation, Frequency, 2=Occasionally | 0 | 0
  Pain in the Abdomen, Pre-IDS Evaluation, Frequency, 3=Frequently: number analyzed (Participants) | 2 | 1
  Pain in the Abdomen, Pre-IDS Evaluation, Frequency, 3=Frequently | 0 | 0
  Pain in the Abdomen, Pre-IDS Evaluation, Frequency, 4=Almost constantly: number analyzed (Participants) | 2 | 1
  Pain in the Abdomen, Pre-IDS Evaluation, Frequency, 4=Almost constantly | 0 | 0
  Pain in the Abdomen, End Of Treatment, Severity, 0=None: number analyzed (Participants) | 0 | 2
  Pain in the Abdomen, End Of Treatment, Severity, 0=None |  | 0
  Pain in the Abdomen, End Of Treatment, Severity, 1=Mild: number analyzed (Participants) | 0 | 2
  Pain in the Abdomen, End Of Treatment, Severity, 1=Mild |  | 1
  Pain in the Abdomen, End Of Treatment, Severity, 2=Moderate: number analyzed (Participants) | 0 | 2
  Pain in the Abdomen, End Of Treatment, Severity, 2=Moderate |  | 1
  Pain in the Abdomen, End Of Treatment, Severity, 3=Severe: number analyzed (Participants) | 0 | 2
  Pain in the Abdomen, End Of Treatment, Severity, 3=Severe |  | 0
  Pain in the Abdomen, End Of Treatment, Severity, 4=Very severe: number analyzed (Participants) | 0 | 2
  Pain in the Abdomen, End Of Treatment, Severity, 4=Very severe |  | 0
  Pain in the Abdomen, End Of Treatment, Frequency, 0=Never: number analyzed (Participants) | 0 | 5
  Pain in the Abdomen, End Of Treatment, Frequency, 0=Never |  | 3
  Pain in the Abdomen, End Of Treatment, Frequency, 1=Rarely: number analyzed (Participants) | 0 | 5
  Pain in the Abdomen, End Of Treatment, Frequency, 1=Rarely |  | 1
  Pain in the Abdomen, End Of Treatment, Frequency, 2=Occasionally: number analyzed (Participants) | 0 | 5
  Pain in the Abdomen, End Of Treatment, Frequency, 2=Occasionally |  | 1
  Pain in the Abdomen, End Of Treatment, Frequency, 3=Frequently: number analyzed (Participants) | 0 | 5
  Pain in the Abdomen, End Of Treatment, Frequency, 3=Frequently |  | 0
  Pain in the Abdomen, End Of Treatment, Frequency, 4=Almost constantly: number analyzed (Participants) | 0 | 5
  Pain in the Abdomen, End Of Treatment, Frequency, 4=Almost constantly |  | 0
  Numb/Tingling Hands/Feet, Baseline, Severity, 0=None: number analyzed (Participants) | 14 | 17
  Numb/Tingling Hands/Feet, Baseline, Severity, 0=None | 7 | 15
  Numb/Tingling Hands/Feet, Baseline, Severity, 1=Mild: number analyzed (Participants) | 14 | 17
  Numb/Tingling Hands/Feet, Baseline, Severity, 1=Mild | 4 | 2
  Numb/Tingling Hands/Feet, Baseline, Severity, 2=Moderate: number analyzed (Participants) | 14 | 17
  Numb/Tingling Hands/Feet, Baseline, Severity, 2=Moderate | 2 | 0
  Numb/Tingling Hands/Feet, Baseline, Severity, 3=Severe: number analyzed (Participants) | 14 | 17
  Numb/Tingling Hands/Feet, Baseline, Severity, 3=Severe | 1 | 0
  Numb/Tingling Hands/Feet, Baseline, Severity, 4=Very severe: number analyzed (Participants) | 14 | 17
  Numb/Tingling Hands/Feet, Baseline, Severity, 4=Very severe | 0 | 0
  Numb/Tingling Hands/Feet, Cycle 1 Day 8, Severity, 0=None: number analyzed (Participants) | 11 | 15
  Numb/Tingling Hands/Feet, Cycle 1 Day 8, Severity, 0=None | 5 | 11
  Numb/Tingling Hands/Feet, Cycle 1 Day 8, Severity, 1=Mild: number analyzed (Participants) | 11 | 15
  Numb/Tingling Hands/Feet, Cycle 1 Day 8, Severity, 1=Mild | 2 | 4
  Numb/Tingling Hands/Feet, Cycle 1 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 11 | 15
  Numb/Tingling Hands/Feet, Cycle 1 Day 8, Severity, 2=Moderate | 2 | 0
  Numb/Tingling Hands/Feet, Cycle 1 Day 8, Severity, 3=Severe: number analyzed (Participants) | 11 | 15
  Numb/Tingling Hands/Feet, Cycle 1 Day 8, Severity, 3=Severe | 2 | 0
  Numb/Tingling Hands/Feet, Cycle 1 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 11 | 15
  Numb/Tingling Hands/Feet, Cycle 1 Day 8, Severity, 4=Very severe | 0 | 0
  Numb/Tingling Hands/Feet, Cycle 1 Day 15, Severity, 0=None: number analyzed (Participants) | 14 | 13
  Numb/Tingling Hands/Feet, Cycle 1 Day 15, Severity, 0=None | 5 | 11
  Numb/Tingling Hands/Feet, Cycle 1 Day 15, Severity, 1=Mild: number analyzed (Participants) | 14 | 13
  Numb/Tingling Hands/Feet, Cycle 1 Day 15, Severity, 1=Mild | 6 | 2
  Numb/Tingling Hands/Feet, Cycle 1 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 14 | 13
  Numb/Tingling Hands/Feet, Cycle 1 Day 15, Severity, 2=Moderate | 3 | 0
  Numb/Tingling Hands/Feet, Cycle 1 Day 15, Severity, 3=Severe: number analyzed (Participants) | 14 | 13
  Numb/Tingling Hands/Feet, Cycle 1 Day 15, Severity, 3=Severe | 0 | 0
  Numb/Tingling Hands/Feet, Cycle 1 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 14 | 13
  Numb/Tingling Hands/Feet, Cycle 1 Day 15, Severity, 4=Very severe | 0 | 0
  Numb/Tingling Hands/Feet, Cycle 2 Day 1, Severity, 0=None: number analyzed (Participants) | 11 | 14
  Numb/Tingling Hands/Feet, Cycle 2 Day 1, Severity, 0=None | 6 | 14
  Numb/Tingling Hands/Feet, Cycle 2 Day 1, Severity, 1=Mild: number analyzed (Participants) | 11 | 14
  Numb/Tingling Hands/Feet, Cycle 2 Day 1, Severity, 1=Mild | 2 | 0
  Numb/Tingling Hands/Feet, Cycle 2 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 11 | 14
  Numb/Tingling Hands/Feet, Cycle 2 Day 1, Severity, 2=Moderate | 3 | 0
  Numb/Tingling Hands/Feet, Cycle 2 Day 1, Severity, 3=Severe: number analyzed (Participants) | 11 | 14
  Numb/Tingling Hands/Feet, Cycle 2 Day 1, Severity, 3=Severe | 0 | 0
  Numb/Tingling Hands/Feet, Cycle 2 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 11 | 14
  Numb/Tingling Hands/Feet, Cycle 2 Day 1, Severity, 4=Very severe | 0 | 0
  Numb/Tingling Hands/Feet, Cycle 2 Day 8, Severity, 0=None: number analyzed (Participants) | 11 | 11
  Numb/Tingling Hands/Feet, Cycle 2 Day 8, Severity, 0=None | 2 | 10
  Numb/Tingling Hands/Feet, Cycle 2 Day 8, Severity, 1=Mild: number analyzed (Participants) | 11 | 11
  Numb/Tingling Hands/Feet, Cycle 2 Day 8, Severity, 1=Mild | 5 | 1
  Numb/Tingling Hands/Feet, Cycle 2 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 11 | 11
  Numb/Tingling Hands/Feet, Cycle 2 Day 8, Severity, 2=Moderate | 2 | 0
  Numb/Tingling Hands/Feet, Cycle 2 Day 8, Severity, 3=Severe: number analyzed (Participants) | 11 | 11
  Numb/Tingling Hands/Feet, Cycle 2 Day 8, Severity, 3=Severe | 2 | 0
  Numb/Tingling Hands/Feet, Cycle 2 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 11 | 11
  Numb/Tingling Hands/Feet, Cycle 2 Day 8, Severity, 4=Very severe | 0 | 0
  Numb/Tingling Hands/Feet, Cycle 2 Day 15, Severity, 0=None: number analyzed (Participants) | 13 | 14
  Numb/Tingling Hands/Feet, Cycle 2 Day 15, Severity, 0=None | 1 | 13
  Numb/Tingling Hands/Feet, Cycle 2 Day 15, Severity, 1=Mild: number analyzed (Participants) | 13 | 14
  Numb/Tingling Hands/Feet, Cycle 2 Day 15, Severity, 1=Mild | 5 | 1
  Numb/Tingling Hands/Feet, Cycle 2 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 13 | 14
  Numb/Tingling Hands/Feet, Cycle 2 Day 15, Severity, 2=Moderate | 5 | 0
  Numb/Tingling Hands/Feet, Cycle 2 Day 15, Severity, 3=Severe: number analyzed (Participants) | 13 | 14
  Numb/Tingling Hands/Feet, Cycle 2 Day 15, Severity, 3=Severe | 2 | 0
  Numb/Tingling Hands/Feet, Cycle 2 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 13 | 14
  Numb/Tingling Hands/Feet, Cycle 2 Day 15, Severity, 4=Very severe | 0 | 0
  Numb/Tingling Hands/Feet, Cycle 3 Day 1, Severity, 0=None: number analyzed (Participants) | 14 | 14
  Numb/Tingling Hands/Feet, Cycle 3 Day 1, Severity, 0=None | 3 | 13
  Numb/Tingling Hands/Feet, Cycle 3 Day 1, Severity, 1=Mild: number analyzed (Participants) | 14 | 14
  Numb/Tingling Hands/Feet, Cycle 3 Day 1, Severity, 1=Mild | 8 | 1
  Numb/Tingling Hands/Feet, Cycle 3 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 14 | 14
  Numb/Tingling Hands/Feet, Cycle 3 Day 1, Severity, 2=Moderate | 3 | 0
  Numb/Tingling Hands/Feet, Cycle 3 Day 1, Severity, 3=Severe: number analyzed (Participants) | 14 | 14
  Numb/Tingling Hands/Feet, Cycle 3 Day 1, Severity, 3=Severe | 0 | 0
  Numb/Tingling Hands/Feet, Cycle 3 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 14 | 14
  Numb/Tingling Hands/Feet, Cycle 3 Day 1, Severity, 4=Very severe | 0 | 0
  Numb/Tingling Hands/Feet, Cycle 3 Day 8, Severity, 0=None: number analyzed (Participants) | 10 | 10
  Numb/Tingling Hands/Feet, Cycle 3 Day 8, Severity, 0=None | 1 | 8
  Numb/Tingling Hands/Feet, Cycle 3 Day 8, Severity, 1=Mild: number analyzed (Participants) | 10 | 10
  Numb/Tingling Hands/Feet, Cycle 3 Day 8, Severity, 1=Mild | 2 | 2
  Numb/Tingling Hands/Feet, Cycle 3 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 10 | 10
  Numb/Tingling Hands/Feet, Cycle 3 Day 8, Severity, 2=Moderate | 5 | 0
  Numb/Tingling Hands/Feet, Cycle 3 Day 8, Severity, 3=Severe: number analyzed (Participants) | 10 | 10
  Numb/Tingling Hands/Feet, Cycle 3 Day 8, Severity, 3=Severe | 1 | 0
  Numb/Tingling Hands/Feet, Cycle 3 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 10 | 10
  Numb/Tingling Hands/Feet, Cycle 3 Day 8, Severity, 4=Very severe | 1 | 0
  Numb/Tingling Hands/Feet, Cycle 3 Day 15, Severity, 0=None: number analyzed (Participants) | 5 | 7
  Numb/Tingling Hands/Feet, Cycle 3 Day 15, Severity, 0=None | 0 | 5
  Numb/Tingling Hands/Feet, Cycle 3 Day 15, Severity, 1=Mild: number analyzed (Participants) | 5 | 7
  Numb/Tingling Hands/Feet, Cycle 3 Day 15, Severity, 1=Mild | 3 | 2
  Numb/Tingling Hands/Feet, Cycle 3 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 5 | 7
  Numb/Tingling Hands/Feet, Cycle 3 Day 15, Severity, 2=Moderate | 1 | 0
  Numb/Tingling Hands/Feet, Cycle 3 Day 15, Severity, 3=Severe: number analyzed (Participants) | 5 | 7
  Numb/Tingling Hands/Feet, Cycle 3 Day 15, Severity, 3=Severe | 1 | 0
  Numb/Tingling Hands/Feet, Cycle 3 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 5 | 7
  Numb/Tingling Hands/Feet, Cycle 3 Day 15, Severity, 4=Very severe | 0 | 0
  Numb/Tingling Hands/Feet, Pre-IDS Evaluation, Severity, 0=None: number analyzed (Participants) | 2 | 1
  Numb/Tingling Hands/Feet, Pre-IDS Evaluation, Severity, 0=None | 1 | 1
  Numb/Tingling Hands/Feet, Pre-IDS Evaluation, Severity, 1=Mild: number analyzed (Participants) | 2 | 1
  Numb/Tingling Hands/Feet, Pre-IDS Evaluation, Severity, 1=Mild | 1 | 0
  Numb/Tingling Hands/Feet, Pre-IDS Evaluation, Severity, 2=Moderate: number analyzed (Participants) | 2 | 1
  Numb/Tingling Hands/Feet, Pre-IDS Evaluation, Severity, 2=Moderate | 0 | 0
  Numb/Tingling Hands/Feet, Pre-IDS Evaluation, Severity, 3=Severe: number analyzed (Participants) | 2 | 1
  Numb/Tingling Hands/Feet, Pre-IDS Evaluation, Severity, 3=Severe | 0 | 0
  Numb/Tingling Hands/Feet, Pre-IDS Evaluation, Severity, 4=Very severe: number analyzed (Participants) | 2 | 1
  Numb/Tingling Hands/Feet, Pre-IDS Evaluation, Severity, 4=Very severe | 0 | 0
  Numb/Tingling Hands/Feet, End Of Treatment, Severity, 0=None: number analyzed (Participants) | 0 | 5
  Numb/Tingling Hands/Feet, End Of Treatment, Severity, 0=None |  | 4
  Numb/Tingling Hands/Feet, End Of Treatment, Severity, 1=Mild: number analyzed (Participants) | 0 | 5
  Numb/Tingling Hands/Feet, End Of Treatment, Severity, 1=Mild |  | 0
  Numb/Tingling Hands/Feet, End Of Treatment, Severity, 2=Moderate: number analyzed (Participants) | 0 | 5
  Numb/Tingling Hands/Feet, End Of Treatment, Severity, 2=Moderate |  | 1
  Numb/Tingling Hands/Feet, End Of Treatment, Severity, 3=Severe: number analyzed (Participants) | 0 | 5
  Numb/Tingling Hands/Feet, End Of Treatment, Severity, 3=Severe |  | 0
  Numb/Tingling Hands/Feet, End Of Treatment, Severity, 4=Very severe: number analyzed (Participants) | 0 | 5
  Numb/Tingling Hands/Feet, End Of Treatment, Severity, 4=Very severe |  | 0
  Probs w/Concentration, Baseline, Severity, 0=None: number analyzed (Participants) | 14 | 17
  Probs w/Concentration, Baseline, Severity, 0=None | 4 | 7
  Probs w/Concentration, Baseline, Severity, 1=Mild: number analyzed (Participants) | 14 | 17
  Probs w/Concentration, Baseline, Severity, 1=Mild | 8 | 7
  Probs w/Concentration, Baseline, Severity, 2=Moderate: number analyzed (Participants) | 14 | 17
  Probs w/Concentration, Baseline, Severity, 2=Moderate | 1 | 3
  Probs w/Concentration, Baseline, Severity, 3=Severe: number analyzed (Participants) | 14 | 17
  Probs w/Concentration, Baseline, Severity, 3=Severe | 1 | 0
  Probs w/Concentration, Baseline, Severity, 4=Very severe: number analyzed (Participants) | 14 | 17
  Probs w/Concentration, Baseline, Severity, 4=Very severe | 0 | 0
  Probs w/Concentration, Cycle 1 Day 8, Severity, 0=None: number analyzed (Participants) | 11 | 15
  Probs w/Concentration, Cycle 1 Day 8, Severity, 0=None | 3 | 4
  Probs w/Concentration, Cycle 1 Day 8, Severity, 1=Mild: number analyzed (Participants) | 11 | 15
  Probs w/Concentration, Cycle 1 Day 8, Severity, 1=Mild | 2 | 10
  Probs w/Concentration, Cycle 1 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 11 | 15
  Probs w/Concentration, Cycle 1 Day 8, Severity, 2=Moderate | 6 | 1
  Probs w/Concentration, Cycle 1 Day 8, Severity, 3=Severe: number analyzed (Participants) | 11 | 15
  Probs w/Concentration, Cycle 1 Day 8, Severity, 3=Severe | 0 | 0
  Probs w/Concentration, Cycle 1 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 11 | 15
  Probs w/Concentration, Cycle 1 Day 8, Severity, 4=Very severe | 0 | 0
  Probs w/Concentration, Cycle 1 Day 15, Severity, 0=None: number analyzed (Participants) | 14 | 13
  Probs w/Concentration, Cycle 1 Day 15, Severity, 0=None | 7 | 7
  Probs w/Concentration, Cycle 1 Day 15, Severity, 1=Mild: number analyzed (Participants) | 14 | 13
  Probs w/Concentration, Cycle 1 Day 15, Severity, 1=Mild | 5 | 3
  Probs w/Concentration, Cycle 1 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 14 | 13
  Probs w/Concentration, Cycle 1 Day 15, Severity, 2=Moderate | 2 | 3
  Probs w/Concentration, Cycle 1 Day 15, Severity, 3=Severe: number analyzed (Participants) | 14 | 13
  Probs w/Concentration, Cycle 1 Day 15, Severity, 3=Severe | 0 | 0
  Probs w/Concentration, Cycle 1 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 14 | 13
  Probs w/Concentration, Cycle 1 Day 15, Severity, 4=Very severe | 0 | 0
  Probs w/Concentration, Cycle 2 Day 1, Severity, 0=None: number analyzed (Participants) | 11 | 14
  Probs w/Concentration, Cycle 2 Day 1, Severity, 0=None | 5 | 6
  Probs w/Concentration, Cycle 2 Day 1, Severity, 1=Mild: number analyzed (Participants) | 11 | 14
  Probs w/Concentration, Cycle 2 Day 1, Severity, 1=Mild | 4 | 6
  Probs w/Concentration, Cycle 2 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 11 | 14
  Probs w/Concentration, Cycle 2 Day 1, Severity, 2=Moderate | 2 | 2
  Probs w/Concentration, Cycle 2 Day 1, Severity, 3=Severe: number analyzed (Participants) | 11 | 14
  Probs w/Concentration, Cycle 2 Day 1, Severity, 3=Severe | 0 | 0
  Probs w/Concentration, Cycle 2 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 11 | 14
  Probs w/Concentration, Cycle 2 Day 1, Severity, 4=Very severe | 0 | 0
  Probs w/Concentration, Cycle 2 Day 8, Severity, 0=None: number analyzed (Participants) | 11 | 11
  Probs w/Concentration, Cycle 2 Day 8, Severity, 0=None | 3 | 7
  Probs w/Concentration, Cycle 2 Day 8, Severity, 1=Mild: number analyzed (Participants) | 11 | 11
  Probs w/Concentration, Cycle 2 Day 8, Severity, 1=Mild | 4 | 4
  Probs w/Concentration, Cycle 2 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 11 | 11
  Probs w/Concentration, Cycle 2 Day 8, Severity, 2=Moderate | 3 | 0
  Probs w/Concentration, Cycle 2 Day 8, Severity, 3=Severe: number analyzed (Participants) | 11 | 11
  Probs w/Concentration, Cycle 2 Day 8, Severity, 3=Severe | 0 | 0
  Probs w/Concentration, Cycle 2 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 11 | 11
  Probs w/Concentration, Cycle 2 Day 8, Severity, 4=Very severe | 1 | 0
  Probs w/Concentration, Cycle 2 Day 15, Severity, 0=None: number analyzed (Participants) | 13 | 14
  Probs w/Concentration, Cycle 2 Day 15, Severity, 0=None | 4 | 9
  Probs w/Concentration, Cycle 2 Day 15, Severity, 1=Mild: number analyzed (Participants) | 13 | 14
  Probs w/Concentration, Cycle 2 Day 15, Severity, 1=Mild | 8 | 4
  Probs w/Concentration, Cycle 2 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 13 | 14
  Probs w/Concentration, Cycle 2 Day 15, Severity, 2=Moderate | 1 | 1
  Probs w/Concentration, Cycle 2 Day 15, Severity, 3=Severe: number analyzed (Participants) | 13 | 14
  Probs w/Concentration, Cycle 2 Day 15, Severity, 3=Severe | 0 | 0
  Probs w/Concentration, Cycle 2 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 13 | 14
  Probs w/Concentration, Cycle 2 Day 15, Severity, 4=Very severe | 0 | 0
  Probs w/Concentration, Cycle 3 Day 1, Severity, 0=None: number analyzed (Participants) | 14 | 14
  Probs w/Concentration, Cycle 3 Day 1, Severity, 0=None | 8 | 9
  Probs w/Concentration, Cycle 3 Day 1, Severity, 1=Mild: number analyzed (Participants) | 14 | 14
  Probs w/Concentration, Cycle 3 Day 1, Severity, 1=Mild | 5 | 3
  Probs w/Concentration, Cycle 3 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 14 | 14
  Probs w/Concentration, Cycle 3 Day 1, Severity, 2=Moderate | 1 | 1
  Probs w/Concentration, Cycle 3 Day 1, Severity, 3=Severe: number analyzed (Participants) | 14 | 14
  Probs w/Concentration, Cycle 3 Day 1, Severity, 3=Severe | 0 | 1
  Probs w/Concentration, Cycle 3 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 14 | 14
  Probs w/Concentration, Cycle 3 Day 1, Severity, 4=Very severe | 0 | 0
  Probs w/Concentration, Cycle 3 Day 8, Severity, 0=None: number analyzed (Participants) | 10 | 10
  Probs w/Concentration, Cycle 3 Day 8, Severity, 0=None | 4 | 5
  Probs w/Concentration, Cycle 3 Day 8, Severity, 1=Mild: number analyzed (Participants) | 10 | 10
  Probs w/Concentration, Cycle 3 Day 8, Severity, 1=Mild | 1 | 4
  Probs w/Concentration, Cycle 3 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 10 | 10
  Probs w/Concentration, Cycle 3 Day 8, Severity, 2=Moderate | 4 | 1
  Probs w/Concentration, Cycle 3 Day 8, Severity, 3=Severe: number analyzed (Participants) | 10 | 10
  Probs w/Concentration, Cycle 3 Day 8, Severity, 3=Severe | 1 | 0
  Probs w/Concentration, Cycle 3 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 10 | 10
  Probs w/Concentration, Cycle 3 Day 8, Severity, 4=Very severe | 0 | 0
  Probs w/Concentration, Cycle 3 Day 15, Severity, 0=None: number analyzed (Participants) | 5 | 7
  Probs w/Concentration, Cycle 3 Day 15, Severity, 0=None | 1 | 4
  Probs w/Concentration, Cycle 3 Day 15, Severity, 1=Mild: number analyzed (Participants) | 5 | 7
  Probs w/Concentration, Cycle 3 Day 15, Severity, 1=Mild | 3 | 2
  Probs w/Concentration, Cycle 3 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 5 | 7
  Probs w/Concentration, Cycle 3 Day 15, Severity, 2=Moderate | 1 | 1
  Probs w/Concentration, Cycle 3 Day 15, Severity, 3=Severe: number analyzed (Participants) | 5 | 7
  Probs w/Concentration, Cycle 3 Day 15, Severity, 3=Severe | 0 | 0
  Probs w/Concentration, Cycle 3 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 5 | 7
  Probs w/Concentration, Cycle 3 Day 15, Severity, 4=Very severe | 0 | 0
  Probs w/Concentration, Pre-IDS Evaluation, Severity, 0=None: number analyzed (Participants) | 2 | 1
  Probs w/Concentration, Pre-IDS Evaluation, Severity, 0=None | 2 | 0
  Probs w/Concentration, Pre-IDS Evaluation, Severity, 1=Mild: number analyzed (Participants) | 2 | 1
  Probs w/Concentration, Pre-IDS Evaluation, Severity, 1=Mild | 0 | 0
  Probs w/Concentration, Pre-IDS Evaluation, Severity, 2=Moderate: number analyzed (Participants) | 2 | 1
  Probs w/Concentration, Pre-IDS Evaluation, Severity, 2=Moderate | 0 | 0
  Probs w/Concentration, Pre-IDS Evaluation, Severity, 3=Severe: number analyzed (Participants) | 2 | 1
  Probs w/Concentration, Pre-IDS Evaluation, Severity, 3=Severe | 0 | 1
  Probs w/Concentration, Pre-IDS Evaluation, Severity, 4=Very severe: number analyzed (Participants) | 2 | 1
  Probs w/Concentration, Pre-IDS Evaluation, Severity, 4=Very severe | 0 | 0
  Probs w/Concentration, End Of Treatment, Severity, 0=None: number analyzed (Participants) | 0 | 5
  Probs w/Concentration, End Of Treatment, Severity, 0=None |  | 3
  Probs w/Concentration, End Of Treatment, Severity, 1=Mild: number analyzed (Participants) | 0 | 5
  Probs w/Concentration, End Of Treatment, Severity, 1=Mild |  | 1
  Probs w/Concentration, End Of Treatment, Severity, 2=Moderate: number analyzed (Participants) | 0 | 5
  Probs w/Concentration, End Of Treatment, Severity, 2=Moderate |  | 1
  Probs w/Concentration, End Of Treatment, Severity, 3=Severe: number analyzed (Participants) | 0 | 5
  Probs w/Concentration, End Of Treatment, Severity, 3=Severe |  | 0
  Probs w/Concentration, End Of Treatment, Severity, 4=Very severe: number analyzed (Participants) | 0 | 5
  Probs w/Concentration, End Of Treatment, Severity, 4=Very severe |  | 0
  Problems w/Memory, Baseline, Severity, 0=None: number analyzed (Participants) | 14 | 17
  Problems w/Memory, Baseline, Severity, 0=None | 7 | 6
  Problems w/Memory, Baseline, Severity, 1=Mild: number analyzed (Participants) | 14 | 17
  Problems w/Memory, Baseline, Severity, 1=Mild | 6 | 8
  Problems w/Memory, Baseline, Severity, 2=Moderate: number analyzed (Participants) | 14 | 17
  Problems w/Memory, Baseline, Severity, 2=Moderate | 0 | 2
  Problems w/Memory, Baseline, Severity, 3=Severe: number analyzed (Participants) | 14 | 17
  Problems w/Memory, Baseline, Severity, 3=Severe | 0 | 1
  Problems w/Memory, Baseline, Severity, 4=Very severe: number analyzed (Participants) | 14 | 17
  Problems w/Memory, Baseline, Severity, 4=Very severe | 1 | 0
  Problems w/Memory, Cycle 1 Day 8, Severity, 0=None: number analyzed (Participants) | 11 | 15
  Problems w/Memory, Cycle 1 Day 8, Severity, 0=None | 7 | 5
  Problems w/Memory, Cycle 1 Day 8, Severity, 1=Mild: number analyzed (Participants) | 11 | 15
  Problems w/Memory, Cycle 1 Day 8, Severity, 1=Mild | 3 | 8
  Problems w/Memory, Cycle 1 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 11 | 15
  Problems w/Memory, Cycle 1 Day 8, Severity, 2=Moderate | 1 | 2
  Problems w/Memory, Cycle 1 Day 8, Severity, 3=Severe: number analyzed (Participants) | 11 | 15
  Problems w/Memory, Cycle 1 Day 8, Severity, 3=Severe | 0 | 0
  Problems w/Memory, Cycle 1 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 11 | 15
  Problems w/Memory, Cycle 1 Day 8, Severity, 4=Very severe | 0 | 0
  Problems w/Memory, Cycle 1 Day 15, Severity, 0=None: number analyzed (Participants) | 14 | 13
  Problems w/Memory, Cycle 1 Day 15, Severity, 0=None | 6 | 5
  Problems w/Memory, Cycle 1 Day 15, Severity, 1=Mild: number analyzed (Participants) | 14 | 13
  Problems w/Memory, Cycle 1 Day 15, Severity, 1=Mild | 7 | 6
  Problems w/Memory, Cycle 1 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 14 | 13
  Problems w/Memory, Cycle 1 Day 15, Severity, 2=Moderate | 1 | 2
  Problems w/Memory, Cycle 1 Day 15, Severity, 3=Severe: number analyzed (Participants) | 14 | 13
  Problems w/Memory, Cycle 1 Day 15, Severity, 3=Severe | 0 | 0
  Problems w/Memory, Cycle 1 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 14 | 13
  Problems w/Memory, Cycle 1 Day 15, Severity, 4=Very severe | 0 | 0
  Problems w/Memory, Cycle 2 Day 1, Severity, 0=None: number analyzed (Participants) | 11 | 14
  Problems w/Memory, Cycle 2 Day 1, Severity, 0=None | 5 | 6
  Problems w/Memory, Cycle 2 Day 1, Severity, 1=Mild: number analyzed (Participants) | 11 | 14
  Problems w/Memory, Cycle 2 Day 1, Severity, 1=Mild | 4 | 5
  Problems w/Memory, Cycle 2 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 11 | 14
  Problems w/Memory, Cycle 2 Day 1, Severity, 2=Moderate | 2 | 3
  Problems w/Memory, Cycle 2 Day 1, Severity, 3=Severe: number analyzed (Participants) | 11 | 14
  Problems w/Memory, Cycle 2 Day 1, Severity, 3=Severe | 0 | 0
  Problems w/Memory, Cycle 2 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 11 | 14
  Problems w/Memory, Cycle 2 Day 1, Severity, 4=Very severe | 0 | 0
  Problems w/Memory, Cycle 2 Day 8, Severity, 0=None: number analyzed (Participants) | 11 | 11
  Problems w/Memory, Cycle 2 Day 8, Severity, 0=None | 5 | 6
  Problems w/Memory, Cycle 2 Day 8, Severity, 1=Mild: number analyzed (Participants) | 11 | 11
  Problems w/Memory, Cycle 2 Day 8, Severity, 1=Mild | 5 | 4
  Problems w/Memory, Cycle 2 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 11 | 11
  Problems w/Memory, Cycle 2 Day 8, Severity, 2=Moderate | 1 | 1
  Problems w/Memory, Cycle 2 Day 8, Severity, 3=Severe: number analyzed (Participants) | 11 | 11
  Problems w/Memory, Cycle 2 Day 8, Severity, 3=Severe | 0 | 0
  Problems w/Memory, Cycle 2 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 11 | 11
  Problems w/Memory, Cycle 2 Day 8, Severity, 4=Very severe | 0 | 0
  Problems w/Memory, Cycle 2 Day 15, Severity, 0=None: number analyzed (Participants) | 13 | 14
  Problems w/Memory, Cycle 2 Day 15, Severity, 0=None | 6 | 5
  Problems w/Memory, Cycle 2 Day 15, Severity, 1=Mild: number analyzed (Participants) | 13 | 14
  Problems w/Memory, Cycle 2 Day 15, Severity, 1=Mild | 7 | 7
  Problems w/Memory, Cycle 2 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 13 | 14
  Problems w/Memory, Cycle 2 Day 15, Severity, 2=Moderate | 0 | 1
  Problems w/Memory, Cycle 2 Day 15, Severity, 3=Severe: number analyzed (Participants) | 13 | 14
  Problems w/Memory, Cycle 2 Day 15, Severity, 3=Severe | 0 | 1
  Problems w/Memory, Cycle 2 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 13 | 14
  Problems w/Memory, Cycle 2 Day 15, Severity, 4=Very severe | 0 | 0
  Problems w/Memory, Cycle 3 Day 1, Severity, 0=None: number analyzed (Participants) | 14 | 14
  Problems w/Memory, Cycle 3 Day 1, Severity, 0=None | 8 | 9
  Problems w/Memory, Cycle 3 Day 1, Severity, 1=Mild: number analyzed (Participants) | 14 | 14
  Problems w/Memory, Cycle 3 Day 1, Severity, 1=Mild | 6 | 3
  Problems w/Memory, Cycle 3 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 14 | 14
  Problems w/Memory, Cycle 3 Day 1, Severity, 2=Moderate | 0 | 1
  Problems w/Memory, Cycle 3 Day 1, Severity, 3=Severe: number analyzed (Participants) | 14 | 14
  Problems w/Memory, Cycle 3 Day 1, Severity, 3=Severe | 0 | 0
  Problems w/Memory, Cycle 3 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 14 | 14
  Problems w/Memory, Cycle 3 Day 1, Severity, 4=Very severe | 0 | 1
  Problems w/Memory, Cycle 3 Day 8, Severity, 0=None: number analyzed (Participants) | 10 | 10
  Problems w/Memory, Cycle 3 Day 8, Severity, 0=None | 5 | 4
  Problems w/Memory, Cycle 3 Day 8, Severity, 1=Mild: number analyzed (Participants) | 10 | 10
  Problems w/Memory, Cycle 3 Day 8, Severity, 1=Mild | 1 | 5
  Problems w/Memory, Cycle 3 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 10 | 10
  Problems w/Memory, Cycle 3 Day 8, Severity, 2=Moderate | 3 | 1
  Problems w/Memory, Cycle 3 Day 8, Severity, 3=Severe: number analyzed (Participants) | 10 | 10
  Problems w/Memory, Cycle 3 Day 8, Severity, 3=Severe | 1 | 0
  Problems w/Memory, Cycle 3 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 10 | 10
  Problems w/Memory, Cycle 3 Day 8, Severity, 4=Very severe | 0 | 0
  Problems w/Memory, Cycle 3 Day 15, Severity, 0=None: number analyzed (Participants) | 5 | 7
  Problems w/Memory, Cycle 3 Day 15, Severity, 0=None | 2 | 4
  Problems w/Memory, Cycle 3 Day 15, Severity, 1=Mild: number analyzed (Participants) | 5 | 7
  Problems w/Memory, Cycle 3 Day 15, Severity, 1=Mild | 3 | 2
  Problems w/Memory, Cycle 3 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 5 | 7
  Problems w/Memory, Cycle 3 Day 15, Severity, 2=Moderate | 0 | 1
  Problems w/Memory, Cycle 3 Day 15, Severity, 3=Severe: number analyzed (Participants) | 5 | 7
  Problems w/Memory, Cycle 3 Day 15, Severity, 3=Severe | 0 | 0
  Problems w/Memory, Cycle 3 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 5 | 7
  Problems w/Memory, Cycle 3 Day 15, Severity, 4=Very severe | 0 | 0
  Problems w/Memory, Pre-IDS Evaluation, Severity, 0=None: number analyzed (Participants) | 2 | 1
  Problems w/Memory, Pre-IDS Evaluation, Severity, 0=None | 2 | 0
  Problems w/Memory, Pre-IDS Evaluation, Severity, 1=Mild: number analyzed (Participants) | 2 | 1
  Problems w/Memory, Pre-IDS Evaluation, Severity, 1=Mild | 0 | 0
  Problems w/Memory, Pre-IDS Evaluation, Severity, 2=Moderate: number analyzed (Participants) | 2 | 1
  Problems w/Memory, Pre-IDS Evaluation, Severity, 2=Moderate | 0 | 0
  Problems w/Memory, Pre-IDS Evaluation, Severity, 3=Severe: number analyzed (Participants) | 2 | 1
  Problems w/Memory, Pre-IDS Evaluation, Severity, 3=Severe | 0 | 0
  Problems w/Memory, Pre-IDS Evaluation, Severity, 4=Very severe: number analyzed (Participants) | 2 | 1
  Problems w/Memory, Pre-IDS Evaluation, Severity, 4=Very severe | 0 | 1
  Problems w/Memory, End Of Treatment, Severity, 0=None: number analyzed (Participants) | 0 | 5
  Problems w/Memory, End Of Treatment, Severity, 0=None |  | 4
  Problems w/Memory, End Of Treatment, Severity, 1=Mild: number analyzed (Participants) | 0 | 5
  Problems w/Memory, End Of Treatment, Severity, 1=Mild |  | 1
  Problems w/Memory, End Of Treatment, Severity, 2=Moderate: number analyzed (Participants) | 0 | 5
  Problems w/Memory, End Of Treatment, Severity, 2=Moderate |  | 0
  Problems w/Memory, End Of Treatment, Severity, 3=Severe: number analyzed (Participants) | 0 | 5
  Problems w/Memory, End Of Treatment, Severity, 3=Severe |  | 0
  Problems w/Memory, End Of Treatment, Severity, 4=Very severe: number analyzed (Participants) | 0 | 5
  Problems w/Memory, End Of Treatment, Severity, 4=Very severe |  | 0
  Aching Muscles, Baseline, Severity, 0=None: number analyzed (Participants) | 3 | 10
  Aching Muscles, Baseline, Severity, 0=None | 1 | 0
  Aching Muscles, Baseline, Severity, 1=Mild: number analyzed (Participants) | 3 | 10
  Aching Muscles, Baseline, Severity, 1=Mild | 0 | 4
  Aching Muscles, Baseline, Severity, 2=Moderate: number analyzed (Participants) | 3 | 10
  Aching Muscles, Baseline, Severity, 2=Moderate | 1 | 4
  Aching Muscles, Baseline, Severity, 3=Severe: number analyzed (Participants) | 3 | 10
  Aching Muscles, Baseline, Severity, 3=Severe | 1 | 2
  Aching Muscles, Baseline, Severity, 4=Very severe: number analyzed (Participants) | 3 | 10
  Aching Muscles, Baseline, Severity, 4=Very severe | 0 | 0
  Aching Muscles, Baseline, Frequency, 0=Never: number analyzed (Participants) | 14 | 17
  Aching Muscles, Baseline, Frequency, 0=Never | 11 | 7
  Aching Muscles, Baseline, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 17
  Aching Muscles, Baseline, Frequency, 1=Rarely | 1 | 6
  Aching Muscles, Baseline, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 17
  Aching Muscles, Baseline, Frequency, 2=Occasionally | 1 | 2
  Aching Muscles, Baseline, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 17
  Aching Muscles, Baseline, Frequency, 3=Frequently | 0 | 2
  Aching Muscles, Baseline, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 17
  Aching Muscles, Baseline, Frequency, 4=Almost constantly | 1 | 0
  Aching Muscles, Cycle 1 Day 8, Severity, 0=None: number analyzed (Participants) | 9 | 7
  Aching Muscles, Cycle 1 Day 8, Severity, 0=None | 1 | 0
  Aching Muscles, Cycle 1 Day 8, Severity, 1=Mild: number analyzed (Participants) | 9 | 7
  Aching Muscles, Cycle 1 Day 8, Severity, 1=Mild | 1 | 4
  Aching Muscles, Cycle 1 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 9 | 7
  Aching Muscles, Cycle 1 Day 8, Severity, 2=Moderate | 2 | 3
  Aching Muscles, Cycle 1 Day 8, Severity, 3=Severe: number analyzed (Participants) | 9 | 7
  Aching Muscles, Cycle 1 Day 8, Severity, 3=Severe | 1 | 0
  Aching Muscles, Cycle 1 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 9 | 7
  Aching Muscles, Cycle 1 Day 8, Severity, 4=Very severe | 4 | 0
  Aching Muscles, Cycle 1 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 15
  Aching Muscles, Cycle 1 Day 8, Frequency, 0=Never | 2 | 8
  Aching Muscles, Cycle 1 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 15
  Aching Muscles, Cycle 1 Day 8, Frequency, 1=Rarely | 2 | 3
  Aching Muscles, Cycle 1 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 15
  Aching Muscles, Cycle 1 Day 8, Frequency, 2=Occasionally | 2 | 2
  Aching Muscles, Cycle 1 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 15
  Aching Muscles, Cycle 1 Day 8, Frequency, 3=Frequently | 1 | 2
  Aching Muscles, Cycle 1 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 15
  Aching Muscles, Cycle 1 Day 8, Frequency, 4=Almost constantly | 4 | 0
  Aching Muscles, Cycle 1 Day 15, Severity, 0=None: number analyzed (Participants) | 9 | 5
  Aching Muscles, Cycle 1 Day 15, Severity, 0=None | 1 | 0
  Aching Muscles, Cycle 1 Day 15, Severity, 1=Mild: number analyzed (Participants) | 9 | 5
  Aching Muscles, Cycle 1 Day 15, Severity, 1=Mild | 5 | 1
  Aching Muscles, Cycle 1 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 9 | 5
  Aching Muscles, Cycle 1 Day 15, Severity, 2=Moderate | 2 | 3
  Aching Muscles, Cycle 1 Day 15, Severity, 3=Severe: number analyzed (Participants) | 9 | 5
  Aching Muscles, Cycle 1 Day 15, Severity, 3=Severe | 0 | 1
  Aching Muscles, Cycle 1 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 9 | 5
  Aching Muscles, Cycle 1 Day 15, Severity, 4=Very severe | 1 | 0
  Aching Muscles, Cycle 1 Day 15, Frequency, 0=Never: number analyzed (Participants) | 14 | 13
  Aching Muscles, Cycle 1 Day 15, Frequency, 0=Never | 5 | 8
  Aching Muscles, Cycle 1 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 13
  Aching Muscles, Cycle 1 Day 15, Frequency, 1=Rarely | 3 | 1
  Aching Muscles, Cycle 1 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 13
  Aching Muscles, Cycle 1 Day 15, Frequency, 2=Occasionally | 5 | 4
  Aching Muscles, Cycle 1 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 13
  Aching Muscles, Cycle 1 Day 15, Frequency, 3=Frequently | 0 | 0
  Aching Muscles, Cycle 1 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 13
  Aching Muscles, Cycle 1 Day 15, Frequency, 4=Almost constantly | 1 | 0
  Aching Muscles, Cycle 2 Day 1, Severity, 0=None: number analyzed (Participants) | 3 | 6
  Aching Muscles, Cycle 2 Day 1, Severity, 0=None | 0 | 0
  Aching Muscles, Cycle 2 Day 1, Severity, 1=Mild: number analyzed (Participants) | 3 | 6
  Aching Muscles, Cycle 2 Day 1, Severity, 1=Mild | 3 | 2
  Aching Muscles, Cycle 2 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 3 | 6
  Aching Muscles, Cycle 2 Day 1, Severity, 2=Moderate | 0 | 4
  Aching Muscles, Cycle 2 Day 1, Severity, 3=Severe: number analyzed (Participants) | 3 | 6
  Aching Muscles, Cycle 2 Day 1, Severity, 3=Severe | 0 | 0
  Aching Muscles, Cycle 2 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 3 | 6
  Aching Muscles, Cycle 2 Day 1, Severity, 4=Very severe | 0 | 0
  Aching Muscles, Cycle 2 Day 1, Frequency, 0=Never: number analyzed (Participants) | 11 | 14
  Aching Muscles, Cycle 2 Day 1, Frequency, 0=Never | 8 | 8
  Aching Muscles, Cycle 2 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 14
  Aching Muscles, Cycle 2 Day 1, Frequency, 1=Rarely | 1 | 1
  Aching Muscles, Cycle 2 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 14
  Aching Muscles, Cycle 2 Day 1, Frequency, 2=Occasionally | 2 | 3
  Aching Muscles, Cycle 2 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 14
  Aching Muscles, Cycle 2 Day 1, Frequency, 3=Frequently | 0 | 2
  Aching Muscles, Cycle 2 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 14
  Aching Muscles, Cycle 2 Day 1, Frequency, 4=Almost constantly | 0 | 0
  Aching Muscles, Cycle 2 Day 8, Severity, 0=None: number analyzed (Participants) | 10 | 5
  Aching Muscles, Cycle 2 Day 8, Severity, 0=None | 0 | 0
  Aching Muscles, Cycle 2 Day 8, Severity, 1=Mild: number analyzed (Participants) | 10 | 5
  Aching Muscles, Cycle 2 Day 8, Severity, 1=Mild | 3 | 2
  Aching Muscles, Cycle 2 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 10 | 5
  Aching Muscles, Cycle 2 Day 8, Severity, 2=Moderate | 4 | 2
  Aching Muscles, Cycle 2 Day 8, Severity, 3=Severe: number analyzed (Participants) | 10 | 5
  Aching Muscles, Cycle 2 Day 8, Severity, 3=Severe | 2 | 1
  Aching Muscles, Cycle 2 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 10 | 5
  Aching Muscles, Cycle 2 Day 8, Severity, 4=Very severe | 1 | 0
  Aching Muscles, Cycle 2 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 11
  Aching Muscles, Cycle 2 Day 8, Frequency, 0=Never | 1 | 6
  Aching Muscles, Cycle 2 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 11
  Aching Muscles, Cycle 2 Day 8, Frequency, 1=Rarely | 4 | 2
  Aching Muscles, Cycle 2 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 11
  Aching Muscles, Cycle 2 Day 8, Frequency, 2=Occasionally | 1 | 2
  Aching Muscles, Cycle 2 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 11
  Aching Muscles, Cycle 2 Day 8, Frequency, 3=Frequently | 4 | 1
  Aching Muscles, Cycle 2 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 11
  Aching Muscles, Cycle 2 Day 8, Frequency, 4=Almost constantly | 1 | 0
  Aching Muscles, Cycle 2 Day 15, Severity, 0=None: number analyzed (Participants) | 9 | 7
  Aching Muscles, Cycle 2 Day 15, Severity, 0=None | 0 | 0
  Aching Muscles, Cycle 2 Day 15, Severity, 1=Mild: number analyzed (Participants) | 9 | 7
  Aching Muscles, Cycle 2 Day 15, Severity, 1=Mild | 5 | 6
  Aching Muscles, Cycle 2 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 9 | 7
  Aching Muscles, Cycle 2 Day 15, Severity, 2=Moderate | 1 | 0
  Aching Muscles, Cycle 2 Day 15, Severity, 3=Severe: number analyzed (Participants) | 9 | 7
  Aching Muscles, Cycle 2 Day 15, Severity, 3=Severe | 2 | 1
  Aching Muscles, Cycle 2 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 9 | 7
  Aching Muscles, Cycle 2 Day 15, Severity, 4=Very severe | 1 | 0
  Aching Muscles, Cycle 2 Day 15, Frequency, 0=Never: number analyzed (Participants) | 13 | 14
  Aching Muscles, Cycle 2 Day 15, Frequency, 0=Never | 4 | 7
  Aching Muscles, Cycle 2 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 13 | 14
  Aching Muscles, Cycle 2 Day 15, Frequency, 1=Rarely | 3 | 5
  Aching Muscles, Cycle 2 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 13 | 14
  Aching Muscles, Cycle 2 Day 15, Frequency, 2=Occasionally | 4 | 1
  Aching Muscles, Cycle 2 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 13 | 14
  Aching Muscles, Cycle 2 Day 15, Frequency, 3=Frequently | 1 | 1
  Aching Muscles, Cycle 2 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 13 | 14
  Aching Muscles, Cycle 2 Day 15, Frequency, 4=Almost constantly | 1 | 0
  Aching Muscles, Cycle 3 Day 1, Severity, 0=None: number analyzed (Participants) | 9 | 8
  Aching Muscles, Cycle 3 Day 1, Severity, 0=None | 1 | 0
  Aching Muscles, Cycle 3 Day 1, Severity, 1=Mild: number analyzed (Participants) | 9 | 8
  Aching Muscles, Cycle 3 Day 1, Severity, 1=Mild | 5 | 6
  Aching Muscles, Cycle 3 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 9 | 8
  Aching Muscles, Cycle 3 Day 1, Severity, 2=Moderate | 1 | 1
  Aching Muscles, Cycle 3 Day 1, Severity, 3=Severe: number analyzed (Participants) | 9 | 8
  Aching Muscles, Cycle 3 Day 1, Severity, 3=Severe | 1 | 1
  Aching Muscles, Cycle 3 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 9 | 8
  Aching Muscles, Cycle 3 Day 1, Severity, 4=Very severe | 1 | 0
  Aching Muscles, Cycle 3 Day 1, Frequency, 0=Never: number analyzed (Participants) | 14 | 14
  Aching Muscles, Cycle 3 Day 1, Frequency, 0=Never | 5 | 6
  Aching Muscles, Cycle 3 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 14
  Aching Muscles, Cycle 3 Day 1, Frequency, 1=Rarely | 5 | 5
  Aching Muscles, Cycle 3 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 14
  Aching Muscles, Cycle 3 Day 1, Frequency, 2=Occasionally | 2 | 1
  Aching Muscles, Cycle 3 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 14
  Aching Muscles, Cycle 3 Day 1, Frequency, 3=Frequently | 1 | 1
  Aching Muscles, Cycle 3 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 14
  Aching Muscles, Cycle 3 Day 1, Frequency, 4=Almost constantly | 1 | 1
  Aching Muscles, Cycle 3 Day 8, Severity, 0=None: number analyzed (Participants) | 6 | 5
  Aching Muscles, Cycle 3 Day 8, Severity, 0=None | 0 | 0
  Aching Muscles, Cycle 3 Day 8, Severity, 1=Mild: number analyzed (Participants) | 6 | 5
  Aching Muscles, Cycle 3 Day 8, Severity, 1=Mild | 1 | 2
  Aching Muscles, Cycle 3 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 6 | 5
  Aching Muscles, Cycle 3 Day 8, Severity, 2=Moderate | 2 | 2
  Aching Muscles, Cycle 3 Day 8, Severity, 3=Severe: number analyzed (Participants) | 6 | 5
  Aching Muscles, Cycle 3 Day 8, Severity, 3=Severe | 3 | 1
  Aching Muscles, Cycle 3 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 6 | 5
  Aching Muscles, Cycle 3 Day 8, Severity, 4=Very severe | 0 | 0
  Aching Muscles, Cycle 3 Day 8, Frequency, 0=Never: number analyzed (Participants) | 10 | 10
  Aching Muscles, Cycle 3 Day 8, Frequency, 0=Never | 4 | 5
  Aching Muscles, Cycle 3 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 10 | 10
  Aching Muscles, Cycle 3 Day 8, Frequency, 1=Rarely | 1 | 2
  Aching Muscles, Cycle 3 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 10 | 10
  Aching Muscles, Cycle 3 Day 8, Frequency, 2=Occasionally | 2 | 2
  Aching Muscles, Cycle 3 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 10 | 10
  Aching Muscles, Cycle 3 Day 8, Frequency, 3=Frequently | 3 | 1
  Aching Muscles, Cycle 3 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 10 | 10
  Aching Muscles, Cycle 3 Day 8, Frequency, 4=Almost constantly | 0 | 0
  Aching Muscles, Cycle 3 Day 15, Severity, 0=None: number analyzed (Participants) | 3 | 3
  Aching Muscles, Cycle 3 Day 15, Severity, 0=None | 1 | 0
  Aching Muscles, Cycle 3 Day 15, Severity, 1=Mild: number analyzed (Participants) | 3 | 3
  Aching Muscles, Cycle 3 Day 15, Severity, 1=Mild | 1 | 3
  Aching Muscles, Cycle 3 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 3 | 3
  Aching Muscles, Cycle 3 Day 15, Severity, 2=Moderate | 1 | 0
  Aching Muscles, Cycle 3 Day 15, Severity, 3=Severe: number analyzed (Participants) | 3 | 3
  Aching Muscles, Cycle 3 Day 15, Severity, 3=Severe | 0 | 0
  Aching Muscles, Cycle 3 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 3 | 3
  Aching Muscles, Cycle 3 Day 15, Severity, 4=Very severe | 0 | 0
  Aching Muscles, Cycle 3 Day 15, Frequency, 0=Never: number analyzed (Participants) | 5 | 7
  Aching Muscles, Cycle 3 Day 15, Frequency, 0=Never | 2 | 4
  Aching Muscles, Cycle 3 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 5 | 7
  Aching Muscles, Cycle 3 Day 15, Frequency, 1=Rarely | 1 | 2
  Aching Muscles, Cycle 3 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 5 | 7
  Aching Muscles, Cycle 3 Day 15, Frequency, 2=Occasionally | 1 | 1
  Aching Muscles, Cycle 3 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 5 | 7
  Aching Muscles, Cycle 3 Day 15, Frequency, 3=Frequently | 1 | 0
  Aching Muscles, Cycle 3 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 5 | 7
  Aching Muscles, Cycle 3 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Aching Muscles, Pre-IDS Evaluation, Severity, 0=None: number analyzed (Participants) | 1 | 0
  Aching Muscles, Pre-IDS Evaluation, Severity, 0=None | 0 |
  Aching Muscles, Pre-IDS Evaluation, Severity, 1=Mild: number analyzed (Participants) | 1 | 0
  Aching Muscles, Pre-IDS Evaluation, Severity, 1=Mild | 1 |
  Aching Muscles, Pre-IDS Evaluation, Severity, 2=Moderate: number analyzed (Participants) | 1 | 0
  Aching Muscles, Pre-IDS Evaluation, Severity, 2=Moderate | 0 |
  Aching Muscles, Pre-IDS Evaluation, Severity, 3=Severe: number analyzed (Participants) | 1 | 0
  Aching Muscles, Pre-IDS Evaluation, Severity, 3=Severe | 0 |
  Aching Muscles, Pre-IDS Evaluation, Severity, 4=Very severe: number analyzed (Participants) | 1 | 0
  Aching Muscles, Pre-IDS Evaluation, Severity, 4=Very severe | 0 |
  Aching Muscles, Pre-IDS Evaluation, Frequency, 0=Never: number analyzed (Participants) | 2 | 1
  Aching Muscles, Pre-IDS Evaluation, Frequency, 0=Never | 1 | 1
  Aching Muscles, Pre-IDS Evaluation, Frequency, 1=Rarely: number analyzed (Participants) | 2 | 1
  Aching Muscles, Pre-IDS Evaluation, Frequency, 1=Rarely | 1 | 0
  Aching Muscles, Pre-IDS Evaluation, Frequency, 2=Occasionally: number analyzed (Participants) | 2 | 1
  Aching Muscles, Pre-IDS Evaluation, Frequency, 2=Occasionally | 0 | 0
  Aching Muscles, Pre-IDS Evaluation, Frequency, 3=Frequently: number analyzed (Participants) | 2 | 1
  Aching Muscles, Pre-IDS Evaluation, Frequency, 3=Frequently | 0 | 0
  Aching Muscles, Pre-IDS Evaluation, Frequency, 4=Almost constantly: number analyzed (Participants) | 2 | 1
  Aching Muscles, Pre-IDS Evaluation, Frequency, 4=Almost constantly | 0 | 0
  Aching Muscles, End Of Treatment, Severity, 0=None: number analyzed (Participants) | 0 | 4
  Aching Muscles, End Of Treatment, Severity, 0=None |  | 0
  Aching Muscles, End Of Treatment, Severity, 1=Mild: number analyzed (Participants) | 0 | 4
  Aching Muscles, End Of Treatment, Severity, 1=Mild |  | 4
  Aching Muscles, End Of Treatment, Severity, 2=Moderate: number analyzed (Participants) | 0 | 4
  Aching Muscles, End Of Treatment, Severity, 2=Moderate |  | 0
  Aching Muscles, End Of Treatment, Severity, 3=Severe: number analyzed (Participants) | 0 | 4
  Aching Muscles, End Of Treatment, Severity, 3=Severe |  | 0
  Aching Muscles, End Of Treatment, Severity, 4=Very severe: number analyzed (Participants) | 0 | 4
  Aching Muscles, End Of Treatment, Severity, 4=Very severe |  | 0
  Aching Muscles, End Of Treatment, Frequency, 0=Never: number analyzed (Participants) | 0 | 5
  Aching Muscles, End Of Treatment, Frequency, 0=Never |  | 1
  Aching Muscles, End Of Treatment, Frequency, 1=Rarely: number analyzed (Participants) | 0 | 5
  Aching Muscles, End Of Treatment, Frequency, 1=Rarely |  | 4
  Aching Muscles, End Of Treatment, Frequency, 2=Occasionally: number analyzed (Participants) | 0 | 5
  Aching Muscles, End Of Treatment, Frequency, 2=Occasionally |  | 0
  Aching Muscles, End Of Treatment, Frequency, 3=Frequently: number analyzed (Participants) | 0 | 5
  Aching Muscles, End Of Treatment, Frequency, 3=Frequently |  | 0
  Aching Muscles, End Of Treatment, Frequency, 4=Almost constantly: number analyzed (Participants) | 0 | 5
  Aching Muscles, End Of Treatment, Frequency, 4=Almost constantly |  | 0
  Aching Joints, Baseline, Severity, 0=None: number analyzed (Participants) | 5 | 6
  Aching Joints, Baseline, Severity, 0=None | 0 | 0
  Aching Joints, Baseline, Severity, 1=Mild: number analyzed (Participants) | 5 | 6
  Aching Joints, Baseline, Severity, 1=Mild | 3 | 3
  Aching Joints, Baseline, Severity, 2=Moderate: number analyzed (Participants) | 5 | 6
  Aching Joints, Baseline, Severity, 2=Moderate | 1 | 1
  Aching Joints, Baseline, Severity, 3=Severe: number analyzed (Participants) | 5 | 6
  Aching Joints, Baseline, Severity, 3=Severe | 1 | 2
  Aching Joints, Baseline, Severity, 4=Very severe: number analyzed (Participants) | 5 | 6
  Aching Joints, Baseline, Severity, 4=Very severe | 0 | 0
  Aching Joints, Baseline, Frequency, 0=Never: number analyzed (Participants) | 14 | 17
  Aching Joints, Baseline, Frequency, 0=Never | 9 | 11
  Aching Joints, Baseline, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 17
  Aching Joints, Baseline, Frequency, 1=Rarely | 3 | 3
  Aching Joints, Baseline, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 17
  Aching Joints, Baseline, Frequency, 2=Occasionally | 1 | 1
  Aching Joints, Baseline, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 17
  Aching Joints, Baseline, Frequency, 3=Frequently | 1 | 1
  Aching Joints, Baseline, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 17
  Aching Joints, Baseline, Frequency, 4=Almost constantly | 0 | 1
  Aching Joints, Cycle 1 Day 8, Severity, 0=None: number analyzed (Participants) | 8 | 3
  Aching Joints, Cycle 1 Day 8, Severity, 0=None | 0 | 0
  Aching Joints, Cycle 1 Day 8, Severity, 1=Mild: number analyzed (Participants) | 8 | 3
  Aching Joints, Cycle 1 Day 8, Severity, 1=Mild | 3 | 1
  Aching Joints, Cycle 1 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 8 | 3
  Aching Joints, Cycle 1 Day 8, Severity, 2=Moderate | 1 | 1
  Aching Joints, Cycle 1 Day 8, Severity, 3=Severe: number analyzed (Participants) | 8 | 3
  Aching Joints, Cycle 1 Day 8, Severity, 3=Severe | 3 | 1
  Aching Joints, Cycle 1 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 8 | 3
  Aching Joints, Cycle 1 Day 8, Severity, 4=Very severe | 1 | 0
  Aching Joints, Cycle 1 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 15
  Aching Joints, Cycle 1 Day 8, Frequency, 0=Never | 3 | 12
  Aching Joints, Cycle 1 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 15
  Aching Joints, Cycle 1 Day 8, Frequency, 1=Rarely | 4 | 0
  Aching Joints, Cycle 1 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 15
  Aching Joints, Cycle 1 Day 8, Frequency, 2=Occasionally | 0 | 2
  Aching Joints, Cycle 1 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 15
  Aching Joints, Cycle 1 Day 8, Frequency, 3=Frequently | 2 | 0
  Aching Joints, Cycle 1 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 15
  Aching Joints, Cycle 1 Day 8, Frequency, 4=Almost constantly | 2 | 1
  Aching Joints, Cycle 1 Day 15, Severity, 0=None: number analyzed (Participants) | 7 | 5
  Aching Joints, Cycle 1 Day 15, Severity, 0=None | 0 | 0
  Aching Joints, Cycle 1 Day 15, Severity, 1=Mild: number analyzed (Participants) | 7 | 5
  Aching Joints, Cycle 1 Day 15, Severity, 1=Mild | 4 | 3
  Aching Joints, Cycle 1 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 7 | 5
  Aching Joints, Cycle 1 Day 15, Severity, 2=Moderate | 2 | 2
  Aching Joints, Cycle 1 Day 15, Severity, 3=Severe: number analyzed (Participants) | 7 | 5
  Aching Joints, Cycle 1 Day 15, Severity, 3=Severe | 0 | 0
  Aching Joints, Cycle 1 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 7 | 5
  Aching Joints, Cycle 1 Day 15, Severity, 4=Very severe | 1 | 0
  Aching Joints, Cycle 1 Day 15, Frequency, 0=Never: number analyzed (Participants) | 14 | 13
  Aching Joints, Cycle 1 Day 15, Frequency, 0=Never | 7 | 8
  Aching Joints, Cycle 1 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 13
  Aching Joints, Cycle 1 Day 15, Frequency, 1=Rarely | 4 | 3
  Aching Joints, Cycle 1 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 13
  Aching Joints, Cycle 1 Day 15, Frequency, 2=Occasionally | 2 | 2
  Aching Joints, Cycle 1 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 13
  Aching Joints, Cycle 1 Day 15, Frequency, 3=Frequently | 0 | 0
  Aching Joints, Cycle 1 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 13
  Aching Joints, Cycle 1 Day 15, Frequency, 4=Almost constantly | 1 | 0
  Aching Joints, Cycle 2 Day 1, Severity, 0=None: number analyzed (Participants) | 6 | 6
  Aching Joints, Cycle 2 Day 1, Severity, 0=None | 1 | 1
  Aching Joints, Cycle 2 Day 1, Severity, 1=Mild: number analyzed (Participants) | 6 | 6
  Aching Joints, Cycle 2 Day 1, Severity, 1=Mild | 4 | 1
  Aching Joints, Cycle 2 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 6 | 6
  Aching Joints, Cycle 2 Day 1, Severity, 2=Moderate | 1 | 3
  Aching Joints, Cycle 2 Day 1, Severity, 3=Severe: number analyzed (Participants) | 6 | 6
  Aching Joints, Cycle 2 Day 1, Severity, 3=Severe | 0 | 1
  Aching Joints, Cycle 2 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 6 | 6
  Aching Joints, Cycle 2 Day 1, Severity, 4=Very severe | 0 | 0
  Aching Joints, Cycle 2 Day 1, Frequency, 0=Never: number analyzed (Participants) | 11 | 14
  Aching Joints, Cycle 2 Day 1, Frequency, 0=Never | 5 | 8
  Aching Joints, Cycle 2 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 14
  Aching Joints, Cycle 2 Day 1, Frequency, 1=Rarely | 4 | 2
  Aching Joints, Cycle 2 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 14
  Aching Joints, Cycle 2 Day 1, Frequency, 2=Occasionally | 1 | 3
  Aching Joints, Cycle 2 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 14
  Aching Joints, Cycle 2 Day 1, Frequency, 3=Frequently | 1 | 1
  Aching Joints, Cycle 2 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 14
  Aching Joints, Cycle 2 Day 1, Frequency, 4=Almost constantly | 0 | 0
  Aching Joints, Cycle 2 Day 8, Severity, 0=None: number analyzed (Participants) | 10 | 4
  Aching Joints, Cycle 2 Day 8, Severity, 0=None | 1 | 0
  Aching Joints, Cycle 2 Day 8, Severity, 1=Mild: number analyzed (Participants) | 10 | 4
  Aching Joints, Cycle 2 Day 8, Severity, 1=Mild | 2 | 3
  Aching Joints, Cycle 2 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 10 | 4
  Aching Joints, Cycle 2 Day 8, Severity, 2=Moderate | 4 | 0
  Aching Joints, Cycle 2 Day 8, Severity, 3=Severe: number analyzed (Participants) | 10 | 4
  Aching Joints, Cycle 2 Day 8, Severity, 3=Severe | 2 | 1
  Aching Joints, Cycle 2 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 10 | 4
  Aching Joints, Cycle 2 Day 8, Severity, 4=Very severe | 1 | 0
  Aching Joints, Cycle 2 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 11
  Aching Joints, Cycle 2 Day 8, Frequency, 0=Never | 1 | 7
  Aching Joints, Cycle 2 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 11
  Aching Joints, Cycle 2 Day 8, Frequency, 1=Rarely | 3 | 2
  Aching Joints, Cycle 2 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 11
  Aching Joints, Cycle 2 Day 8, Frequency, 2=Occasionally | 4 | 1
  Aching Joints, Cycle 2 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 11
  Aching Joints, Cycle 2 Day 8, Frequency, 3=Frequently | 2 | 1
  Aching Joints, Cycle 2 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 11
  Aching Joints, Cycle 2 Day 8, Frequency, 4=Almost constantly | 1 | 0
  Aching Joints, Cycle 2 Day 15, Severity, 0=None: number analyzed (Participants) | 10 | 5
  Aching Joints, Cycle 2 Day 15, Severity, 0=None | 2 | 0
  Aching Joints, Cycle 2 Day 15, Severity, 1=Mild: number analyzed (Participants) | 10 | 5
  Aching Joints, Cycle 2 Day 15, Severity, 1=Mild | 5 | 3
  Aching Joints, Cycle 2 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 10 | 5
  Aching Joints, Cycle 2 Day 15, Severity, 2=Moderate | 2 | 1
  Aching Joints, Cycle 2 Day 15, Severity, 3=Severe: number analyzed (Participants) | 10 | 5
  Aching Joints, Cycle 2 Day 15, Severity, 3=Severe | 0 | 1
  Aching Joints, Cycle 2 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 10 | 5
  Aching Joints, Cycle 2 Day 15, Severity, 4=Very severe | 1 | 0
  Aching Joints, Cycle 2 Day 15, Frequency, 0=Never: number analyzed (Participants) | 13 | 14
  Aching Joints, Cycle 2 Day 15, Frequency, 0=Never | 3 | 9
  Aching Joints, Cycle 2 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 13 | 14
  Aching Joints, Cycle 2 Day 15, Frequency, 1=Rarely | 5 | 3
  Aching Joints, Cycle 2 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 13 | 14
  Aching Joints, Cycle 2 Day 15, Frequency, 2=Occasionally | 3 | 1
  Aching Joints, Cycle 2 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 13 | 14
  Aching Joints, Cycle 2 Day 15, Frequency, 3=Frequently | 1 | 1
  Aching Joints, Cycle 2 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 13 | 14
  Aching Joints, Cycle 2 Day 15, Frequency, 4=Almost constantly | 1 | 0
  Aching Joints, Cycle 3 Day 1, Severity, 0=None: number analyzed (Participants) | 8 | 6
  Aching Joints, Cycle 3 Day 1, Severity, 0=None | 0 | 1
  Aching Joints, Cycle 3 Day 1, Severity, 1=Mild: number analyzed (Participants) | 8 | 6
  Aching Joints, Cycle 3 Day 1, Severity, 1=Mild | 3 | 3
  Aching Joints, Cycle 3 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 8 | 6
  Aching Joints, Cycle 3 Day 1, Severity, 2=Moderate | 4 | 1
  Aching Joints, Cycle 3 Day 1, Severity, 3=Severe: number analyzed (Participants) | 8 | 6
  Aching Joints, Cycle 3 Day 1, Severity, 3=Severe | 1 | 1
  Aching Joints, Cycle 3 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 8 | 6
  Aching Joints, Cycle 3 Day 1, Severity, 4=Very severe | 0 | 0
  Aching Joints, Cycle 3 Day 1, Frequency, 0=Never: number analyzed (Participants) | 14 | 14
  Aching Joints, Cycle 3 Day 1, Frequency, 0=Never | 6 | 8
  Aching Joints, Cycle 3 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 14
  Aching Joints, Cycle 3 Day 1, Frequency, 1=Rarely | 3 | 4
  Aching Joints, Cycle 3 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 14
  Aching Joints, Cycle 3 Day 1, Frequency, 2=Occasionally | 3 | 0
  Aching Joints, Cycle 3 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 14
  Aching Joints, Cycle 3 Day 1, Frequency, 3=Frequently | 2 | 1
  Aching Joints, Cycle 3 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 14
  Aching Joints, Cycle 3 Day 1, Frequency, 4=Almost constantly | 0 | 1
  Aching Joints, Cycle 3 Day 8, Severity, 0=None: number analyzed (Participants) | 6 | 5
  Aching Joints, Cycle 3 Day 8, Severity, 0=None | 1 | 0
  Aching Joints, Cycle 3 Day 8, Severity, 1=Mild: number analyzed (Participants) | 6 | 5
  Aching Joints, Cycle 3 Day 8, Severity, 1=Mild | 0 | 4
  Aching Joints, Cycle 3 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 6 | 5
  Aching Joints, Cycle 3 Day 8, Severity, 2=Moderate | 2 | 0
  Aching Joints, Cycle 3 Day 8, Severity, 3=Severe: number analyzed (Participants) | 6 | 5
  Aching Joints, Cycle 3 Day 8, Severity, 3=Severe | 3 | 1
  Aching Joints, Cycle 3 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 6 | 5
  Aching Joints, Cycle 3 Day 8, Severity, 4=Very severe | 0 | 0
  Aching Joints, Cycle 3 Day 8, Frequency, 0=Never: number analyzed (Participants) | 10 | 10
  Aching Joints, Cycle 3 Day 8, Frequency, 0=Never | 4 | 5
  Aching Joints, Cycle 3 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 10 | 10
  Aching Joints, Cycle 3 Day 8, Frequency, 1=Rarely | 1 | 3
  Aching Joints, Cycle 3 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 10 | 10
  Aching Joints, Cycle 3 Day 8, Frequency, 2=Occasionally | 0 | 1
  Aching Joints, Cycle 3 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 10 | 10
  Aching Joints, Cycle 3 Day 8, Frequency, 3=Frequently | 4 | 1
  Aching Joints, Cycle 3 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 10 | 10
  Aching Joints, Cycle 3 Day 8, Frequency, 4=Almost constantly | 1 | 0
  Aching Joints, Cycle 3 Day 15, Severity, 0=None: number analyzed (Participants) | 4 | 2
  Aching Joints, Cycle 3 Day 15, Severity, 0=None | 1 | 0
  Aching Joints, Cycle 3 Day 15, Severity, 1=Mild: number analyzed (Participants) | 4 | 2
  Aching Joints, Cycle 3 Day 15, Severity, 1=Mild | 1 | 2
  Aching Joints, Cycle 3 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 4 | 2
  Aching Joints, Cycle 3 Day 15, Severity, 2=Moderate | 1 | 0
  Aching Joints, Cycle 3 Day 15, Severity, 3=Severe: number analyzed (Participants) | 4 | 2
  Aching Joints, Cycle 3 Day 15, Severity, 3=Severe | 1 | 0
  Aching Joints, Cycle 3 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 4 | 2
  Aching Joints, Cycle 3 Day 15, Severity, 4=Very severe | 0 | 0
  Aching Joints, Cycle 3 Day 15, Frequency, 0=Never: number analyzed (Participants) | 5 | 7
  Aching Joints, Cycle 3 Day 15, Frequency, 0=Never | 1 | 5
  Aching Joints, Cycle 3 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 5 | 7
  Aching Joints, Cycle 3 Day 15, Frequency, 1=Rarely | 2 | 1
  Aching Joints, Cycle 3 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 5 | 7
  Aching Joints, Cycle 3 Day 15, Frequency, 2=Occasionally | 1 | 1
  Aching Joints, Cycle 3 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 5 | 7
  Aching Joints, Cycle 3 Day 15, Frequency, 3=Frequently | 0 | 0
  Aching Joints, Cycle 3 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 5 | 7
  Aching Joints, Cycle 3 Day 15, Frequency, 4=Almost constantly | 1 | 0
  Aching Joints, Pre-IDS Evaluation, Frequency, 0=Never: number analyzed (Participants) | 2 | 1
  Aching Joints, Pre-IDS Evaluation, Frequency, 0=Never | 2 | 1
  Aching Joints, Pre-IDS Evaluation, Frequency, 1=Rarely: number analyzed (Participants) | 2 | 1
  Aching Joints, Pre-IDS Evaluation, Frequency, 1=Rarely | 0 | 0
  Aching Joints, Pre-IDS Evaluation, Frequency, 2=Occasionally: number analyzed (Participants) | 2 | 1
  Aching Joints, Pre-IDS Evaluation, Frequency, 2=Occasionally | 0 | 0
  Aching Joints, Pre-IDS Evaluation, Frequency, 3=Frequently: number analyzed (Participants) | 2 | 1
  Aching Joints, Pre-IDS Evaluation, Frequency, 3=Frequently | 0 | 0
  Aching Joints, Pre-IDS Evaluation, Frequency, 4=Almost constantly: number analyzed (Participants) | 2 | 1
  Aching Joints, Pre-IDS Evaluation, Frequency, 4=Almost constantly | 0 | 0
  Aching Joints, End Of Treatment, Severity, 0=None: number analyzed (Participants) | 0 | 2
  Aching Joints, End Of Treatment, Severity, 0=None |  | 1
  Aching Joints, End Of Treatment, Severity, 1=Mild: number analyzed (Participants) | 0 | 2
  Aching Joints, End Of Treatment, Severity, 1=Mild |  | 1
  Aching Joints, End Of Treatment, Severity, 2=Moderate: number analyzed (Participants) | 0 | 2
  Aching Joints, End Of Treatment, Severity, 2=Moderate |  | 0
  Aching Joints, End Of Treatment, Severity, 3=Severe: number analyzed (Participants) | 0 | 2
  Aching Joints, End Of Treatment, Severity, 3=Severe |  | 0
  Aching Joints, End Of Treatment, Severity, 4=Very severe: number analyzed (Participants) | 0 | 2
  Aching Joints, End Of Treatment, Severity, 4=Very severe |  | 0
  Aching Joints, End Of Treatment, Frequency, 0=Never: number analyzed (Participants) | 0 | 5
  Aching Joints, End Of Treatment, Frequency, 0=Never |  | 3
  Aching Joints, End Of Treatment, Frequency, 1=Rarely: number analyzed (Participants) | 0 | 5
  Aching Joints, End Of Treatment, Frequency, 1=Rarely |  | 2
  Aching Joints, End Of Treatment, Frequency, 2=Occasionally: number analyzed (Participants) | 0 | 5
  Aching Joints, End Of Treatment, Frequency, 2=Occasionally |  | 0
  Aching Joints, End Of Treatment, Frequency, 3=Frequently: number analyzed (Participants) | 0 | 5
  Aching Joints, End Of Treatment, Frequency, 3=Frequently |  | 0
  Aching Joints, End Of Treatment, Frequency, 4=Almost constantly: number analyzed (Participants) | 0 | 5
  Aching Joints, End Of Treatment, Frequency, 4=Almost constantly |  | 0
  Fatigue/Lack of Energy, Baseline, Severity, 0=None: number analyzed (Participants) | 14 | 17
  Fatigue/Lack of Energy, Baseline, Severity, 0=None | 3 | 3
  Fatigue/Lack of Energy, Baseline, Severity, 1=Mild: number analyzed (Participants) | 14 | 17
  Fatigue/Lack of Energy, Baseline, Severity, 1=Mild | 2 | 5
  Fatigue/Lack of Energy, Baseline, Severity, 2=Moderate: number analyzed (Participants) | 14 | 17
  Fatigue/Lack of Energy, Baseline, Severity, 2=Moderate | 8 | 6
  Fatigue/Lack of Energy, Baseline, Severity, 3=Severe: number analyzed (Participants) | 14 | 17
  Fatigue/Lack of Energy, Baseline, Severity, 3=Severe | 1 | 3
  Fatigue/Lack of Energy, Baseline, Severity, 4=Very severe: number analyzed (Participants) | 14 | 17
  Fatigue/Lack of Energy, Baseline, Severity, 4=Very severe | 0 | 0
  Fatigue/Lack of Energy, Cycle 1 Day 8, Severity, 0=None: number analyzed (Participants) | 11 | 15
  Fatigue/Lack of Energy, Cycle 1 Day 8, Severity, 0=None | 0 | 0
  Fatigue/Lack of Energy, Cycle 1 Day 8, Severity, 1=Mild: number analyzed (Participants) | 11 | 15
  Fatigue/Lack of Energy, Cycle 1 Day 8, Severity, 1=Mild | 1 | 7
  Fatigue/Lack of Energy, Cycle 1 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 11 | 15
  Fatigue/Lack of Energy, Cycle 1 Day 8, Severity, 2=Moderate | 3 | 2
  Fatigue/Lack of Energy, Cycle 1 Day 8, Severity, 3=Severe: number analyzed (Participants) | 11 | 15
  Fatigue/Lack of Energy, Cycle 1 Day 8, Severity, 3=Severe | 7 | 6
  Fatigue/Lack of Energy, Cycle 1 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 11 | 15
  Fatigue/Lack of Energy, Cycle 1 Day 8, Severity, 4=Very severe | 0 | 0
  Fatigue/Lack of Energy, Cycle 1 Day 15, Severity, 0=None: number analyzed (Participants) | 14 | 13
  Fatigue/Lack of Energy, Cycle 1 Day 15, Severity, 0=None | 2 | 2
  Fatigue/Lack of Energy, Cycle 1 Day 15, Severity, 1=Mild: number analyzed (Participants) | 14 | 13
  Fatigue/Lack of Energy, Cycle 1 Day 15, Severity, 1=Mild | 5 | 3
  Fatigue/Lack of Energy, Cycle 1 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 14 | 13
  Fatigue/Lack of Energy, Cycle 1 Day 15, Severity, 2=Moderate | 5 | 4
  Fatigue/Lack of Energy, Cycle 1 Day 15, Severity, 3=Severe: number analyzed (Participants) | 14 | 13
  Fatigue/Lack of Energy, Cycle 1 Day 15, Severity, 3=Severe | 1 | 4
  Fatigue/Lack of Energy, Cycle 1 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 14 | 13
  Fatigue/Lack of Energy, Cycle 1 Day 15, Severity, 4=Very severe | 1 | 0
  Fatigue/Lack of Energy, Cycle 2 Day 1, Severity, 0=None: number analyzed (Participants) | 11 | 14
  Fatigue/Lack of Energy, Cycle 2 Day 1, Severity, 0=None | 3 | 1
  Fatigue/Lack of Energy, Cycle 2 Day 1, Severity, 1=Mild: number analyzed (Participants) | 11 | 14
  Fatigue/Lack of Energy, Cycle 2 Day 1, Severity, 1=Mild | 4 | 6
  Fatigue/Lack of Energy, Cycle 2 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 11 | 14
  Fatigue/Lack of Energy, Cycle 2 Day 1, Severity, 2=Moderate | 4 | 5
  Fatigue/Lack of Energy, Cycle 2 Day 1, Severity, 3=Severe: number analyzed (Participants) | 11 | 14
  Fatigue/Lack of Energy, Cycle 2 Day 1, Severity, 3=Severe | 0 | 2
  Fatigue/Lack of Energy, Cycle 2 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 11 | 14
  Fatigue/Lack of Energy, Cycle 2 Day 1, Severity, 4=Very severe | 0 | 0
  Fatigue/Lack of Energy, Cycle 2 Day 8, Severity, 0=None: number analyzed (Participants) | 11 | 11
  Fatigue/Lack of Energy, Cycle 2 Day 8, Severity, 0=None | 0 | 1
  Fatigue/Lack of Energy, Cycle 2 Day 8, Severity, 1=Mild: number analyzed (Participants) | 11 | 11
  Fatigue/Lack of Energy, Cycle 2 Day 8, Severity, 1=Mild | 4 | 6
  Fatigue/Lack of Energy, Cycle 2 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 11 | 11
  Fatigue/Lack of Energy, Cycle 2 Day 8, Severity, 2=Moderate | 3 | 3
  Fatigue/Lack of Energy, Cycle 2 Day 8, Severity, 3=Severe: number analyzed (Participants) | 11 | 11
  Fatigue/Lack of Energy, Cycle 2 Day 8, Severity, 3=Severe | 2 | 1
  Fatigue/Lack of Energy, Cycle 2 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 11 | 11
  Fatigue/Lack of Energy, Cycle 2 Day 8, Severity, 4=Very severe | 2 | 0
  Fatigue/Lack of Energy, Cycle 2 Day 15, Severity, 0=None: number analyzed (Participants) | 13 | 14
  Fatigue/Lack of Energy, Cycle 2 Day 15, Severity, 0=None | 2 | 2
  Fatigue/Lack of Energy, Cycle 2 Day 15, Severity, 1=Mild: number analyzed (Participants) | 13 | 14
  Fatigue/Lack of Energy, Cycle 2 Day 15, Severity, 1=Mild | 2 | 5
  Fatigue/Lack of Energy, Cycle 2 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 13 | 14
  Fatigue/Lack of Energy, Cycle 2 Day 15, Severity, 2=Moderate | 7 | 6
  Fatigue/Lack of Energy, Cycle 2 Day 15, Severity, 3=Severe: number analyzed (Participants) | 13 | 14
  Fatigue/Lack of Energy, Cycle 2 Day 15, Severity, 3=Severe | 2 | 1
  Fatigue/Lack of Energy, Cycle 2 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 13 | 14
  Fatigue/Lack of Energy, Cycle 2 Day 15, Severity, 4=Very severe | 0 | 0
  Fatigue/Lack of Energy, Cycle 3 Day 1, Severity, 0=None: number analyzed (Participants) | 14 | 14
  Fatigue/Lack of Energy, Cycle 3 Day 1, Severity, 0=None | 2 | 2
  Fatigue/Lack of Energy, Cycle 3 Day 1, Severity, 1=Mild: number analyzed (Participants) | 14 | 14
  Fatigue/Lack of Energy, Cycle 3 Day 1, Severity, 1=Mild | 7 | 6
  Fatigue/Lack of Energy, Cycle 3 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 14 | 14
  Fatigue/Lack of Energy, Cycle 3 Day 1, Severity, 2=Moderate | 5 | 4
  Fatigue/Lack of Energy, Cycle 3 Day 1, Severity, 3=Severe: number analyzed (Participants) | 14 | 14
  Fatigue/Lack of Energy, Cycle 3 Day 1, Severity, 3=Severe | 0 | 2
  Fatigue/Lack of Energy, Cycle 3 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 14 | 14
  Fatigue/Lack of Energy, Cycle 3 Day 1, Severity, 4=Very severe | 0 | 0
  Fatigue/Lack of Energy, Cycle 3 Day 8, Severity, 0=None: number analyzed (Participants) | 10 | 10
  Fatigue/Lack of Energy, Cycle 3 Day 8, Severity, 0=None | 0 | 1
  Fatigue/Lack of Energy, Cycle 3 Day 8, Severity, 1=Mild: number analyzed (Participants) | 10 | 10
  Fatigue/Lack of Energy, Cycle 3 Day 8, Severity, 1=Mild | 2 | 3
  Fatigue/Lack of Energy, Cycle 3 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 10 | 10
  Fatigue/Lack of Energy, Cycle 3 Day 8, Severity, 2=Moderate | 3 | 5
  Fatigue/Lack of Energy, Cycle 3 Day 8, Severity, 3=Severe: number analyzed (Participants) | 10 | 10
  Fatigue/Lack of Energy, Cycle 3 Day 8, Severity, 3=Severe | 3 | 1
  Fatigue/Lack of Energy, Cycle 3 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 10 | 10
  Fatigue/Lack of Energy, Cycle 3 Day 8, Severity, 4=Very severe | 2 | 0
  Fatigue/Lack of Energy, Cycle 3 Day 15, Severity, 0=None: number analyzed (Participants) | 5 | 7
  Fatigue/Lack of Energy, Cycle 3 Day 15, Severity, 0=None | 0 | 0
  Fatigue/Lack of Energy, Cycle 3 Day 15, Severity, 1=Mild: number analyzed (Participants) | 5 | 7
  Fatigue/Lack of Energy, Cycle 3 Day 15, Severity, 1=Mild | 4 | 3
  Fatigue/Lack of Energy, Cycle 3 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 5 | 7
  Fatigue/Lack of Energy, Cycle 3 Day 15, Severity, 2=Moderate | 1 | 4
  Fatigue/Lack of Energy, Cycle 3 Day 15, Severity, 3=Severe: number analyzed (Participants) | 5 | 7
  Fatigue/Lack of Energy, Cycle 3 Day 15, Severity, 3=Severe | 0 | 0
  Fatigue/Lack of Energy, Cycle 3 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 5 | 7
  Fatigue/Lack of Energy, Cycle 3 Day 15, Severity, 4=Very severe | 0 | 0
  Fatigue/Lack of Energy, Pre-IDS Evaluation, Severity, 0=None: number analyzed (Participants) | 2 | 1
  Fatigue/Lack of Energy, Pre-IDS Evaluation, Severity, 0=None | 1 | 0
  Fatigue/Lack of Energy, Pre-IDS Evaluation, Severity, 1=Mild: number analyzed (Participants) | 2 | 1
  Fatigue/Lack of Energy, Pre-IDS Evaluation, Severity, 1=Mild | 1 | 0
  Fatigue/Lack of Energy, Pre-IDS Evaluation, Severity, 2=Moderate: number analyzed (Participants) | 2 | 1
  Fatigue/Lack of Energy, Pre-IDS Evaluation, Severity, 2=Moderate | 0 | 1
  Fatigue/Lack of Energy, Pre-IDS Evaluation, Severity, 3=Severe: number analyzed (Participants) | 2 | 1
  Fatigue/Lack of Energy, Pre-IDS Evaluation, Severity, 3=Severe | 0 | 0
  Fatigue/Lack of Energy, Pre-IDS Evaluation, Severity, 4=Very severe: number analyzed (Participants) | 2 | 1
  Fatigue/Lack of Energy, Pre-IDS Evaluation, Severity, 4=Very severe | 0 | 0
  Fatigue/Lack of Energy, End Of Treatment, Severity, 0=None: number analyzed (Participants) | 0 | 5
  Fatigue/Lack of Energy, End Of Treatment, Severity, 0=None |  | 2
  Fatigue/Lack of Energy, End Of Treatment, Severity, 1=Mild: number analyzed (Participants) | 0 | 5
  Fatigue/Lack of Energy, End Of Treatment, Severity, 1=Mild |  | 2
  Fatigue/Lack of Energy, End Of Treatment, Severity, 2=Moderate: number analyzed (Participants) | 0 | 5
  Fatigue/Lack of Energy, End Of Treatment, Severity, 2=Moderate |  | 1
  Fatigue/Lack of Energy, End Of Treatment, Severity, 3=Severe: number analyzed (Participants) | 0 | 5
  Fatigue/Lack of Energy, End Of Treatment, Severity, 3=Severe |  | 0
  Fatigue/Lack of Energy, End Of Treatment, Severity, 4=Very severe: number analyzed (Participants) | 0 | 5
  Fatigue/Lack of Energy, End Of Treatment, Severity, 4=Very severe |  | 0
  Anxiety, Baseline, Severity, 0=None: number analyzed (Participants) | 10 | 12
  Anxiety, Baseline, Severity, 0=None | 1 | 1
  Anxiety, Baseline, Severity, 1=Mild: number analyzed (Participants) | 10 | 12
  Anxiety, Baseline, Severity, 1=Mild | 5 | 6
  Anxiety, Baseline, Severity, 2=Moderate: number analyzed (Participants) | 10 | 12
  Anxiety, Baseline, Severity, 2=Moderate | 4 | 3
  Anxiety, Baseline, Severity, 3=Severe: number analyzed (Participants) | 10 | 12
  Anxiety, Baseline, Severity, 3=Severe | 0 | 1
  Anxiety, Baseline, Severity, 4=Very severe: number analyzed (Participants) | 10 | 12
  Anxiety, Baseline, Severity, 4=Very severe | 0 | 1
  Anxiety, Baseline, Frequency, 0=Never: number analyzed (Participants) | 14 | 17
  Anxiety, Baseline, Frequency, 0=Never | 4 | 5
  Anxiety, Baseline, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 17
  Anxiety, Baseline, Frequency, 1=Rarely | 4 | 6
  Anxiety, Baseline, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 17
  Anxiety, Baseline, Frequency, 2=Occasionally | 5 | 4
  Anxiety, Baseline, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 17
  Anxiety, Baseline, Frequency, 3=Frequently | 0 | 0
  Anxiety, Baseline, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 17
  Anxiety, Baseline, Frequency, 4=Almost constantly | 1 | 2
  Anxiety, Cycle 1 Day 8, Severity, 0=None: number analyzed (Participants) | 8 | 8
  Anxiety, Cycle 1 Day 8, Severity, 0=None | 2 | 0
  Anxiety, Cycle 1 Day 8, Severity, 1=Mild: number analyzed (Participants) | 8 | 8
  Anxiety, Cycle 1 Day 8, Severity, 1=Mild | 4 | 3
  Anxiety, Cycle 1 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 8 | 8
  Anxiety, Cycle 1 Day 8, Severity, 2=Moderate | 1 | 3
  Anxiety, Cycle 1 Day 8, Severity, 3=Severe: number analyzed (Participants) | 8 | 8
  Anxiety, Cycle 1 Day 8, Severity, 3=Severe | 1 | 2
  Anxiety, Cycle 1 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 8 | 8
  Anxiety, Cycle 1 Day 8, Severity, 4=Very severe | 0 | 0
  Anxiety, Cycle 1 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 15
  Anxiety, Cycle 1 Day 8, Frequency, 0=Never | 3 | 7
  Anxiety, Cycle 1 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 15
  Anxiety, Cycle 1 Day 8, Frequency, 1=Rarely | 6 | 3
  Anxiety, Cycle 1 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 15
  Anxiety, Cycle 1 Day 8, Frequency, 2=Occasionally | 1 | 2
  Anxiety, Cycle 1 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 15
  Anxiety, Cycle 1 Day 8, Frequency, 3=Frequently | 1 | 2
  Anxiety, Cycle 1 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 15
  Anxiety, Cycle 1 Day 8, Frequency, 4=Almost constantly | 0 | 1
  Anxiety, Cycle 1 Day 15, Severity, 0=None: number analyzed (Participants) | 7 | 7
  Anxiety, Cycle 1 Day 15, Severity, 0=None | 1 | 0
  Anxiety, Cycle 1 Day 15, Severity, 1=Mild: number analyzed (Participants) | 7 | 7
  Anxiety, Cycle 1 Day 15, Severity, 1=Mild | 4 | 3
  Anxiety, Cycle 1 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 7 | 7
  Anxiety, Cycle 1 Day 15, Severity, 2=Moderate | 2 | 2
  Anxiety, Cycle 1 Day 15, Severity, 3=Severe: number analyzed (Participants) | 7 | 7
  Anxiety, Cycle 1 Day 15, Severity, 3=Severe | 0 | 2
  Anxiety, Cycle 1 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 7 | 7
  Anxiety, Cycle 1 Day 15, Severity, 4=Very severe | 0 | 0
  Anxiety, Cycle 1 Day 15, Frequency, 0=Never: number analyzed (Participants) | 14 | 13
  Anxiety, Cycle 1 Day 15, Frequency, 0=Never | 7 | 6
  Anxiety, Cycle 1 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 13
  Anxiety, Cycle 1 Day 15, Frequency, 1=Rarely | 6 | 3
  Anxiety, Cycle 1 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 13
  Anxiety, Cycle 1 Day 15, Frequency, 2=Occasionally | 0 | 3
  Anxiety, Cycle 1 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 13
  Anxiety, Cycle 1 Day 15, Frequency, 3=Frequently | 1 | 1
  Anxiety, Cycle 1 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 13
  Anxiety, Cycle 1 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Anxiety, Cycle 2 Day 1, Severity, 0=None: number analyzed (Participants) | 6 | 8
  Anxiety, Cycle 2 Day 1, Severity, 0=None | 0 | 1
  Anxiety, Cycle 2 Day 1, Severity, 1=Mild: number analyzed (Participants) | 6 | 8
  Anxiety, Cycle 2 Day 1, Severity, 1=Mild | 4 | 6
  Anxiety, Cycle 2 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 6 | 8
  Anxiety, Cycle 2 Day 1, Severity, 2=Moderate | 2 | 0
  Anxiety, Cycle 2 Day 1, Severity, 3=Severe: number analyzed (Participants) | 6 | 8
  Anxiety, Cycle 2 Day 1, Severity, 3=Severe | 0 | 1
  Anxiety, Cycle 2 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 6 | 8
  Anxiety, Cycle 2 Day 1, Severity, 4=Very severe | 0 | 0
  Anxiety, Cycle 2 Day 1, Frequency, 0=Never: number analyzed (Participants) | 11 | 14
  Anxiety, Cycle 2 Day 1, Frequency, 0=Never | 5 | 6
  Anxiety, Cycle 2 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 14
  Anxiety, Cycle 2 Day 1, Frequency, 1=Rarely | 4 | 6
  Anxiety, Cycle 2 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 14
  Anxiety, Cycle 2 Day 1, Frequency, 2=Occasionally | 2 | 2
  Anxiety, Cycle 2 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 14
  Anxiety, Cycle 2 Day 1, Frequency, 3=Frequently | 0 | 0
  Anxiety, Cycle 2 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 14
  Anxiety, Cycle 2 Day 1, Frequency, 4=Almost constantly | 0 | 0
  Anxiety, Cycle 2 Day 8, Severity, 0=None: number analyzed (Participants) | 7 | 4
  Anxiety, Cycle 2 Day 8, Severity, 0=None | 1 | 0
  Anxiety, Cycle 2 Day 8, Severity, 1=Mild: number analyzed (Participants) | 7 | 4
  Anxiety, Cycle 2 Day 8, Severity, 1=Mild | 2 | 3
  Anxiety, Cycle 2 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 7 | 4
  Anxiety, Cycle 2 Day 8, Severity, 2=Moderate | 3 | 1
  Anxiety, Cycle 2 Day 8, Severity, 3=Severe: number analyzed (Participants) | 7 | 4
  Anxiety, Cycle 2 Day 8, Severity, 3=Severe | 1 | 0
  Anxiety, Cycle 2 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 7 | 4
  Anxiety, Cycle 2 Day 8, Severity, 4=Very severe | 0 | 0
  Anxiety, Cycle 2 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 11
  Anxiety, Cycle 2 Day 8, Frequency, 0=Never | 4 | 7
  Anxiety, Cycle 2 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 11
  Anxiety, Cycle 2 Day 8, Frequency, 1=Rarely | 2 | 3
  Anxiety, Cycle 2 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 11
  Anxiety, Cycle 2 Day 8, Frequency, 2=Occasionally | 4 | 1
  Anxiety, Cycle 2 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 11
  Anxiety, Cycle 2 Day 8, Frequency, 3=Frequently | 1 | 0
  Anxiety, Cycle 2 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 11
  Anxiety, Cycle 2 Day 8, Frequency, 4=Almost constantly | 0 | 0
  Anxiety, Cycle 2 Day 15, Severity, 0=None: number analyzed (Participants) | 8 | 6
  Anxiety, Cycle 2 Day 15, Severity, 0=None | 0 | 0
  Anxiety, Cycle 2 Day 15, Severity, 1=Mild: number analyzed (Participants) | 8 | 6
  Anxiety, Cycle 2 Day 15, Severity, 1=Mild | 4 | 3
  Anxiety, Cycle 2 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 8 | 6
  Anxiety, Cycle 2 Day 15, Severity, 2=Moderate | 4 | 2
  Anxiety, Cycle 2 Day 15, Severity, 3=Severe: number analyzed (Participants) | 8 | 6
  Anxiety, Cycle 2 Day 15, Severity, 3=Severe | 0 | 1
  Anxiety, Cycle 2 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 8 | 6
  Anxiety, Cycle 2 Day 15, Severity, 4=Very severe | 0 | 0
  Anxiety, Cycle 2 Day 15, Frequency, 0=Never: number analyzed (Participants) | 13 | 14
  Anxiety, Cycle 2 Day 15, Frequency, 0=Never | 5 | 8
  Anxiety, Cycle 2 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 13 | 14
  Anxiety, Cycle 2 Day 15, Frequency, 1=Rarely | 2 | 2
  Anxiety, Cycle 2 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 13 | 14
  Anxiety, Cycle 2 Day 15, Frequency, 2=Occasionally | 6 | 1
  Anxiety, Cycle 2 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 13 | 14
  Anxiety, Cycle 2 Day 15, Frequency, 3=Frequently | 0 | 2
  Anxiety, Cycle 2 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 13 | 14
  Anxiety, Cycle 2 Day 15, Frequency, 4=Almost constantly | 0 | 1
  Anxiety, Cycle 3 Day 1, Severity, 0=None: number analyzed (Participants) | 9 | 8
  Anxiety, Cycle 3 Day 1, Severity, 0=None | 1 | 0
  Anxiety, Cycle 3 Day 1, Severity, 1=Mild: number analyzed (Participants) | 9 | 8
  Anxiety, Cycle 3 Day 1, Severity, 1=Mild | 7 | 5
  Anxiety, Cycle 3 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 9 | 8
  Anxiety, Cycle 3 Day 1, Severity, 2=Moderate | 1 | 3
  Anxiety, Cycle 3 Day 1, Severity, 3=Severe: number analyzed (Participants) | 9 | 8
  Anxiety, Cycle 3 Day 1, Severity, 3=Severe | 0 | 0
  Anxiety, Cycle 3 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 9 | 8
  Anxiety, Cycle 3 Day 1, Severity, 4=Very severe | 0 | 0
  Anxiety, Cycle 3 Day 1, Frequency, 0=Never: number analyzed (Participants) | 14 | 14
  Anxiety, Cycle 3 Day 1, Frequency, 0=Never | 5 | 6
  Anxiety, Cycle 3 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 14
  Anxiety, Cycle 3 Day 1, Frequency, 1=Rarely | 5 | 5
  Anxiety, Cycle 3 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 14
  Anxiety, Cycle 3 Day 1, Frequency, 2=Occasionally | 4 | 2
  Anxiety, Cycle 3 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 14
  Anxiety, Cycle 3 Day 1, Frequency, 3=Frequently | 0 | 1
  Anxiety, Cycle 3 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 14
  Anxiety, Cycle 3 Day 1, Frequency, 4=Almost constantly | 0 | 0
  Anxiety, Cycle 3 Day 8, Severity, 0=None: number analyzed (Participants) | 5 | 6
  Anxiety, Cycle 3 Day 8, Severity, 0=None | 1 | 0
  Anxiety, Cycle 3 Day 8, Severity, 1=Mild: number analyzed (Participants) | 5 | 6
  Anxiety, Cycle 3 Day 8, Severity, 1=Mild | 1 | 3
  Anxiety, Cycle 3 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 5 | 6
  Anxiety, Cycle 3 Day 8, Severity, 2=Moderate | 3 | 3
  Anxiety, Cycle 3 Day 8, Severity, 3=Severe: number analyzed (Participants) | 5 | 6
  Anxiety, Cycle 3 Day 8, Severity, 3=Severe | 0 | 0
  Anxiety, Cycle 3 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 5 | 6
  Anxiety, Cycle 3 Day 8, Severity, 4=Very severe | 0 | 0
  Anxiety, Cycle 3 Day 8, Frequency, 0=Never: number analyzed (Participants) | 10 | 10
  Anxiety, Cycle 3 Day 8, Frequency, 0=Never | 5 | 4
  Anxiety, Cycle 3 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 10 | 10
  Anxiety, Cycle 3 Day 8, Frequency, 1=Rarely | 1 | 3
  Anxiety, Cycle 3 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 10 | 10
  Anxiety, Cycle 3 Day 8, Frequency, 2=Occasionally | 2 | 2
  Anxiety, Cycle 3 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 10 | 10
  Anxiety, Cycle 3 Day 8, Frequency, 3=Frequently | 2 | 1
  Anxiety, Cycle 3 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 10 | 10
  Anxiety, Cycle 3 Day 8, Frequency, 4=Almost constantly | 0 | 0
  Anxiety, Cycle 3 Day 15, Severity, 0=None: number analyzed (Participants) | 4 | 4
  Anxiety, Cycle 3 Day 15, Severity, 0=None | 1 | 0
  Anxiety, Cycle 3 Day 15, Severity, 1=Mild: number analyzed (Participants) | 4 | 4
  Anxiety, Cycle 3 Day 15, Severity, 1=Mild | 1 | 4
  Anxiety, Cycle 3 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 4 | 4
  Anxiety, Cycle 3 Day 15, Severity, 2=Moderate | 2 | 0
  Anxiety, Cycle 3 Day 15, Severity, 3=Severe: number analyzed (Participants) | 4 | 4
  Anxiety, Cycle 3 Day 15, Severity, 3=Severe | 0 | 0
  Anxiety, Cycle 3 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 4 | 4
  Anxiety, Cycle 3 Day 15, Severity, 4=Very severe | 0 | 0
  Anxiety, Cycle 3 Day 15, Frequency, 0=Never: number analyzed (Participants) | 5 | 7
  Anxiety, Cycle 3 Day 15, Frequency, 0=Never | 1 | 3
  Anxiety, Cycle 3 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 5 | 7
  Anxiety, Cycle 3 Day 15, Frequency, 1=Rarely | 2 | 3
  Anxiety, Cycle 3 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 5 | 7
  Anxiety, Cycle 3 Day 15, Frequency, 2=Occasionally | 2 | 1
  Anxiety, Cycle 3 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 5 | 7
  Anxiety, Cycle 3 Day 15, Frequency, 3=Frequently | 0 | 0
  Anxiety, Cycle 3 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 5 | 7
  Anxiety, Cycle 3 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Anxiety, Pre-IDS Evaluation, Severity, 0=None: number analyzed (Participants) | 0 | 1
  Anxiety, Pre-IDS Evaluation, Severity, 0=None |  | 0
  Anxiety, Pre-IDS Evaluation, Severity, 1=Mild: number analyzed (Participants) | 0 | 1
  Anxiety, Pre-IDS Evaluation, Severity, 1=Mild |  | 1
  Anxiety, Pre-IDS Evaluation, Severity, 2=Moderate: number analyzed (Participants) | 0 | 1
  Anxiety, Pre-IDS Evaluation, Severity, 2=Moderate |  | 0
  Anxiety, Pre-IDS Evaluation, Severity, 3=Severe: number analyzed (Participants) | 0 | 1
  Anxiety, Pre-IDS Evaluation, Severity, 3=Severe |  | 0
  Anxiety, Pre-IDS Evaluation, Severity, 4=Very severe: number analyzed (Participants) | 0 | 1
  Anxiety, Pre-IDS Evaluation, Severity, 4=Very severe |  | 0
  Anxiety, Pre-IDS Evaluation, Frequency, 0=Never: number analyzed (Participants) | 2 | 1
  Anxiety, Pre-IDS Evaluation, Frequency, 0=Never | 2 | 0
  Anxiety, Pre-IDS Evaluation, Frequency, 1=Rarely: number analyzed (Participants) | 2 | 1
  Anxiety, Pre-IDS Evaluation, Frequency, 1=Rarely | 0 | 1
  Anxiety, Pre-IDS Evaluation, Frequency, 2=Occasionally: number analyzed (Participants) | 2 | 1
  Anxiety, Pre-IDS Evaluation, Frequency, 2=Occasionally | 0 | 0
  Anxiety, Pre-IDS Evaluation, Frequency, 3=Frequently: number analyzed (Participants) | 2 | 1
  Anxiety, Pre-IDS Evaluation, Frequency, 3=Frequently | 0 | 0
  Anxiety, Pre-IDS Evaluation, Frequency, 4=Almost constantly: number analyzed (Participants) | 2 | 1
  Anxiety, Pre-IDS Evaluation, Frequency, 4=Almost constantly | 0 | 0
  Anxiety, End Of Treatment, Severity, 0=None: number analyzed (Participants) | 0 | 4
  Anxiety, End Of Treatment, Severity, 0=None |  | 1
  Anxiety, End Of Treatment, Severity, 1=Mild: number analyzed (Participants) | 0 | 4
  Anxiety, End Of Treatment, Severity, 1=Mild |  | 2
  Anxiety, End Of Treatment, Severity, 2=Moderate: number analyzed (Participants) | 0 | 4
  Anxiety, End Of Treatment, Severity, 2=Moderate |  | 1
  Anxiety, End Of Treatment, Severity, 3=Severe: number analyzed (Participants) | 0 | 4
  Anxiety, End Of Treatment, Severity, 3=Severe |  | 0
  Anxiety, End Of Treatment, Severity, 4=Very severe: number analyzed (Participants) | 0 | 4
  Anxiety, End Of Treatment, Severity, 4=Very severe |  | 0
  Anxiety, End Of Treatment, Frequency, 0=Never: number analyzed (Participants) | 0 | 5
  Anxiety, End Of Treatment, Frequency, 0=Never |  | 1
  Anxiety, End Of Treatment, Frequency, 1=Rarely: number analyzed (Participants) | 0 | 5
  Anxiety, End Of Treatment, Frequency, 1=Rarely |  | 2
  Anxiety, End Of Treatment, Frequency, 2=Occasionally: number analyzed (Participants) | 0 | 5
  Anxiety, End Of Treatment, Frequency, 2=Occasionally |  | 2
  Anxiety, End Of Treatment, Frequency, 3=Frequently: number analyzed (Participants) | 0 | 5
  Anxiety, End Of Treatment, Frequency, 3=Frequently |  | 0
  Anxiety, End Of Treatment, Frequency, 4=Almost constantly: number analyzed (Participants) | 0 | 5
  Anxiety, End Of Treatment, Frequency, 4=Almost constantly |  | 0
  Sad or Unhappy Feelings, Baseline, Severity, 0=None: number analyzed (Participants) | 12 | 13
  Sad or Unhappy Feelings, Baseline, Severity, 0=None | 1 | 2
  Sad or Unhappy Feelings, Baseline, Severity, 1=Mild: number analyzed (Participants) | 12 | 13
  Sad or Unhappy Feelings, Baseline, Severity, 1=Mild | 8 | 5
  Sad or Unhappy Feelings, Baseline, Severity, 2=Moderate: number analyzed (Participants) | 12 | 13
  Sad or Unhappy Feelings, Baseline, Severity, 2=Moderate | 3 | 4
  Sad or Unhappy Feelings, Baseline, Severity, 3=Severe: number analyzed (Participants) | 12 | 13
  Sad or Unhappy Feelings, Baseline, Severity, 3=Severe | 0 | 1
  Sad or Unhappy Feelings, Baseline, Severity, 4=Very severe: number analyzed (Participants) | 12 | 13
  Sad or Unhappy Feelings, Baseline, Severity, 4=Very severe | 0 | 1
  Sad or Unhappy Feelings, Baseline, Frequency, 0=Never: number analyzed (Participants) | 14 | 17
  Sad or Unhappy Feelings, Baseline, Frequency, 0=Never | 2 | 4
  Sad or Unhappy Feelings, Baseline, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 17
  Sad or Unhappy Feelings, Baseline, Frequency, 1=Rarely | 4 | 6
  Sad or Unhappy Feelings, Baseline, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 17
  Sad or Unhappy Feelings, Baseline, Frequency, 2=Occasionally | 8 | 5
  Sad or Unhappy Feelings, Baseline, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 17
  Sad or Unhappy Feelings, Baseline, Frequency, 3=Frequently | 0 | 1
  Sad or Unhappy Feelings, Baseline, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 17
  Sad or Unhappy Feelings, Baseline, Frequency, 4=Almost constantly | 0 | 1
  Sad or Unhappy Feelings, Cycle 1 Day 8, Severity, 0=None: number analyzed (Participants) | 10 | 10
  Sad or Unhappy Feelings, Cycle 1 Day 8, Severity, 0=None | 1 | 1
  Sad or Unhappy Feelings, Cycle 1 Day 8, Severity, 1=Mild: number analyzed (Participants) | 10 | 10
  Sad or Unhappy Feelings, Cycle 1 Day 8, Severity, 1=Mild | 6 | 5
  Sad or Unhappy Feelings, Cycle 1 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 10 | 10
  Sad or Unhappy Feelings, Cycle 1 Day 8, Severity, 2=Moderate | 2 | 2
  Sad or Unhappy Feelings, Cycle 1 Day 8, Severity, 3=Severe: number analyzed (Participants) | 10 | 10
  Sad or Unhappy Feelings, Cycle 1 Day 8, Severity, 3=Severe | 1 | 2
  Sad or Unhappy Feelings, Cycle 1 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 10 | 10
  Sad or Unhappy Feelings, Cycle 1 Day 8, Severity, 4=Very severe | 0 | 0
  Sad or Unhappy Feelings, Cycle 1 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 15
  Sad or Unhappy Feelings, Cycle 1 Day 8, Frequency, 0=Never | 1 | 5
  Sad or Unhappy Feelings, Cycle 1 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 15
  Sad or Unhappy Feelings, Cycle 1 Day 8, Frequency, 1=Rarely | 5 | 6
  Sad or Unhappy Feelings, Cycle 1 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 15
  Sad or Unhappy Feelings, Cycle 1 Day 8, Frequency, 2=Occasionally | 4 | 3
  Sad or Unhappy Feelings, Cycle 1 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 15
  Sad or Unhappy Feelings, Cycle 1 Day 8, Frequency, 3=Frequently | 1 | 0
  Sad or Unhappy Feelings, Cycle 1 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 15
  Sad or Unhappy Feelings, Cycle 1 Day 8, Frequency, 4=Almost constantly | 0 | 1
  Sad or Unhappy Feelings, Cycle 1 Day 15, Severity, 0=None: number analyzed (Participants) | 8 | 9
  Sad or Unhappy Feelings, Cycle 1 Day 15, Severity, 0=None | 1 | 0
  Sad or Unhappy Feelings, Cycle 1 Day 15, Severity, 1=Mild: number analyzed (Participants) | 8 | 9
  Sad or Unhappy Feelings, Cycle 1 Day 15, Severity, 1=Mild | 5 | 5
  Sad or Unhappy Feelings, Cycle 1 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 8 | 9
  Sad or Unhappy Feelings, Cycle 1 Day 15, Severity, 2=Moderate | 2 | 2
  Sad or Unhappy Feelings, Cycle 1 Day 15, Severity, 3=Severe: number analyzed (Participants) | 8 | 9
  Sad or Unhappy Feelings, Cycle 1 Day 15, Severity, 3=Severe | 0 | 2
  Sad or Unhappy Feelings, Cycle 1 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 8 | 9
  Sad or Unhappy Feelings, Cycle 1 Day 15, Severity, 4=Very severe | 0 | 0
  Sad or Unhappy Feelings, Cycle 1 Day 15, Frequency, 0=Never: number analyzed (Participants) | 14 | 13
  Sad or Unhappy Feelings, Cycle 1 Day 15, Frequency, 0=Never | 6 | 4
  Sad or Unhappy Feelings, Cycle 1 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 13
  Sad or Unhappy Feelings, Cycle 1 Day 15, Frequency, 1=Rarely | 5 | 5
  Sad or Unhappy Feelings, Cycle 1 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 13
  Sad or Unhappy Feelings, Cycle 1 Day 15, Frequency, 2=Occasionally | 2 | 3
  Sad or Unhappy Feelings, Cycle 1 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 13
  Sad or Unhappy Feelings, Cycle 1 Day 15, Frequency, 3=Frequently | 1 | 1
  Sad or Unhappy Feelings, Cycle 1 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 13
  Sad or Unhappy Feelings, Cycle 1 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Sad or Unhappy Feelings, Cycle 2 Day 1, Severity, 0=None: number analyzed (Participants) | 5 | 9
  Sad or Unhappy Feelings, Cycle 2 Day 1, Severity, 0=None | 0 | 1
  Sad or Unhappy Feelings, Cycle 2 Day 1, Severity, 1=Mild: number analyzed (Participants) | 5 | 9
  Sad or Unhappy Feelings, Cycle 2 Day 1, Severity, 1=Mild | 3 | 7
  Sad or Unhappy Feelings, Cycle 2 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 5 | 9
  Sad or Unhappy Feelings, Cycle 2 Day 1, Severity, 2=Moderate | 2 | 1
  Sad or Unhappy Feelings, Cycle 2 Day 1, Severity, 3=Severe: number analyzed (Participants) | 5 | 9
  Sad or Unhappy Feelings, Cycle 2 Day 1, Severity, 3=Severe | 0 | 0
  Sad or Unhappy Feelings, Cycle 2 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 5 | 9
  Sad or Unhappy Feelings, Cycle 2 Day 1, Severity, 4=Very severe | 0 | 0
  Sad or Unhappy Feelings, Cycle 2 Day 1, Frequency, 0=Never: number analyzed (Participants) | 11 | 14
  Sad or Unhappy Feelings, Cycle 2 Day 1, Frequency, 0=Never | 6 | 5
  Sad or Unhappy Feelings, Cycle 2 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 14
  Sad or Unhappy Feelings, Cycle 2 Day 1, Frequency, 1=Rarely | 1 | 8
  Sad or Unhappy Feelings, Cycle 2 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 14
  Sad or Unhappy Feelings, Cycle 2 Day 1, Frequency, 2=Occasionally | 4 | 1
  Sad or Unhappy Feelings, Cycle 2 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 14
  Sad or Unhappy Feelings, Cycle 2 Day 1, Frequency, 3=Frequently | 0 | 0
  Sad or Unhappy Feelings, Cycle 2 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 14
  Sad or Unhappy Feelings, Cycle 2 Day 1, Frequency, 4=Almost constantly | 0 | 0
  Sad or Unhappy Feelings, Cycle 2 Day 8, Severity, 0=None: number analyzed (Participants) | 7 | 8
  Sad or Unhappy Feelings, Cycle 2 Day 8, Severity, 0=None | 1 | 2
  Sad or Unhappy Feelings, Cycle 2 Day 8, Severity, 1=Mild: number analyzed (Participants) | 7 | 8
  Sad or Unhappy Feelings, Cycle 2 Day 8, Severity, 1=Mild | 3 | 6
  Sad or Unhappy Feelings, Cycle 2 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 7 | 8
  Sad or Unhappy Feelings, Cycle 2 Day 8, Severity, 2=Moderate | 2 | 0
  Sad or Unhappy Feelings, Cycle 2 Day 8, Severity, 3=Severe: number analyzed (Participants) | 7 | 8
  Sad or Unhappy Feelings, Cycle 2 Day 8, Severity, 3=Severe | 0 | 0
  Sad or Unhappy Feelings, Cycle 2 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 7 | 8
  Sad or Unhappy Feelings, Cycle 2 Day 8, Severity, 4=Very severe | 1 | 0
  Sad or Unhappy Feelings, Cycle 2 Day 8, Frequency, 0=Never: number analyzed (Participants) | 11 | 11
  Sad or Unhappy Feelings, Cycle 2 Day 8, Frequency, 0=Never | 4 | 3
  Sad or Unhappy Feelings, Cycle 2 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 11 | 11
  Sad or Unhappy Feelings, Cycle 2 Day 8, Frequency, 1=Rarely | 3 | 8
  Sad or Unhappy Feelings, Cycle 2 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 11 | 11
  Sad or Unhappy Feelings, Cycle 2 Day 8, Frequency, 2=Occasionally | 2 | 0
  Sad or Unhappy Feelings, Cycle 2 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 11 | 11
  Sad or Unhappy Feelings, Cycle 2 Day 8, Frequency, 3=Frequently | 1 | 0
  Sad or Unhappy Feelings, Cycle 2 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 11 | 11
  Sad or Unhappy Feelings, Cycle 2 Day 8, Frequency, 4=Almost constantly | 1 | 0
  Sad or Unhappy Feelings, Cycle 2 Day 15, Severity, 0=None: number analyzed (Participants) | 9 | 11
  Sad or Unhappy Feelings, Cycle 2 Day 15, Severity, 0=None | 0 | 3
  Sad or Unhappy Feelings, Cycle 2 Day 15, Severity, 1=Mild: number analyzed (Participants) | 9 | 11
  Sad or Unhappy Feelings, Cycle 2 Day 15, Severity, 1=Mild | 5 | 6
  Sad or Unhappy Feelings, Cycle 2 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 9 | 11
  Sad or Unhappy Feelings, Cycle 2 Day 15, Severity, 2=Moderate | 4 | 2
  Sad or Unhappy Feelings, Cycle 2 Day 15, Severity, 3=Severe: number analyzed (Participants) | 9 | 11
  Sad or Unhappy Feelings, Cycle 2 Day 15, Severity, 3=Severe | 0 | 0
  Sad or Unhappy Feelings, Cycle 2 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 9 | 11
  Sad or Unhappy Feelings, Cycle 2 Day 15, Severity, 4=Very severe | 0 | 0
  Sad or Unhappy Feelings, Cycle 2 Day 15, Frequency, 0=Never: number analyzed (Participants) | 13 | 14
  Sad or Unhappy Feelings, Cycle 2 Day 15, Frequency, 0=Never | 4 | 3
  Sad or Unhappy Feelings, Cycle 2 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 13 | 14
  Sad or Unhappy Feelings, Cycle 2 Day 15, Frequency, 1=Rarely | 4 | 7
  Sad or Unhappy Feelings, Cycle 2 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 13 | 14
  Sad or Unhappy Feelings, Cycle 2 Day 15, Frequency, 2=Occasionally | 4 | 3
  Sad or Unhappy Feelings, Cycle 2 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 13 | 14
  Sad or Unhappy Feelings, Cycle 2 Day 15, Frequency, 3=Frequently | 1 | 1
  Sad or Unhappy Feelings, Cycle 2 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 13 | 14
  Sad or Unhappy Feelings, Cycle 2 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Sad or Unhappy Feelings, Cycle 3 Day 1, Severity, 0=None: number analyzed (Participants) | 8 | 10
  Sad or Unhappy Feelings, Cycle 3 Day 1, Severity, 0=None | 1 | 1
  Sad or Unhappy Feelings, Cycle 3 Day 1, Severity, 1=Mild: number analyzed (Participants) | 8 | 10
  Sad or Unhappy Feelings, Cycle 3 Day 1, Severity, 1=Mild | 6 | 8
  Sad or Unhappy Feelings, Cycle 3 Day 1, Severity, 2=Moderate: number analyzed (Participants) | 8 | 10
  Sad or Unhappy Feelings, Cycle 3 Day 1, Severity, 2=Moderate | 1 | 1
  Sad or Unhappy Feelings, Cycle 3 Day 1, Severity, 3=Severe: number analyzed (Participants) | 8 | 10
  Sad or Unhappy Feelings, Cycle 3 Day 1, Severity, 3=Severe | 0 | 0
  Sad or Unhappy Feelings, Cycle 3 Day 1, Severity, 4=Very severe: number analyzed (Participants) | 8 | 10
  Sad or Unhappy Feelings, Cycle 3 Day 1, Severity, 4=Very severe | 0 | 0
  Sad or Unhappy Feelings, Cycle 3 Day 1, Frequency, 0=Never: number analyzed (Participants) | 14 | 14
  Sad or Unhappy Feelings, Cycle 3 Day 1, Frequency, 0=Never | 6 | 4
  Sad or Unhappy Feelings, Cycle 3 Day 1, Frequency, 1=Rarely: number analyzed (Participants) | 14 | 14
  Sad or Unhappy Feelings, Cycle 3 Day 1, Frequency, 1=Rarely | 6 | 9
  Sad or Unhappy Feelings, Cycle 3 Day 1, Frequency, 2=Occasionally: number analyzed (Participants) | 14 | 14
  Sad or Unhappy Feelings, Cycle 3 Day 1, Frequency, 2=Occasionally | 1 | 1
  Sad or Unhappy Feelings, Cycle 3 Day 1, Frequency, 3=Frequently: number analyzed (Participants) | 14 | 14
  Sad or Unhappy Feelings, Cycle 3 Day 1, Frequency, 3=Frequently | 1 | 0
  Sad or Unhappy Feelings, Cycle 3 Day 1, Frequency, 4=Almost constantly: number analyzed (Participants) | 14 | 14
  Sad or Unhappy Feelings, Cycle 3 Day 1, Frequency, 4=Almost constantly | 0 | 0
  Sad or Unhappy Feelings, Cycle 3 Day 8, Severity, 0=None: number analyzed (Participants) | 5 | 7
  Sad or Unhappy Feelings, Cycle 3 Day 8, Severity, 0=None | 2 | 1
  Sad or Unhappy Feelings, Cycle 3 Day 8, Severity, 1=Mild: number analyzed (Participants) | 5 | 7
  Sad or Unhappy Feelings, Cycle 3 Day 8, Severity, 1=Mild | 0 | 4
  Sad or Unhappy Feelings, Cycle 3 Day 8, Severity, 2=Moderate: number analyzed (Participants) | 5 | 7
  Sad or Unhappy Feelings, Cycle 3 Day 8, Severity, 2=Moderate | 2 | 2
  Sad or Unhappy Feelings, Cycle 3 Day 8, Severity, 3=Severe: number analyzed (Participants) | 5 | 7
  Sad or Unhappy Feelings, Cycle 3 Day 8, Severity, 3=Severe | 1 | 0
  Sad or Unhappy Feelings, Cycle 3 Day 8, Severity, 4=Very severe: number analyzed (Participants) | 5 | 7
  Sad or Unhappy Feelings, Cycle 3 Day 8, Severity, 4=Very severe | 0 | 0
  Sad or Unhappy Feelings, Cycle 3 Day 8, Frequency, 0=Never: number analyzed (Participants) | 10 | 10
  Sad or Unhappy Feelings, Cycle 3 Day 8, Frequency, 0=Never | 5 | 3
  Sad or Unhappy Feelings, Cycle 3 Day 8, Frequency, 1=Rarely: number analyzed (Participants) | 10 | 10
  Sad or Unhappy Feelings, Cycle 3 Day 8, Frequency, 1=Rarely | 2 | 5
  Sad or Unhappy Feelings, Cycle 3 Day 8, Frequency, 2=Occasionally: number analyzed (Participants) | 10 | 10
  Sad or Unhappy Feelings, Cycle 3 Day 8, Frequency, 2=Occasionally | 2 | 1
  Sad or Unhappy Feelings, Cycle 3 Day 8, Frequency, 3=Frequently: number analyzed (Participants) | 10 | 10
  Sad or Unhappy Feelings, Cycle 3 Day 8, Frequency, 3=Frequently | 1 | 1
  Sad or Unhappy Feelings, Cycle 3 Day 8, Frequency, 4=Almost constantly: number analyzed (Participants) | 10 | 10
  Sad or Unhappy Feelings, Cycle 3 Day 8, Frequency, 4=Almost constantly | 0 | 0
  Sad or Unhappy Feelings, Cycle 3 Day 15, Severity, 0=None: number analyzed (Participants) | 5 | 4
  Sad or Unhappy Feelings, Cycle 3 Day 15, Severity, 0=None | 1 | 0
  Sad or Unhappy Feelings, Cycle 3 Day 15, Severity, 1=Mild: number analyzed (Participants) | 5 | 4
  Sad or Unhappy Feelings, Cycle 3 Day 15, Severity, 1=Mild | 4 | 4
  Sad or Unhappy Feelings, Cycle 3 Day 15, Severity, 2=Moderate: number analyzed (Participants) | 5 | 4
  Sad or Unhappy Feelings, Cycle 3 Day 15, Severity, 2=Moderate | 0 | 0
  Sad or Unhappy Feelings, Cycle 3 Day 15, Severity, 3=Severe: number analyzed (Participants) | 5 | 4
  Sad or Unhappy Feelings, Cycle 3 Day 15, Severity, 3=Severe | 0 | 0
  Sad or Unhappy Feelings, Cycle 3 Day 15, Severity, 4=Very severe: number analyzed (Participants) | 5 | 4
  Sad or Unhappy Feelings, Cycle 3 Day 15, Severity, 4=Very severe | 0 | 0
  Sad or Unhappy Feelings, Cycle 3 Day 15, Frequency, 0=Never: number analyzed (Participants) | 5 | 7
  Sad or Unhappy Feelings, Cycle 3 Day 15, Frequency, 0=Never | 0 | 3
  Sad or Unhappy Feelings, Cycle 3 Day 15, Frequency, 1=Rarely: number analyzed (Participants) | 5 | 7
  Sad or Unhappy Feelings, Cycle 3 Day 15, Frequency, 1=Rarely | 4 | 3
  Sad or Unhappy Feelings, Cycle 3 Day 15, Frequency, 2=Occasionally: number analyzed (Participants) | 5 | 7
  Sad or Unhappy Feelings, Cycle 3 Day 15, Frequency, 2=Occasionally | 1 | 1
  Sad or Unhappy Feelings, Cycle 3 Day 15, Frequency, 3=Frequently: number analyzed (Participants) | 5 | 7
  Sad or Unhappy Feelings, Cycle 3 Day 15, Frequency, 3=Frequently | 0 | 0
  Sad or Unhappy Feelings, Cycle 3 Day 15, Frequency, 4=Almost constantly: number analyzed (Participants) | 5 | 7
  Sad or Unhappy Feelings, Cycle 3 Day 15, Frequency, 4=Almost constantly | 0 | 0
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Severity, 0=None: number analyzed (Participants) | 0 | 1
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Severity, 0=None |  | 0
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Severity, 1=Mild: number analyzed (Participants) | 0 | 1
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Severity, 1=Mild |  | 1
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Severity, 2=Moderate: number analyzed (Participants) | 0 | 1
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Severity, 2=Moderate |  | 0
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Severity, 3=Severe: number analyzed (Participants) | 0 | 1
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Severity, 3=Severe |  | 0
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Severity, 4=Very severe: number analyzed (Participants) | 0 | 1
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Severity, 4=Very severe |  | 0
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Frequency, 0=Never: number analyzed (Participants) | 2 | 1
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Frequency, 0=Never | 2 | 0
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Frequency, 1=Rarely: number analyzed (Participants) | 2 | 1
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Frequency, 1=Rarely | 0 | 0
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Frequency, 2=Occasionally: number analyzed (Participants) | 2 | 1
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Frequency, 2=Occasionally | 0 | 1
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Frequency, 3=Frequently: number analyzed (Participants) | 2 | 1
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Frequency, 3=Frequently | 0 | 0
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Frequency, 4=Almost constantly: number analyzed (Participants) | 2 | 1
  Sad or Unhappy Feelings, Pre-IDS Evaluation, Frequency, 4=Almost constantly | 0 | 0
  Sad or Unhappy Feelings, End Of Treatment, Severity, 0=None: number analyzed (Participants) | 0 | 2
  Sad or Unhappy Feelings, End Of Treatment, Severity, 0=None |  | 1
  Sad or Unhappy Feelings, End Of Treatment, Severity, 1=Mild: number analyzed (Participants) | 0 | 2
  Sad or Unhappy Feelings, End Of Treatment, Severity, 1=Mild |  | 1
  Sad or Unhappy Feelings, End Of Treatment, Severity, 2=Moderate: number analyzed (Participants) | 0 | 2
  Sad or Unhappy Feelings, End Of Treatment, Severity, 2=Moderate |  | 0
  Sad or Unhappy Feelings, End Of Treatment, Severity, 3=Severe: number analyzed (Participants) | 0 | 2
  Sad or Unhappy Feelings, End Of Treatment, Severity, 3=Severe |  | 0
  Sad or Unhappy Feelings, End Of Treatment, Severity, 4=Very severe: number analyzed (Participants) | 0 | 2
  Sad or Unhappy Feelings, End Of Treatment, Severity, 4=Very severe |  | 0
  Sad or Unhappy Feelings, End Of Treatment, Frequency, 0=Never: number analyzed (Participants) | 0 | 5
  Sad or Unhappy Feelings, End Of Treatment, Frequency, 0=Never |  | 3
  Sad or Unhappy Feelings, End Of Treatment, Frequency, 1=Rarely: number analyzed (Participants) | 0 | 5
  Sad or Unhappy Feelings, End Of Treatment, Frequency, 1=Rarely |  | 2
  Sad or Unhappy Feelings, End Of Treatment, Frequency, 2=Occasionally: number analyzed (Participants) | 0 | 5
  Sad or Unhappy Feelings, End Of Treatment, Frequency, 2=Occasionally |  | 0
  Sad or Unhappy Feelings, End Of Treatment, Frequency, 3=Frequently: number analyzed (Participants) | 0 | 5
  Sad or Unhappy Feelings, End Of Treatment, Frequency, 3=Frequently |  | 0
  Sad or Unhappy Feelings, End Of Treatment, Frequency, 4=Almost constantly: number analyzed (Participants) | 0 | 5
  Sad or Unhappy Feelings, End Of Treatment, Frequency, 4=Almost constantly |  | 0

7. Secondary Outcome: Number of Participants With Overall Side Effect Bother as Measured by Functional Assessment of Cancer Therapy - Item FACT-GP5
Description: The FACT-GP5 item is a single item from the FACT-G that assesses how bothersome the side effects of treatment are for participants with cancer. It evaluates the extent to which side effects of treatment are bothersome for cancer participants. This outcome is measured using a 5-category response scale, where responses include 0="Not at all," 1="A little bit," 2="Somewhat," 3="Quite a bit," and 4="Very much." A higher score on this measure indicates that the participant experiences a greater level of bother from the side effects of treatment.
Time Frame: Baseline (Predose), Day 8 and 15 of Cycle 1; Day 1, 8, and 15 of Cycle 2 and Cycle 3; Pre-IDS Evaluation, and End of Treatment (Up to approximately 154 weeks)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-taxane | Niraparib
Number analyzed (Participants) | 17 | 19
Participants
  Baseline, 0=Not at all: number analyzed (Participants) | 14 | 17
  Baseline, 0=Not at all | 4 | 4
  Baseline, 1=A little bit: number analyzed (Participants) | 14 | 17
  Baseline, 1=A little bit | 4 | 6
  Baseline, 2=Somewhat: number analyzed (Participants) | 14 | 17
  Baseline, 2=Somewhat | 1 | 7
  Baseline, 3=Quite a bit: number analyzed (Participants) | 14 | 17
  Baseline, 3=Quite a bit | 4 | 0
  Baseline, 4=Very much: number analyzed (Participants) | 14 | 17
  Baseline, 4=Very much | 1 | 0
  Cycle 1 Day 8, 0=Not at all: number analyzed (Participants) | 11 | 15
  Cycle 1 Day 8, 0=Not at all | 0 | 2
  Cycle 1 Day 8, 1=A little bit: number analyzed (Participants) | 11 | 15
  Cycle 1 Day 8, 1=A little bit | 2 | 5
  Cycle 1 Day 8, 2=Somewhat: number analyzed (Participants) | 11 | 15
  Cycle 1 Day 8, 2=Somewhat | 2 | 7
  Cycle 1 Day 8, 3=Quite a bit: number analyzed (Participants) | 11 | 15
  Cycle 1 Day 8, 3=Quite a bit | 6 | 1
  Cycle 1 Day 8, 4=Very much: number analyzed (Participants) | 11 | 15
  Cycle 1 Day 8, 4=Very much | 1 | 0
  Cycle 1 Day 15, 0=Not at all: number analyzed (Participants) | 14 | 14
  Cycle 1 Day 15, 0=Not at all | 4 | 5
  Cycle 1 Day 15, 1=A little bit: number analyzed (Participants) | 14 | 14
  Cycle 1 Day 15, 1=A little bit | 2 | 2
  Cycle 1 Day 15, 2=Somewhat: number analyzed (Participants) | 14 | 14
  Cycle 1 Day 15, 2=Somewhat | 4 | 7
  Cycle 1 Day 15, 3=Quite a bit: number analyzed (Participants) | 14 | 14
  Cycle 1 Day 15, 3=Quite a bit | 2 | 0
  Cycle 1 Day 15, 4=Very much: number analyzed (Participants) | 14 | 14
  Cycle 1 Day 15, 4=Very much | 2 | 0
  Cycle 2 Day 1, 0=Not at all: number analyzed (Participants) | 11 | 14
  Cycle 2 Day 1, 0=Not at all | 4 | 5
  Cycle 2 Day 1, 1=A little bit: number analyzed (Participants) | 11 | 14
  Cycle 2 Day 1, 1=A little bit | 4 | 2
  Cycle 2 Day 1, 2=Somewhat: number analyzed (Participants) | 11 | 14
  Cycle 2 Day 1, 2=Somewhat | 2 | 5
  Cycle 2 Day 1, 3=Quite a bit: number analyzed (Participants) | 11 | 14
  Cycle 2 Day 1, 3=Quite a bit | 1 | 2
  Cycle 2 Day 1, 4=Very much: number analyzed (Participants) | 11 | 14
  Cycle 2 Day 1, 4=Very much | 0 | 0
  Cycle 2 Day 8, 0=Not at all: number analyzed (Participants) | 11 | 12
  Cycle 2 Day 8, 0=Not at all | 1 | 3
  Cycle 2 Day 8, 1=A little bit: number analyzed (Participants) | 11 | 12
  Cycle 2 Day 8, 1=A little bit | 4 | 3
  Cycle 2 Day 8, 2=Somewhat: number analyzed (Participants) | 11 | 12
  Cycle 2 Day 8, 2=Somewhat | 3 | 6
  Cycle 2 Day 8, 3=Quite a bit: number analyzed (Participants) | 11 | 12
  Cycle 2 Day 8, 3=Quite a bit | 1 | 0
  Cycle 2 Day 8, 4=Very much: number analyzed (Participants) | 11 | 12
  Cycle 2 Day 8, 4=Very much | 2 | 0
  Cycle 2 Day 15, 0=Not at all: number analyzed (Participants) | 13 | 14
  Cycle 2 Day 15, 0=Not at all | 2 | 4
  Cycle 2 Day 15, 1=A little bit: number analyzed (Participants) | 13 | 14
  Cycle 2 Day 15, 1=A little bit | 3 | 5
  Cycle 2 Day 15, 2=Somewhat: number analyzed (Participants) | 13 | 14
  Cycle 2 Day 15, 2=Somewhat | 5 | 4
  Cycle 2 Day 15, 3=Quite a bit: number analyzed (Participants) | 13 | 14
  Cycle 2 Day 15, 3=Quite a bit | 2 | 1
  Cycle 2 Day 15, 4=Very much: number analyzed (Participants) | 13 | 14
  Cycle 2 Day 15, 4=Very much | 1 | 0
  Cycle 3 Day 1, 0=Not at all: number analyzed (Participants) | 14 | 14
  Cycle 3 Day 1, 0=Not at all | 1 | 4
  Cycle 3 Day 1, 1=A little bit: number analyzed (Participants) | 14 | 14
  Cycle 3 Day 1, 1=A little bit | 9 | 3
  Cycle 3 Day 1, 2=Somewhat: number analyzed (Participants) | 14 | 14
  Cycle 3 Day 1, 2=Somewhat | 4 | 6
  Cycle 3 Day 1, 3=Quite a bit: number analyzed (Participants) | 14 | 14
  Cycle 3 Day 1, 3=Quite a bit | 0 | 1
  Cycle 3 Day 1, 4=Very much: number analyzed (Participants) | 14 | 14
  Cycle 3 Day 1, 4=Very much | 0 | 0
  Cycle 3 Day 8, 0=Not at all: number analyzed (Participants) | 10 | 10
  Cycle 3 Day 8, 0=Not at all | 1 | 1
  Cycle 3 Day 8, 1=A little bit: number analyzed (Participants) | 10 | 10
  Cycle 3 Day 8, 1=A little bit | 3 | 3
  Cycle 3 Day 8, 2=Somewhat: number analyzed (Participants) | 10 | 10
  Cycle 3 Day 8, 2=Somewhat | 0 | 6
  Cycle 3 Day 8, 3=Quite a bit: number analyzed (Participants) | 10 | 10
  Cycle 3 Day 8, 3=Quite a bit | 5 | 0
  Cycle 3 Day 8, 4=Very much: number analyzed (Participants) | 10 | 10
  Cycle 3 Day 8, 4=Very much | 1 | 0
  Cycle 3 Day 15, 0=Not at all: number analyzed (Participants) | 5 | 7
  Cycle 3 Day 15, 0=Not at all | 0 | 2
  Cycle 3 Day 15, 1=A little bit: number analyzed (Participants) | 5 | 7
  Cycle 3 Day 15, 1=A little bit | 3 | 2
  Cycle 3 Day 15, 2=Somewhat: number analyzed (Participants) | 5 | 7
  Cycle 3 Day 15, 2=Somewhat | 1 | 3
  Cycle 3 Day 15, 3=Quite a bit: number analyzed (Participants) | 5 | 7
  Cycle 3 Day 15, 3=Quite a bit | 1 | 0
  Cycle 3 Day 15, 4=Very much: number analyzed (Participants) | 5 | 7
  Cycle 3 Day 15, 4=Very much | 0 | 0
  Pre-IDS Evaluation, 0=Not at all: number analyzed (Participants) | 15 | 7
  Pre-IDS Evaluation, 0=Not at all | 2 | 2
  Pre-IDS Evaluation, 1=A little bit: number analyzed (Participants) | 15 | 7
  Pre-IDS Evaluation, 1=A little bit | 7 | 1
  Pre-IDS Evaluation, 2=Somewhat: number analyzed (Participants) | 15 | 7
  Pre-IDS Evaluation, 2=Somewhat | 6 | 4
  Pre-IDS Evaluation, 3=Quite a bit: number analyzed (Participants) | 15 | 7
  Pre-IDS Evaluation, 3=Quite a bit | 0 | 0
  Pre-IDS Evaluation, 4=Very much: number analyzed (Participants) | 15 | 7
  Pre-IDS Evaluation, 4=Very much | 0 | 0
  End Of Treatment, 0=Not at all: number analyzed (Participants) | 0 | 5
  End Of Treatment, 0=Not at all |  | 2
  End Of Treatment, 1=A little bit: number analyzed (Participants) | 0 | 5
  End Of Treatment, 1=A little bit |  | 1
  End Of Treatment, 2=Somewhat: number analyzed (Participants) | 0 | 5
  End Of Treatment, 2=Somewhat |  | 2
  End Of Treatment, 3=Quite a bit: number analyzed (Participants) | 0 | 5
  End Of Treatment, 3=Quite a bit |  | 0
  End Of Treatment, 4=Very much: number analyzed (Participants) | 0 | 5
  End Of Treatment, 4=Very much |  | 0

8. Secondary Outcome: Change From Baseline (CFB) in European Organisation for Research and Treatment of Cancer Item Library 136 (EORTC IL136) Questionnaire
Description: EORTC IL136 includes items from the EORTC QLQ-C30, a 30-item survey assessing health-related quality of life (HRQoL) in cancer patients, featuring 5 functional scales, 3 symptom scales, 6 single items, and a global health status/HRQoL scale. Functional and symptom scales/items are rated on 4-point scale with options "Not at all," "A little," "Quite a bit," and "Very much". 2 items measuring global health status/quality of life use a 7-point scale ranging from 1 ("Very Poor") to 7 ("Excellent"). Each item has a specific scoring system, and scores were transformed to a 0-100 scale, where higher scores on functional scales and global health status/HRQoL scale indicate better functioning or quality of life, while higher scores on symptom scales/items indicate greater symptom burden. Baseline is defined as the latest assessment with a non-missing value prior to Cycle 1 Day 1 (C1D1), including those from unscheduled visits.
Time Frame: Baseline (Predose), Day 1 of Cycle 2 and Cycle 3; Pre-IDS Evaluation, and End of Treatment (Up to approximately 154 weeks).
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Platinum-taxane | Niraparib
Number analyzed (Participants) | 17 | 19
Scores on scale
  Global Health Status/QoL, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 11 | 11
  Global Health Status/QoL, CFB to CYCLE 2 DAY 1 | 0.00 (19.365) | 3.79 (27.224)
  Global Health Status/QoL, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Global Health Status/QoL, CFB to CYCLE 3 DAY 1 | 7.64 (16.460) | 10.19 (38.814)
  Global Health Status/QoL, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Global Health Status/QoL, CFB to Pre-IDS EVALUATION | -4.17 (22.349) | 9.72 (27.597)
  Global Health Status/QoL, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Global Health Status/QoL, CFB to END OF TREATMENT |  | -23.33 (23.863)
  Rate Your Overall Health, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 11 | 11
  Rate Your Overall Health, CFB to CYCLE 2 DAY 1 | -1.52 (22.918) | 4.55 (27.979)
  Rate Your Overall Health, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Rate Your Overall Health, CFB to CYCLE 3 DAY 1 | 9.72 (16.603) | 9.26 (40.062)
  Rate Your Overall Health, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Rate Your Overall Health, CFB to Pre-IDS EVALUATION | -4.76 (23.956) | 11.11 (29.187)
  Rate Your Overall Health, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Rate Your Overall Health, CFB to END OF TREATMENT |  | -20.00 (18.257)
  Rate Your Overall Quality of Life, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 11 | 11
  Rate Your Overall Quality of Life, CFB to CYCLE 2 DAY 1 | 1.52 (18.936) | 3.03 (28.692)
  Rate Your Overall Quality of Life, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Rate Your Overall Quality of Life, CFB to CYCLE 3 DAY 1 | 5.56 (19.245) | 11.11 (38.188)
  Rate Your Overall Quality of Life, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Rate Your Overall Quality of Life, CFB to Pre-IDS EVALUATION | -3.57 (21.857) | 8.33 (27.386)
  Rate Your Overall Quality of Life, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Rate Your Overall Quality of Life, CFB to END OF TREATMENT |  | -26.67 (32.489)
  Physical Functioning Scale, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 11 | 11
  Physical Functioning Scale, CFB to CYCLE 2 DAY 1 | 0.61 (13.150) | 7.27 (12.808)
  Physical Functioning Scale, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Physical Functioning Scale, CFB to CYCLE 3 DAY 1 | 1.53 (12.702) | 10.37 (16.025)
  Physical Functioning Scale, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Physical Functioning Scale, CFB to Pre-IDS EVALUATION | -1.43 (10.838) | 14.44 (20.403)
  Physical Functioning Scale, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Physical Functioning Scale, CFB to END OF TREATMENT |  | -9.33 (17.385)
  Trouble Doing Strenuous Activity, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 11 | 11
  Trouble Doing Strenuous Activity, CFB to CYCLE 2 DAY 1 | 0.00 (21.082) | 3.03 (27.707)
  Trouble Doing Strenuous Activity, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Trouble Doing Strenuous Activity, CFB to CYCLE 3 DAY 1 | -2.78 (9.623) | 22.22 (23.570)
  Trouble Doing Strenuous Activity, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Trouble Doing Strenuous Activity, CFB to Pre-IDS EVALUATION | -7.14 (19.298) | 22.22 (34.427)
  Trouble Doing Strenuous Activity, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Trouble Doing Strenuous Activity, CFB to END OF TREATMENT |  | 0.00 (33.333)
  Have Trouble Taking a Long Walk, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 11 | 11
  Have Trouble Taking a Long Walk, CFB to CYCLE 2 DAY 1 | 0.00 (21.082) | 21.21 (30.814)
  Have Trouble Taking a Long Walk, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Have Trouble Taking a Long Walk, CFB to CYCLE 3 DAY 1 | 13.89 (30.011) | 11.11 (28.868)
  Have Trouble Taking a Long Walk, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Have Trouble Taking a Long Walk, CFB to Pre-IDS EVALUATION | 4.76 (22.100) | 22.22 (34.427)
  Have Trouble Taking a Long Walk, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Have Trouble Taking a Long Walk, CFB to END OF TREATMENT |  | -6.67 (14.907)
  Have Trouble Taking Short Walk, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 11 | 11
  Have Trouble Taking Short Walk, CFB to CYCLE 2 DAY 1 | 6.06 (20.101) | 9.09 (15.570)
  Have Trouble Taking Short Walk, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 11 | 9
  Have Trouble Taking Short Walk, CFB to CYCLE 3 DAY 1 | 0.00 (33.333) | 7.41 (14.699)
  Have Trouble Taking Short Walk, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Have Trouble Taking Short Walk, CFB to Pre-IDS EVALUATION | -4.76 (17.817) | 16.67 (27.889)
  Have Trouble Taking Short Walk, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Have Trouble Taking Short Walk, CFB to END OF TREATMENT |  | -13.33 (18.257)
  Stay in Bed or Chair During Day, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 11 | 11
  Stay in Bed or Chair During Day, CFB to CYCLE 2 DAY 1 | -3.03 (17.979) | 0.00 (25.820)
  Stay in Bed or Chair During Day, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Stay in Bed or Chair During Day, CFB to CYCLE 3 DAY 1 | -2.78 (22.285) | 7.41 (22.222)
  Stay in Bed or Chair During Day, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Stay in Bed or Chair During Day, CFB to Pre-IDS EVALUATION | 0.00 (18.490) | 0.00 (21.082)
  Stay in Bed or Chair During Day, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Stay in Bed or Chair During Day, CFB to END OF TREATMENT |  | -13.33 (18.257)
  Need Help Eating Dressing Washing, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 11 | 11
  Need Help Eating Dressing Washing, CFB to CYCLE 2 DAY 1 | 0.00 (0.000) | 3.03 (17.979)
  Need Help Eating Dressing Washing, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Need Help Eating Dressing Washing, CFB to CYCLE 3 DAY 1 | 0.00 (0.000) | 3.70 (20.031)
  Need Help Eating Dressing Washing, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Need Help Eating Dressing Washing, CFB to Pre-IDS EVALUATION | 0.00 (0.000) | 11.11 (17.213)
  Need Help Eating Dressing Washing, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Need Help Eating Dressing Washing, CFB to END OF TREATMENT |  | -13.33 (18.257)
  Social Functioning Scale, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 11 | 11
  Social Functioning Scale, CFB to CYCLE 2 DAY 1 | 13.64 (27.707) | 7.58 (36.027)
  Social Functioning Scale, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Social Functioning Scale, CFB to CYCLE 3 DAY 1 | 13.89 (30.841) | 1.85 (22.737)
  Social Functioning Scale, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Social Functioning Scale, CFB to Pre-IDS EVALUATION | 7.14 (27.514) | 8.33 (25.276)
  Social Functioning Scale, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Social Functioning Scale, CFB to END OF TREATMENT |  | 3.33 (18.257)
  Cond Interfere With Family Life, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 11 | 11
  Cond Interfere With Family Life, CFB to CYCLE 2 DAY 1 | 18.18 (31.140) | 6.06 (44.267)
  Cond Interfere With Family Life, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Cond Interfere With Family Life, CFB to CYCLE 3 DAY 1 | 13.89 (33.207) | -7.41 (27.778)
  Cond Interfere With Family Life, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Cond Interfere With Family Life, CFB to Pre-IDS EVALUATION | 14.29 (36.314) | -5.56 (38.968)
  Cond Interfere With Family Life, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Cond Interfere With Family Life, CFB to END OF TREATMENT |  | -6.67 (27.889)
  Cond Interfere Social Activity, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 11 | 11
  Cond Interfere Social Activity, CFB to CYCLE 2 DAY 1 | 9.09 (30.151) | 9.09 (33.635)
  Cond Interfere Social Activity, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Cond Interfere Social Activity, CFB to CYCLE 3 DAY 1 | 13.89 (30.011) | 11.11 (28.868)
  Cond Interfere Social Activity, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Cond Interfere Social Activity, CFB to Pre-IDS EVALUATION | 0.00 (26.149) | 22.22 (17.213)
  Cond Interfere Social Activity, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Cond Interfere Social Activity, CFB to END OF TREATMENT |  | 13.33 (18.257)
  Dyspnea Symptom Scale, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 11 | 11
  Dyspnea Symptom Scale, CFB to CYCLE 2 DAY 1 | -3.03 (10.050) | 3.03 (17.979)
  Dyspnea Symptom Scale, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Dyspnea Symptom Scale, CFB to CYCLE 3 DAY 1 | 0.00 (14.213) | 0.00 (28.868)
  Dyspnea Symptom Scale, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Dyspnea Symptom Scale, CFB to Pre-IDS EVALUATION | 0.00 (13.074) | 0.00 (47.140)
  Dyspnea Symptom Scale, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Dyspnea Symptom Scale, CFB to END OF TREATMENT |  | 6.67 (27.889)
  Were You Short of Breath, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 11 | 11
  Were You Short of Breath, CFB to CYCLE 2 DAY 1 | -3.03 (10.050) | 3.03 (17.979)
  Were You Short of Breath, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Were You Short of Breath, CFB to CYCLE 3 DAY 1 | 0.00 (14.213) | 0.00 (28.868)
  Were You Short of Breath, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Were You Short of Breath, CFB to Pre-IDS EVALUATION | 0.00 (13.074) | 0.00 (47.140)
  Were You Short of Breath, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Were You Short of Breath, CFB to END OF TREATMENT |  | 6.67 (27.889)

9. Secondary Outcome: Change From Baseline (CFB) in European Organisation for Research and Treatment of Cancer Item Library 137 (EORTC IL137) Questionnaire
Description: The OC module (QLQ-OV28) supplements the QLQ-C30 and was designed for participants with local or advanced disease who receive treatment by surgery with or without chemotherapy. It consists of 28 items including 3 functional scales (body image, sexuality, attitude to disease/treatment burden) and 5 symptom scales/items (abdominal/gastrointestinal symptoms, peripheral neuropathy, hormonal/menopausal symptoms, other chemotherapy side effects, and hair loss). A subset of 9 questions will be utilized for this cohort, referred to as the EORTC IL137. The scoring approach is identical to the EORTC QLQ-C30. Scores are transformed to a 0-100 scale, where higher functional scale scores indicate better functioning, and higher symptom scale scores indicate greater symptom burden. Baseline is defined as the latest assessment with a non-missing value prior to C1D1, including unscheduled visits.
Time Frame: as for outcome 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Platinum-taxane | Niraparib
Number analyzed (Participants) | 17 | 19
Scores on scale
  Felt physically Less Attractive, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 12 | 10
  Felt physically Less Attractive, CFB to CYCLE 2 DAY 1 | -2.78 (17.164) | -3.33 (33.148)
  Felt physically Less Attractive, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Felt physically Less Attractive, CFB to CYCLE 3 DAY 1 | -2.78 (33.207) | 7.41 (52.116)
  Felt physically Less Attractive, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Felt physically Less Attractive, CFB to Pre-IDS EVALUATION | 0.00 (18.490) | -16.67 (27.889)
  Felt physically Less Attractive, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Felt physically Less Attractive, CFB to END OF TREATMENT |  | 13.33 (38.006)
  Disease Burden, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 12 | 10
  Disease Burden, CFB to CYCLE 2 DAY 1 | 5.56 (19.245) | 10.00 (27.442)
  Disease Burden, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Disease Burden, CFB to CYCLE 3 DAY 1 | 11.11 (25.950) | 14.81 (50.308)
  Disease Burden, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Disease Burden, CFB to Pre-IDS EVALUATION | 11.90 (24.832) | 0.00 (42.164)
  Disease Burden, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Disease Burden, CFB to END OF TREATMENT |  | 13.33 (44.721)
  Treatment Burden, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 12 | 10
  Treatment Burden, CFB to CYCLE 2 DAY 1 | -8.33 (32.177) | 3.33 (39.907)
  Treatment Burden, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Treatment Burden, CFB to CYCLE 3 DAY 1 | 0.00 (24.618) | 7.41 (32.394)
  Treatment Burden, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Treatment Burden, CFB to Pre-IDS EVALUATION | 2.38 (27.625) | 11.11 (27.217)
  Treatment Burden, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Treatment Burden, CFB to END OF TREATMENT |  | 13.33 (18.257)
  Bloated Feeling Abdomen, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 12 | 10
  Bloated Feeling Abdomen, CFB to CYCLE 2 DAY 1 | -8.33 (35.176) | -10.00 (41.722)
  Bloated Feeling Abdomen, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Bloated Feeling Abdomen, CFB to CYCLE 3 DAY 1 | 0.00 (42.640) | -14.81 (29.397)
  Bloated Feeling Abdomen, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Bloated Feeling Abdomen, CFB to Pre-IDS EVALUATION | 0.00 (29.235) | -5.56 (49.065)
  Bloated Feeling Abdomen, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Bloated Feeling Abdomen, CFB to END OF TREATMENT |  | 6.67 (43.461)
  Change Bowel Habit, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 12 | 10
  Change Bowel Habit, CFB to CYCLE 2 DAY 1 | -33.33 (34.816) | 0.00 (41.574)
  Change Bowel Habit, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Change Bowel Habit, CFB to CYCLE 3 DAY 1 | -13.89 (45.965) | -7.41 (22.222)
  Change Bowel Habit, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Change Bowel Habit, CFB to Pre-IDS EVALUATION | -16.67 (31.351) | -11.11 (40.369)
  Change Bowel Habit, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Change Bowel Habit, CFB to END OF TREATMENT |  | -6.67 (14.907)
  Troubled Pass Flatulence, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 12 | 10
  Troubled Pass Flatulence, CFB to CYCLE 2 DAY 1 | 8.33 (25.126) | -3.33 (24.595)
  Troubled Pass Flatulence, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Troubled Pass Flatulence, CFB to CYCLE 3 DAY 1 | -2.78 (22.285) | -3.70 (35.136)
  Troubled Pass Flatulence, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Troubled Pass Flatulence, CFB to Pre-IDS EVALUATION | 7.14 (26.726) | 0.00 (29.814)
  Troubled Pass Flatulence, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Troubled Pass Flatulence, CFB to END OF TREATMENT |  | -20.00 (29.814)
  Felt Full Quick after Begin Eat, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 12 | 10
  Felt Full Quick after Begin Eat, CFB to CYCLE 2 DAY 1 | -13.89 (22.285) | 0.00 (41.574)
  Felt Full Quick after Begin Eat, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 11 | 9
  Felt Full Quick after Begin Eat, CFB to CYCLE 3 DAY 1 | -15.15 (22.918) | -14.81 (33.793)
  Felt Full Quick after Begin Eat, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Felt Full Quick after Begin Eat, CFB to Pre-IDS EVALUATION | -11.90 (28.063) | 5.56 (25.092)
  Felt Full Quick after Begin Eat, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Felt Full Quick after Begin Eat, CFB to END OF TREATMENT |  | -6.67 (59.628)
  Acid Indigestion or Heartburn, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 12 | 10
  Acid Indigestion or Heartburn, CFB to CYCLE 2 DAY 1 | 2.78 (17.164) | -3.33 (29.187)
  Acid Indigestion or Heartburn, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 12 | 9
  Acid Indigestion or Heartburn, CFB to CYCLE 3 DAY 1 | 5.56 (12.975) | -7.41 (32.394)
  Acid Indigestion or Heartburn, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Acid Indigestion or Heartburn, CFB to Pre-IDS EVALUATION | 7.14 (14.194) | -11.11 (27.217)
  Acid Indigestion or Heartburn, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Acid Indigestion or Heartburn, CFB to END OF TREATMENT |  | 6.67 (27.889)
  Felt Weak in Your Arms or Legs, CFB to CYCLE 2 DAY 1: number analyzed (Participants) | 12 | 10
  Felt Weak in Your Arms or Legs, CFB to CYCLE 2 DAY 1 | -5.56 (19.245) | -6.67 (21.082)
  Felt Weak in Your Arms or Legs, CFB to CYCLE 3 DAY 1: number analyzed (Participants) | 11 | 9
  Felt Weak in Your Arms or Legs, CFB to CYCLE 3 DAY 1 | 18.18 (34.524) | -18.52 (33.793)
  Felt Weak in Your Arms or Legs, CFB to Pre-IDS EVALUATION: number analyzed (Participants) | 14 | 6
  Felt Weak in Your Arms or Legs, CFB to Pre-IDS EVALUATION | 4.76 (34.237) | -11.11 (34.427)
  Felt Weak in Your Arms or Legs, CFB to END OF TREATMENT: number analyzed (Participants) | 0 | 5
  Felt Weak in Your Arms or Legs, CFB to END OF TREATMENT |  | 6.67 (27.889)

10. Secondary Outcome: Number of Participants With Treatment Emergent (TE) Non-serious Adverse Events (Non-SAEs), Treatment Emergent Serious Adverse Events (TESAEs) and Adverse Events of Treatment Emergent (TE) Special Interest (AESIs) by Severity
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose resulted in death, is life threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity, is a congenital anomaly/birth defect, other situations and is associated with liver injury or impaired liver function. SAEs are subsets of AEs. TEAE is an event that emerged during treatment having been absent pretreatment or worsened relative to the pretreatment state. AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding system.
Time Frame: Up to approximately 154 weeks
Population: Safety population included all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-taxane | Niraparib
Number analyzed (Participants) | 17 | 19
Participants
  TE Non-SAEs | 17 | 19
  TESAEs | 4 | 2
  TE AESIs | 0 | 0

11. Secondary Outcome: Number of Participants With Dose Modification Due to TEAEs
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAE is an event that emerged during treatment having been absent pretreatment or worsened relative to the pretreatment state. Number of participants with dose modifications : permanent discontinuation, dose reduction and treatment interruption/delay due to AEs is summarized.
Time Frame: Up to approximately 154 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Platinum-taxane | Niraparib
Number analyzed (Participants) | 17 | 19
Participants
  Permanent Discontinuation | 5 | 4
  Dose Reduction | 14 | 7
  Treatment Interruption/delay | 11 | 11

ADVERSE EVENTS:
Time Frame: All-cause mortality, Treatment-Emergent Serious Adverse Events (TESAEs), and TE Non-SAEs were collected up to approximately 154 weeks.
Description: Safety population included all randomized participants who received at least one dose of study treatment.
Arm/Group | Platinum-taxane | Niraparib
All-Cause Mortality (participants affected / at risk) | 4/17 | 4/19
Serious Adverse Events (participants affected / at risk) | 4/17 | 2/19
Other Adverse Events (participants affected / at risk) | 17/17 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platinum-taxane (N=17) | Niraparib (N=19)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (3) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Pelvic haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Platinum-taxane (N=17) | Niraparib (N=19)
Anaemia (Blood and lymphatic system disorders) | 11 (40) | 10 (24)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (5) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 8 (16) | 3 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (20) | 5 (13)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (4) | 0 (0)
Palpitations (Cardiac disorders) | 3 (4) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eczema eyelids (Eye disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Narrow anterior chamber angle (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 3 (3)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (16) | 6 (9)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal wall pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (14) | 8 (13)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (9) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (2) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (7) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 3 (5) | 1 (1)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (25) | 4 (5)
Peritoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (4) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (3)
Vomiting (Gastrointestinal disorders) | 8 (14) | 4 (7)
Asthenia (General disorders) | 4 (10) | 4 (6)
Early satiety (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 14 (46) | 7 (12)
General physical health deterioration (General disorders) | 1 (2) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 3 (4)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (5) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (2)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (9) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural constipation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative adhesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 2 (3) | 3 (5)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 3 (3) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (17) | 4 (8)
Oxygen saturation decreased (Investigations) | 1 (2) | 0 (0)
Platelet count decreased (Investigations) | 6 (10) | 1 (3)
Weight decreased (Investigations) | 2 (2) | 1 (1)
Weight increased (Investigations) | 4 (8) | 1 (2)
White blood cell count decreased (Investigations) | 2 (5) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 6 (11) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 (5) | 3 (4)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (11) | 3 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (11) | 3 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0)
Temporomandibular pain and dysfunction syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness (Nervous system disorders) | 6 (9) | 1 (1)
Dysaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 7 (18) | 4 (5)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 13 (34) | 1 (1)
Paraesthesia (Nervous system disorders) | 4 (9) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 8 (11) | 9 (9)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast haematoma (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Pelvic haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal haematoma (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 (4) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 4 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (12) | 3 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (11) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 7 (17) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (2)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 3 (3) | 4 (4)
Hypertension (Vascular disorders) | 5 (8) | 6 (11)
Hypotension (Vascular disorders) | 2 (5) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT06964165/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/65/NCT06964165/SAP_002.pdf